

# STATISTICAL ANALYSIS PLAN

A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy, Safety, and Pharmacokinetics of Femoral Nerve Block with EXPAREL for Postsurgical Analgesia in Subjects Undergoing Total Knee Arthroplasty

**Protocol No.:** 402-C-326

**IND No.:** 69,198

**Study Phase:** 3

**Study Drug:** EXPAREL (bupivacaine liposome injectable

suspension)

**Date/Version:** 20 June 2017 / Version 1.0

**Prepared by:** Richard Willey, M.S.

**Sponsor:** Pacira Pharmaceuticals, Inc.

5 Sylvan Way

Parsippany, NJ 07054 Tel: 973-254-3560

#### Confidentiality Statement

The information contained in this document is confidential and the property of Pacira Pharmaceuticals, Inc. It should not be reproduced, revealed, or sent to third parties other than Institutional Review Boards/Independent Ethics Committees and the Investigator's research support staff participating in the conduct of the study without the prior written authorization of Pacira Pharmaceuticals, Inc.

# 1. SIGNATURE PAGE

| Hassan Danesi, MD Senior Medical Director, Clinical Research | 20 Jun 2017 Date |
|---|---|
| James Jones, MD | 26 Jine 2017 |
| Chief Medical Officer | Date |
| Michael Rozycki, PhD Vice President, Regulatory Affairs | 2050N 2017<br>Date |
| Richard Willey, MS | 20JUN2017 |
| Senior Manager, Biostatistics | Date |
| Vincent Yu, PhD | 2/JUN 2017 |
| Senior Director, Biometrics | Date |

# 2. TABLE OF CONTENTS

| 1. | SIGNATURE PAGE | 2 |
|----------|----------------------------------------------------------|----|
| 2. | TABLE OF CONTENTS | 3 |
| 3. | LIST OF ABBREVIATIONS | 5 |
| 4. | INTRODUCTION | 6 |
| 5. | STUDY OBJECTIVES | 7 |
| 5.1. | Primary Objective | 7 |
| 5.2. | Secondary Objectives | 7 |
| 6. | STUDY OVERVIEW | 8 |
| 7. | DEFINITIONS | 11 |
| 8. | ANALYSIS SETS | 15 |
| 9. | STATISTICAL METHODS OF ANALYSIS | 16 |
| 9.1. | General Principles | 16 |
| 9.1.1. | Handling Missing Values | 18 |
| 9.1.1.1. | Area under the VAS-Time Curve | 18 |
| 9.1.1.2. | Exposure, Surgery, and Rescue Medication Date or Time | 19 |
| 9.1.1.3. | Rescue Pain Medication | 19 |
| 9.1.1.4. | Adverse Event or Concomitant Medications Dates or Times | 19 |
| 9.1.1.5. | Adverse Event Severity or Relationship to Study Drug | 20 |
| 9.1.1.6. | Time to Event | 20 |
| 9.1.2. | Multiplicity Adjustments | 20 |
| 9.1.3. | By-Center Analyses | 20 |
| 9.2. | Subject Disposition | 20 |
| 9.3. | Description of Demographics and Baseline Characteristics | 21 |
| 9.3.1. | Demographics | 21 |
| 9.3.2. | Baseline Characteristics | 21 |
| 9.4. | Surgery Characteristics | 22 |
| 9.5. | Intraoperative, Prior and Concomitant Medications | 22 |
| 9.6. | Measurements of Treatment Compliance | 23 |
| 9.7. | Efficacy Analysis | 23 |
| 9.7.1. | Efficacy Endpoints | 23 |
| 9.7.1.1. | Primary Efficacy | 23 |
| 9.7.1.2. | Secondary Efficacy | 23 |
| 9.7.1.3. | Tertiary Efficacy | 24 |
| 9714 | Area under the Curve | 24 |


| Pacira Pharmaceuticals, Inc. EXPAREL® | | 402-C-326 (TKA FNB)<br>Statistical Analysis Plan |
|---|---|---|
| 9.7.1.5. | Opioid Consumption | 24 |
| 9.7.1.6. | Time to First Opioid Rescue Medication Use | 25 |
| 9.7.1.7. | Pain-free | 25 |
| 9.7.1.8. | Overall Benefit of Analgesia Score (OBAS) | 25 |
| 9.7.2. | Methods of Analysis | 26 |
| 9.7.2.1. | Primary Efficacy Analysis | 26 |
| 9.7.2.2. | Secondary Efficacy Analyses | 26 |
| 9.7.2.3. | Tertiary Efficacy Analyses | 27 |
| 9.8. | Safety Analyses | 31 |
| 9.8.1. | Vital Signs | 31 |
| 9.8.2. | Electrocardiograms | 31 |
| 9.8.3. | Neurological Assessments | 32 |
| 9.8.4. | Sensation Tests | 32 |
| 9.8.5. | Degree of motor nerve block Assessments | 33 |
| 9.8.6. | Adverse Events | 33 |
| 9.8.7. | Laboratory Parameters | 35 |
| 9.9. | Pharmacokinetic Analysis | 35 |
| 9.10. | Interim Analysis | 35 |
| 9.10.1. | Pharmacokinetic Review | 35 |
| 9.11. | Significance Testing | 36 |
| 10. | SAMPLE SIZE CALCULATIONS | 38 |
| 11. | REFERENCES | 39 |
| 12. | TIME AND EVENTS SCHEDULE OF STUDY PROCEDURES | 40 |
| 13. | MULTIPLE IMPUTATION EXAMPLE PROGRAM CODE | 41 |
| 14. | TABLE OF CONTENTS FOR TABLE MOCK-UPS | 43 |
| 15. | TABLE OF CONTENTS FOR LISTING MOCK-UPS | 131 |
| 16. | TABLE OF CONTENTS FOR FIGURE MOCK-UPS | 168 |


# 3. LIST OF ABBREVIATIONS

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| AE | Adverse event |
| ANOVA | Analysis of variance |
| ATC | Anatomical therapeutic class |
| AUC | Area under the curve |
| BLOQ | Below the limit of quantification |
| BMI | Body mass index |
| bpm | Beats per minute |
| ĊĪ | Confidence interval |
| CMH | Cochran-Mantel-Haenszel |
| CRF | Case report form |
| CSR | Clinical study report |
| d | Day |
| ECG | Electrocardiogram |
| EMA | European Medicines Agency |
| ER | Emergency room |
| FDA | Food and Drug Administration |
| FNB | Femoral nerve block |
| hr, h | hour |
| ICF | Informed consent form |
| ICH | International Conference on Harmonization |
| ICU | Intensive care unit |
| IV | Intravenous |
| LOCF | Last observation carried forward |
| LS | Least square |
| MedDRA | Medical dictionary for regulatory affairs |
| MMRM | Mixed model repeated measures |
| MPADSS | Modified Postanesthesia Discharge Scoring System |
| min | minutes |
| MED | Morphine equivalent dose in mg |
| n | Number of subjects |
| OBAS | Overall benefit of analgesia |
| OR | Operating room |
| PACU | Postanesthesia care unit |
| PCA | Patient-controlled analgesia |
| PK | Pharmacokinetics |
| PO | Oral |
| ROW | Rest of world |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SE | Standard error |
| SPI | Sum of pain intensity scores |
| TEAE | Treatment-emergent adverse event |
| TKA | Total knee arthroplasty |
| TLF | Table, listings and figures |
| TUG | Timed up-and-go |
| TWT | Timed walk test |
| VAS | Visual analog scale |
| WHO | World Health Organization |
| WHO-DD | World Health Organization – Drug Dictionary |
| wWOCF | Windowed worst observation carried forward |

# 4. INTRODUCTION

This Statistical Analysis Plan (SAP) describes the planned statistical analysis and reporting of the clinical study 402-C-326 titled "A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy, Safety, and Pharmacokinetics of Femoral Nerve Block with EXPAREL for Postsurgical Analgesia in Subjects Undergoing Total Knee Arthroplasty".

This study is intended to evaluate the magnitude and duration of analgesic effect of a single femoral nerve block injection with EXPAREL in subjects undergoing primary unilateral total knee arthroplasty (TKA).

The structure and content of this SAP provide sufficient detail to meet the requirements identified by the US Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials<sup>1</sup>. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association<sup>2</sup> and the Royal Statistical Society<sup>3</sup>, for statistical practice.

The purposes of this SAP are to:

- Outline the types of analyses and presentations of data that will form the basis for drawing conclusions to the study objectives and hypotheses outlined in the protocol.
- Explain in detail how the data will be handled and analyzed, adhering to commonly accepted standards and practices for Good Statistical Practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or manuscripts. Post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc, unplanned, or exploratory analyses performed will be clearly identified as such in the final CSR.

The following documents were reviewed in preparation of this SAP:

- Amendment 3 of Protocol 402-C-326 issued on 7Nov2016.
- Amendment 2 of Protocol 402-C-326 issued on 28Sep2016.
- Amendment 1 of Protocol 402-C-326 issued on 15Feb2016.
- Original Protocol 402-C-326 issued on 16Nov2015.
- CRF version 1.0 issued on 25Nov2015.
- ICH Guidance on Statistical Principles for Clinical Trials (E9).

The reader of this SAP is encouraged to also read the clinical protocol and other identified documents for details on the planned conduct of this study. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analyses.


# 5. STUDY OBJECTIVES

# 5.1. Primary Objective

The primary objective of this study is to evaluate the magnitude and duration of the analgesic effect achieved following single-dose injection femoral nerve block with EXPAREL in subjects undergoing primary unilateral total knee arthroplasty (TKA).

# 5.2. Secondary Objectives

The secondary objectives of this study are to further assess the efficacy, safety, and pharmacokinetic (PK) profiles of EXPAREL as well as the onset and duration of sensory and motor function blockade following administration for analgesia in subjects undergoing primary unilateral TKA.

#### 6. STUDY OVERVIEW

This is a Phase 3, double-blind, placebo-controlled, randomized study. Subjects will be monitored for 5 days after surgery and followed for 30 days after surgery. Subjects will be randomized (1:1:1) to receive a 20mL injection of EXPAREL 133mg (10mL of EXPAREL 266mg/20mL expanded with 10mL of normal saline), EXPAREL 266mg or placebo (normal saline) via an ultrasound guided single-injection femoral nerve block approximately 1 hour before surgery.

Subjects will be allowed rescue medication upon request to control their pain. Rescue medication will be oral (PO) immediate release oxycodone. If subject cannot tolerate PO medication, intravenous (IV) morphine or hydromorphone may be used as rescue medication.

Pain will be assessed using a 10 cm visual analog scale (VAS). Pain will be assessed at multiple timepoints during the study.

Other postsurgical assessments include:

- Postsurgical opioid consumption;
- Overall benefit of analgesia score (OBAS);
- Subject satisfaction with overall analgesia using a 5-point Likert scale;
- Subject's discharge ready as assessed by Modified Postanesthesia Discharge Scoring System (MPADSS);
- Unscheduled phone calls or office visits related to pain;
- Clinical laboratories;
- Vital sign measurements;
- ECGs;
- Neurological assessment;
- Sensory function assessment at 2 locations as measured by:
  - o Cold,
  - o Pinprick,
  - Light touch;
- Degree of motor nerve block, both active and passive, assessment as measured by:
  - o Angle of flexion,
  - o Angle of extension,
- Adverse events;
- Concomitant medications;
- Timed walk test (added with Amendment 2 of protocol);
- Timed up-and-go test (added with Amendment 2 of protocol);


• Stair climb test (added with Amendment 2 of protocol).

Following are the major changes in Amendment 2 of the protocol impacting the statistical analyses (see Amendment 2 of the protocol for a complete record of changes):

- Under Amendment 1 all subjects were to be in-hospital through 120 hours; under Amendment 2 subjects are to remain in-hospital through 108 hours.
- Under Amendment 1 all subjects had PK assessments at the same scheduled time; under Amendment 2 a population PK approach was adopted where subjects were randomized to one of two PK sampling schemes.
- Time points of the motor and sensitivity assessments were changed from baseline (on Day 0 prior to the nerve block); at approximately 15, 30, and 45 minutes; at 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, and 120 hours to baseline (on Day 0 prior to the nerve block); at approximately 15, 30, and 45 minutes; at 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, and 108 hours; and at hospital discharge to align with the T<sub>max</sub> observed in the PK interim analysis.
- Duration of in-house portion of the study was changed from 5 days to 4 days.
- Added physical therapy assessments of timed walk test, timed up-and-go test, and stair climb test scheduled for 8am and  $8pm \pm 2$  hours.
- Assessment schedules were changed for:
  - Pain
    - From 'upon arrival at the PACU; at 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120 hours; and immediately prior to each administration of rescue pain medication through 120 hours';
    - To 'upon arrival at the PACU, every 15 minutes while in the PACU, and prior to PACU discharge; at 6, 12, 24, 36, 48, 60, 72, 84, 96, and 108 hours; and immediately prior to each administration of rescue pain medication through 108 hours.'

#### Vital signs

- From 'baseline (on Day 0 prior to the nerve block); upon arrival at the PACU; at 6, 12, 24, 36, 48, 60, 66, 72, 78, 84, 96, 108, and 120 hours; and on postsurgical Days 7 and 10';
- To 'baseline (on Day 0 prior to the nerve block); every 5 minutes during performance of the block and up to 30 minutes after the end of the injection and then every 15 minutes after the block until entering the operating room; upon arrival at the PACU; at 6, 9, 12, 24, 36, 48, 56, 60, 64, 68, 72, 76, 80, 84, 96, and 108 hours; and on postsurgical Days 6 and 10.'

#### 12-lead ECG

■ From 'baseline (on Day 0 prior to the nerve block); upon arrival at the PACU; at 6, 12, 24, 36, 48, 60, 66, 72, 78, 84, 96, 108, and 120 hours; and on postsurgical Days 7 and 10';


- To 'baseline (on Day 0 prior to the nerve block); upon arrival at the PACU; at 6, 9, 12, 24, 36, 48, 56, 60, 64, 68, 72, 76, 80, 84, 96, and 108 hours; and on postsurgical Days 6 and 10.'
- Sensory and motor function
  - From 'baseline (on Day 0 prior to the nerve block); at approximately 15, 30, and 45 minutes; and at 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, and 120 hours':
  - To 'baseline (on Day 0 prior to the nerve block); at approximately 15, 30, and 45 minutes prior to the OR; prior to discharge from the PACU; at 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, and 108 hours; and at hospital discharge.'

# Neurological

- From 'baseline (on Day 0 prior to the nerve block); upon arrival at the PACU; at 6, 12, 24, 36, 48, 60, 66, 72, 78, 84, 96, 108, and 120 hours; and on postsurgical Days 7 and 10';
- To 'baseline (on Day 0 prior to the nerve block); upon arrival at the PACU; at 6, 9, 12, 24, 36, 48, 56, 60, 64, 68, 72, 76, 80, 84, 96, and 108 hours; and on postsurgical Days 6 and 10.'

Following are the major changes in Amendment 3 of the protocol impacting the statistical analyses are as follows (see Amendment 3 of the protocol for a complete record of changes):

- Sample size calculation changed from 90% power to 80% power. Resulting in a drop in sample size from 300 to 231 subjects.
- Discharge readiness assessments schedule was changed
  - o From 'Discharge readiness at 12, 24, 36, 48, 60, 72, 84, and 96 hours or discharge ready, whichever occurs first';
  - o To '12, 24, 36, 48, 60, 72, 84, and 96 hours or until the subject is determined to be discharge ready, whichever occurs first.'
- Post-surgical medications were amended
  - From 'Patient-controlled analgesia (PCA) is not permitted. No other analgesic agents, including NSAIDs, are permitted through 108 hours (postsurgical Day 4)';
  - To 'Patient-controlled analgesia (PCA) is not permitted. Postsurgically, all subjects will receive the following scheduled medications until hospital discharge: Acetaminophen/paracetamol up to 1000 mg PO or IV every 8 hours (q8h) unless contraindicated. The total daily dose of acetaminophen/paracetamol should not exceed 3000 mg and Cyclobenzaprine (eg, Flexeril®) 10 mg PO x1 dose (PRN at the surgeon's discretion). No other analgesic agents, including NSAIDs, are permitted through 108 hours (postsurgical Day 4).'


#### 7. **DEFINITIONS**

#### Study Day

Study Day is calculated as the date of event minus the date of surgery plus one (1), if the date of event is on or after the date of surgery. Study Day is based on the calendar dates, thus days before the date of surgery have negative values while those on or after the date of surgery are positive.

This Study Day definition differs from the protocol defined Study Day. By this definition Day 1 is the day of the operation while the protocol defines this as Day 0. The definition assigning the operation to Day 1 aligns with the CDISC implementation guidance and FDA expectations.

# Treatment-emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are those with onset between the start date and time of study drug administration and end of study (Study Day 30±3 days).

#### Time 0 (zero)

Time 0 is defined as the date and time of the start of study drug administration.

#### Time Periods

All schedule times have a window associated with them (see Time and Events Schedule for individual timepoint windows). Various time frames are used in the data analyses which are dependent on these windows. The table below defines the actual elapsed times with allowance for the windows that can be included in the window.

| Defined time frame (hrs) | Acceptable elapsed times (hrs) |
|--------------------------|--------------------------------|
| 0-12 | [0 to 13] |
| 0-24 | [0 to 25] |
| 0-48 | [0 to 50] |
| 0-72 | [0 to 76] |
| 0-96 | [0 to 100] |
| 0-Day 6 | [0 to 168] |
| 0-Day 10 | [0 to 264] |
| 24-48 | [23 to 50] |
| 48-72 | [ 46 to 76] |
| 72-96 | [68 to 100] |
| 48-96 | [46 to 100] |

If there are two or more data points that fit the time window, the data point that occurs the latest in the window should be used. For example when selecting the data point for the 48 hour timepoint, if a subject has data points collected at 47 and 49 hours then the 49 hour timepoint should be used. In this example the 49 hour timepoint record will be used as the end and start of all time intervals, thus the 0-48 hour interval will end using the 49 hour record and the 48-72 hour interval will start using the same 49 hour record. In addition, if there are two measurements for a given assessment at the exact same time, the measurement with the highest value should be used.


#### Baseline

Baseline is defined as the last available measurement or assessment prior to start of study treatment.

#### **Sensation Loss**

Sensation loss is when the subject reports absence of sensation for the sensory test (cold, pinprick or light touch) at each location [foot (anterior cutaneous nerve) and thigh (saphenous nerve)]. Subjects may experience loss of sensation multiple times and at different times in different locations. A subject must have a return of sensation in the same sensory test in the same location before another loss of sensation can occur.

# Time to Sensation Loss

Time to first loss of sensation is the first timepoint after baseline at which one of the three sensations (cold, pinprick and light touch) is absent at any location. If sensation is not lost, time to sensation loss will be censored at the last available sensory assessment available for that subject. Subjects who experience multiple losses of sensation will have multiple times to sensation loss but the time to first sensation loss will be used for analysis of time to first sensation loss

#### Return of Sensation

Return of sensation is when a subject reports the presence of sensation after reporting a loss of sensation for the same sensory test (cold, pinprick or light touch) at the same location as the loss. Subjects may experience returns of sensation multiple times. A subject must experience multiple losses of sensation before multiple returns can be experienced. Subjects who experience multiple returns of sensation will have multiple times to sensation return.

#### Time to Return of Sensation

Time to return of sensation is when all three sensations (cold, pinprick and light touch) are present after a subject experienced a loss of sensation in at least one of the sensory tests. If sensation doesn't return, it will be censored at the time of the last sensory assessment available for that subject. Only subjects who experience a loss of sensation can experience a return of sensation.

# **Duration of Sensory Loss**

Duration of sensory loss is defined as the time from sensation loss to the time of sensation return. Subjects who never lose sensation will not be included in any analysis of Duration of Sensory Loss. If sensation doesn't return, then duration will be censored and is defined as the time between sensation loss and last sensory assessment.

Duration will be calculated for each loss-return cycle for those subjects with multiple cycles. If after the last sensation loss there is no return of sensation, the duration of the last cycle will be censored and defined as the time between sensation loss for that cycle and last sensory assessment.

Total duration is the sum of all durations for a subject.

# Onset of Motor Function Loss


Onset of motor function loss is the first timepoint after baseline where at least one of the motor function assessments (angle of flexion [active and passive] or angle of extension [active and passive]) meets the criteria below. Passive assessments are assisted by medical staff while active assessments are done without medical assistance.

Loss of motor function is defined as:

- L1. If the subject's baseline active flexion angle is  $\geq 80^{\circ}$  then an active flexion angle  $< 80^{\circ}$  indicates loss of motor function; otherwise a change (post-baseline) in active flexion angle  $\leq -10^{\circ}$  indicates loss of motor function **OR**
- L2. If the subject's baseline active extension angle is  $\leq 10^{\circ}$  then an active extension angle >  $10^{\circ}$  indicates loss of motor function; otherwise a change (post-baseline) in active extension angle >  $10^{\circ}$  indicates motor function loss.

A subject satisfying at least one of the loss criteria L1 or L2 is considered as having loss of motor function. These individual criteria are used to define loss of function within each specific motor function test.

#### Return of Motor Function

Return of motor function is defined when the following criteria R1 and R2 are met:

- R1. Active flexion angle is either  $\geq 80^{\circ}$  for those subjects whose baseline was  $\geq 80^{\circ}$  or change from baseline is  $\geq -10^{\circ}$  for subjects whose baseline flexion was  $\leq 80^{\circ}$  **AND**
- R2. Active extension angle is  $\leq 10^{\circ}$  for those subjects whose baseline extension was  $\leq 10^{\circ}$  or change from baseline is  $< 10^{\circ}$  for those subjects whose baseline was  $> 10^{\circ}$ .

A subject who satisfies return criteria R1 and R2 is considered as having complete return of motor function. The individual criteria are used to define return of function within a specific motor function test.

#### Time to Return of Motor Function

Time to return of motor function is the time from first loss of motor function to last return of motor function for the motor assessment. If a subjects doesn't have return of motor function, the time to return of motor function will be censored on the date and time of last motor function assessment. For those subjects who never lose motor function, time to return will be missing; these subjects will not be included in any analysis of time to return.

#### Loss-Return Cycle

A loss-return cycle is the event where a subject has loss and return of sensory or motor function. Subjects may experience multiple cycles. Cycles are defined separately for each sensory and motor function tests.

#### Ready for Discharge

Ready for discharge is defined as a total score of 9 or more on the MPADSS. The total score is the sum of all scores. If there are missing data then the total score will not be calculated.

# Sum of Pain Intensity Score (SPIS)


Sum of pain intensity scores (SPIS) are calculated by summing the imputed VAS scores for the time-frames of interest.

# Region

Region is defined as US and ROW where ROW is any site outside of the US.


# 8. ANALYSIS SETS

The safety analysis set will include all subjects who receive study drug. All analyses based on the safety set will be by actual treatment received.

The efficacy analysis set will include all subjects in the safety analysis set who undergo the planned surgery. All analyses based on the efficacy analysis set will be by randomized treatment regardless of treatment actually received.

The per-protocol efficacy analysis set will include all subjects in the efficacy analysis set and do not have any important protocol deviations. Important protocol deviations may include, but are not limited to, the following:

- 1) Bilateral TKA or other concurrent surgical procedure
- 2) 50% or more of the rescue medications are missing a VAS assessment (baseline through 72 hours +/-4 hours) within 30 minutes prior to rescue medication use and at least 4 rescue medication doses are missing the associated VAS assessments within 30 minutes prior to rescue medication use.
- 3) Missing two or more scheduled VAS assessments between start study drug administration as the baseline VAS assessment and the 72 hour VAS assessment.
- 4) Subject did not receive the study treatment to which he/she was randomized (determined after database lock and unblinding).

All analyses for the per-protocol analysis set will be by randomized treatment.


# 9. STATISTICAL METHODS OF ANALYSIS

# 9.1. General Principles

The statistical analyses will be reported using summary tables, listings, and figures (TLFs). All analyses and tabulations will be performed using SAS® Version 9.1 or later. Continuous variables will be summarized using descriptive statistics [sample size (n), mean, standard deviation (SD), minimum, median, and maximum]. Categorical variables will be tabulated with number and percentage of subjects. Unless otherwise noted, percentages will be based on the number of subjects in the treatment group within the population.

Individual subject data will be provided in listings. All listings will be sorted by treatment, site, subject, and, if applicable, collection date and time.

Unless otherwise stated summaries will present data across all sites (overall).

Unless otherwise noted, tabulations of categorical data will present only those categories appearing in the data.

On all figures, the comparator treatment will be represented in black with solid lines and filled squares; EXPAREL will be represented in red with solid lines and dots.

For tables presenting summaries of VAS scores, if more than one VAS score is presented for a specific timeframe/timepoint of interest, the highest score within that specific timeframe/timepoint should be used.

Plots of the VAS scores will show both observed and imputed scores. A change in color and line type will differentiate the imputed VAS scores. Imputed values will be represented by blue and green symbols and dashed lines for the comparator and EXPAREL respectively. VAS scores obtained immediately prior to rescue will be indicated by a change in symbol. For the comparator the symbol should be a triangle, for EXPAREL the symbol is a star. The following table shows the SAS symbol statements:

| Treatment | VAS Score | SAS Statement |
|---|---|---|
| Comparator | Observed | symbol font=marker interpol=j line=1 value=U color=black |
| | Imputed | symbol font=marker interpol=j line=3 value=C color=brown |
| EXPAREL 133 mg | Observed | symbol font=marker interpol=j line=1 value=W color=red |
| | Imputed | symbol font=marker interpol=j line=3 value=V color=crimson |
| EXPAREL 266 mg | Observed | symbol font=marker interpol=j line=1 value=W color=blue |
| _ | Imputed | symbol font=marker interpol=j line=3 value=V color=cadetblue |

Note the symbol statement number will be dependent on the sort order of the treatment and VAS score group indicator variables.

Sites with fewer than 5 subjects per treatment arm will be pooled with other sites for analysis. US sites will be pooled with other small US sites based on the US Census Bureau geographic regions (see Table 1) and European sites will be pooled with other small European sites based on country. Sites meeting the criteria for pooling will be pooled with other similar sites within their census division. If the resulting pooled site within a division still doesn't have enough subjects per treatment group, it will be pooled with the site within the division with the smallest enrollment that doesn't meet the pooling criteria. If all sites within a division are pooled and the resulting pooled site still meets the pooling criteria, the site will be pooled with other small sites


within the region. If the pooled site with the region still meets the pooling criteria it will be pooled with the site with the smallest enrollment from the neighboring regions.

Table 1: US Census Regions and Divisions

| Region | Division | State |
|---|---|---|
| Midwest East North Central | | Illinois, Indiana, Michigan, Ohio, Wisconsin |
| Midwest | West North Central | Iowa, Kansas, Minnesota, Missouri, Nebraska, North Dakota, South Dakota |
| Northeast | Middle Atlantic | New Jersey, New York, Pennsylvania |
| Northeast | New England | Connecticut, Maine, Massachusetts, New Hampshire, Rhode Island, Vermont |
| East South Central South South Atlantic | | Alabama, Kentucky, Mississippi, Tennessee |
| | | Delaware, District of Columbia, Florida, Georgia, Maryland, North Carolina, South Carolina, Virginia, West Virginia |
| | West South Central | Arkansas, Louisiana, Oklahoma, Texas |
| West | Mountain | Arizona, Colorado, Idaho, Montana, Nevada, New Mexico, Utah, Wyoming |
| vv CSt | Pacific | Alaska, California, Hawaii, Oregon, Washington |

Subjects who use opioid rescue medication will have the pain scores obtained after rescue replaced using pain scores obtained prior to rescue medication use. Pain scores obtained during the opioid medication window will be replaced. For this study the prescribed opioid rescue medication is oxycodone; however morphine or hydromorphone may be used. The durations of effect for various opioids are listed in Table 2.

**Table 2: Opioid Windows** 

| Medication | Route | Window Used to Impute VAS |
|---------------------------------|--------------|---------------------------|
| Oxycodone, Oxycocet, Percocet, | PO, IM,IV,SC | 6 hours |
| acetaminophen-oxycodone, | | |
| Oxycontin | | |
| Morphine | IV, PO, SC | 4 hours |
| Hydromorphone (Dilaudid), | IV | 2 hours |
| Hydromorphone hydrochloride | | |
| Hydromorphone (Dilaudid), | PO, IM, SC | 4 hours |
| Hydromorphone hydrochloride | | |
| Hydrocodone | PO | 6 hours |
| Fentanyl | IV, PO, IM | 6 hours |
| Vicodin, Norco, Lorcet, Lortab, | PO | 6 hours |
| hydrocodone-acetaminophen | | |
| Codeine (Tylenol 3, | PO | 6 hours |
| acetaminophen-coedine, | | |
| Paracetamol Forte, Tylenol 4) | | |
| Ultram, Tramadol, Tramacol | PO | 6 hours |
| hydrochloride | | |

PO = oral; IV = intravenous; VAS = visual analog scale.

If other rescue medications are given then the window will be determined post-hoc. If a combination opioid product is given then the window will be determined by the opioid part of the medication. Opioids given post surgically with an indication such as 'anesthesia maintenance' will not be included for imputation purposes.


All non-efficacy tables will present EXPAREL 133 mg, EXPAREL 266 mg, All EXPAREL (combined doses), placebo, and all treatments as separate columns.

Efficacy tables will present EXPAREL 133 mg, EXPAREL 266 mg, and placebo as separate columns.

If there are multiple VAS records with the same actual date/time for a given subject, then the record with the highest VAS score will be used for that actual date/time for all endpoint derivations, summaries, and analyses.

# 9.1.1. Handling Missing Values

- 9.1.1.1. Area under the VAS-Time Curve
- 9.1.1.1.1. Multiple Imputation Method

Rubin's (1987)<sup>4</sup> multiple imputation procedure will be applied to replace each missing value with a set of plausible values that represent the uncertainty about the right value to impute. This multiple imputation method is being implemented per the advice provided in "The prevention and treatment of missing data in clinical trials."<sup>5</sup> For calculation of area under the curve (AUC) of VAS pain intensity scores, the windowed worst observation carried forward (wWOCF) multiple imputation procedure will be used in the following order:

- a) Windowed worst observation carried forward (wWOCF) for rescue medications.
  - For subjects who take a rescue medication, their VAS scores recorded within the window of controlled type of rescue medication (see Table 2) will be replaced by the 'worst' observation. The non-rescue VAS score recorded right before taking a rescue medication (start of Rescue window) is considered as the 'worst' observation. This non-rescue worst VAS score shall be after the end of previous rescue window, where a rescue window ends once a subject is no longer considered under the effect of opioids (see Table 2 for individual rescue medication durations). If there is no value available between the end of previous rescue window and the start of the current rescue window, then the first VAS score recorded on or right after the start of the current rescue window will be used for the imputation. VAS scores recorded prior to the end of surgery will not be considered.
- b) After the wWOCF imputation, described in Step a, subject data still missing scheduled assessments with a non-monotone missing pattern (i.e., all pain scores between the last non-missing score and last timepoint) will have missing scores imputed using the Markov-Chain Monte-Carlo (MCMC) method (Schafer 1997)<sup>6</sup> within each treatment, which will be applied in the multiple imputation procedure for arbitrary missing patterns. This MCMC method will simulate 10 datasets with only monotone missing data. In order to achieve the stationary distribution and to avoid dependency within samples generated by MCMC method, the number of iteration for the burn in period will be set to 2000 and the number of iterations between each sample will be set to 1000 (i.e., NBITER=2000 and NITER=1000.)


- c) The AUC and SPIS at various time intervals will be derived from the VAS scores resulting from Step b.
- d) Rubin's (1987) synthesizing procedure for the multiple imputed data will be applied to synthesize analysis results for each imputation. SAS PROC MIANALYZE will be used for this procedure. The mean parameter estimates, the asymptotic variance for this mean from the imputed data analysis in Step c will be created based on Rubin and Schenker method (1986)<sup>7</sup>.

SAS pseudo-code for multiple imputations is provided in Section 13.

# 9.1.1.2. Exposure, Surgery, and Rescue Medication Date or Time

It is expected that all necessary information on study drug exposure, surgery, and postsurgical rescue medication dates and times will be complete. Any such information that is missing and cannot be obtained through query resolution may be imputed, on a case-by-case basis, in a conservative manner that minimizes bias. For example, if pain medication taken on Day 1 has no time of administration recorded, the imputed time will be the end of surgery.

#### 9.1.1.3. Rescue Pain Medication

For calculation of the total rescue pain medication usage (IV Morphine Equivalent) through a time point, if a subject is discontinued early (e.g., dies, withdraws consent, is withdrawn from the study, or is lost to follow-up) before the end of the time interval (e.g., 24 hours after study drug administration), his or her total rescue pain medication usage through the time interval will be a projected amount. For example, if a subject discontinues early at 6 hours after surgery, the projected amounts through 24 hours will be actual amount + average amount (actual amount/6 hours) multiplied by the number of hours remaining in the time interval (18=24-6).

#### 9.1.1.4. Adverse Event or Concomitant Medications Dates or Times

For AEs or concomitant medications with missing or partially missing start/stop date/time, the following imputation rules will be applied:

For partial start date/time:

- If the year is unknown, then the date will be assigned the date and time of first dose of study treatment.
- If the month is unknown, then:
  - i) If the year matches the year of the dose of study drug date, then the month and day of the dose of study drug date will be used to impute the missing month and corresponding day.
  - ii) Otherwise, 'January' will be assigned.
- If the day is unknown, then:
  - i) If the month and year match the month and year of the dose of study drug date, then the day of the dose of study drug date will be imputed.
  - ii) Otherwise, '01' will be assigned.
- If the time is unknown, then:
  - i) If the date (day, month, and year) matches the date of the administration of study drug, then the time of the dose of study drug time will be imputed.


ii) Otherwise, '00:00' will be assigned.

For partial stop date/time:

- If the year is unknown, then the date will be assigned the date subject discontinued from study, time will be set to the last time of the day ('23:59').
- If the month is unknown, then month subject discontinued from study will be assigned.
- If the day is unknown, then the last day of the month will be assigned.
- If the time is unknown, then the last time of the day will be assigned ('23:59').

#### 9.1.1.5. Adverse Event Severity or Relationship to Study Drug

If severity of an AE is not reported, then for tables of AEs by severity, the event will be classified as 'Severe'. If relationship to study drug is not reported for an AE, then for tables of study-drug related AEs, the event will be assigned the relationship of 'definite'. Tables presenting related AEs will include all AEs with relationships of 'possible', 'probable' or 'definite' as assessed by the investigator.

# 9.1.1.6. Time to Event

For calculating time to an event when only the hour is reported, the minutes will be set to zero.

# 9.1.2. Multiplicity Adjustments

Significance testing will be based on "Graphical approaches for multiple comparison procedures using weighted Bonferroni, Simes, or parametric tests" (Bretz 2011)<sup>8</sup>. The initial alpha will be set to 0.025 for each of the primary efficacy analyses. The diagram for sequential testing is in Section 9.11.

Any analyses of tertiary efficacy endpoints are for sensitivity or exploratory purposes. No multiplicity adjustments need be made for these endpoints.

# 9.1.3. By-Center Analyses

By-site summaries will present descriptive statistics only; no statistical analyses will be performed on individual sites. By-site summaries will be presented for disposition, demographics, primary efficacy endpoint and secondary efficacy endpoints. By-site summaries will present both pooled and individual sites. The pooled site should be presented first immediately followed by the sites within that pool.

#### 9.2. Subject Disposition

Subject disposition summaries will include the number of subjects that were:

- Screened,
  - Screen failure
  - o Enrolled
- Randomized
  - Randomized not treated.
  - o Randomized treated,
- In the safety analysis set,
- In the efficacy analysis set.


- In the per-protocol analysis set,
- Protocol
  - o Enrolled under Amendment 2
  - o Enrolled under Amendment 1
- Completed the study as planned,
- Discontinued from the study, and
- Reasons for discontinuation from the study.

Percentages will be reported for the screen failures and enrolled using the number of subjects screened as the denominator; efficacy analysis set and per-protocol analysis set will use the number of subjects randomized, treated, and having surgery as denominator for percentages; all other percentages will use the number of subjects randomized and treated as denominator.

The safety analysis set and enrollment data will be presented as treated. All other data will be presented as randomized.

The disposition summary will present the data for each treatment group (EXPAREL 133 mg, EXPAREL 266 mg, placebo), EXPAREL treatments combined (All EXPAREL), and across treatment groups (Total). This summary table will present overall sites and for each site separately.

# 9.3. Description of Demographics and Baseline Characteristics

# 9.3.1. Demographics

The summary of demographic data will present:

- Age (years) descriptive statistics
- Sex − n (%)
- Ethnicity n (%)
- Race n (%)
- Country n (%)

Age is calculated from the date the subject signed the informed consent form (ICF) and birth. It is presented as the number of years between, rounding down to the nearest integer year. For partial birthdates, impute the first of the month for missing day and January for missing month to calculate age. It is presumed that birth year is known.

The demographic summary will present the data for each treatment group (EXPAREL 133 mg, EXPAREL 266 mg, placebo), EXPAREL treatments combined (All EXPAREL), and across treatment groups (Total). Summaries will be provided for all (safety, efficacy, and per-protocol) analysis sets. This summary will present overall sites and for each site separately.

#### 9.3.2. Baseline Characteristics

The summary of baseline characteristic data will present:

- American Society of Anesthesiologists (ASA) Classification n (%)
- Baseline VAS scores
- Baseline neurological assessments
- Baseline ECG interpretation
- Baseline degree of motor nerve block assessments (active and passive)


- Flexion
- Extension
- Height (cm)
- Weight (kg)
- Body Mass Index (BMI) (kg/m<sup>2</sup>)
- Baseline vital signs
  - o Heart rate (bpm)
  - Systolic blood pressure (mmHg)
  - Diastolic blood pressure (mmHg)

The formula for BMI is  $w/(h^2)$ , where w is weight in kilograms and h is height in meters. Weight in pounds will be converted to kilograms using the conversion factor of 2.2046 pounds to 1 kilogram. Height in inches will be converted to centimeters using the conversion factor of 2.54 centimeters to 1 inch. Height in centimeters will be converted to meters using the conversion factor of 100 centimeters to 1 meter

Baseline characteristics summaries will present the data for each treatment group (EXPAREL 133 mg, EXPAREL 266 mg, All EXPAREL doses, placebo) and across treatment groups (Total). Summaries will be provided for all (safety, efficacy, and per-protocol) analysis sets. This summary table will show summaries across all sites and for each site separately.

Descriptive statistics (n, mean, SD, median, minimum and maximum) will be provided for VAS scores, degree of motor blockade, height, weight, BMI, and vital signs. The number and percent of subjects will be tabulated for the various categories of sensory assessments, neurological assessments, and ECG interpretation.

#### 9.4. Surgery Characteristics

Surgery characteristics include duration of surgery, tourniquet use (yes/no), duration of tourniquet inflation, maximum tourniquet inflation pressure and drain use (yes/no). Duration of surgery is calculated as the difference between the end of surgery and start of surgery times and reported in hours. Duration of tourniquet use is calculated as the difference between the end of tourniquet inflation and removal and reported in hours. Descriptive statistics will be provided for the duration of surgery, tourniquet inflation and duration of drain by treatment group and across all treatment groups. Use of tourniquet and drains (yes/no) will be tabulated by treatment group and across all treatment groups.

# 9.5. Intraoperative, Prior and Concomitant Medications

Intraoperative, prior and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO-DD) and will be classified according to the anatomical therapeutic chemical (ATC4) classification term and standard medication name.

Intraoperative medications are defined as medications given as part of the surgical procedure. These may include anesthesia, opioids or other medications with start and stop dates on the day of surgery and start and stop times overlapping with the surgery start and stop times.

Prior medications are defined as medications with a stop date and time prior to the start of study drug administration.


Concomitant medications are defined as medications taken after the start of study drug administration (i.e., started prior to the start of study drug administration and continued after or started after the start of study drug administration).

Intraoperative, prior, and concomitant medications will be summarized separately using n (%) of subjects for each treatment group and across treatment groups by ATC class term and standard medication name for the safety analysis set. Subjects may have more than one medication per ATC category and standard medication name. At each level of subject summarization, a subject will be counted once if one or more medications are reported by the subject at that level.

A listing mapping the ATC term and standard medication name to verbatim term will be presented.

# 9.6. Measurements of Treatment Compliance

Study treatment is administered by a party other than the subject, therefore compliance is assured

# 9.7. Efficacy Analysis

For Primary and Secondary Efficacy Analyses, descriptive statistics that are appropriate for the efficacy variable will also be shown by site but no statistical analyses will be performed within a site. The primary and secondary efficacy analyses will be performed on the efficacy and per-protocol analysis sets. Tertiary efficacy analyses will be performed on the efficacy analysis set only.

# 9.7.1. Efficacy Endpoints

#### 9.7.1.1. Primary Efficacy

The primary endpoint is AUC of the VAS pain intensity scores through 72 hours [AUC(0-72)].

#### 9.7.1.2. Secondary Efficacy

The following secondary endpoints will be analyzed as described in Section 9.1.2:

- Total postsurgical opioid consumption (mg) through 72 hours.
- Percentage of opioid-free subjects through 72 hours.
- Time to first rescue medication (opioid) dose through 72 hours.


# 9.7.1.3. Tertiary Efficacy

- The AUC of the VAS pain intensity scores through 12, 24, 48 and 96 hours.
- The AUC of VAS pain intensity scores from 24-48, 48-72 and 72-96 hours.
- VAS pain intensity scores at each assessed timepoint.
- Proportion of subjects who are pain free (VAS score of  $\leq 1.5$ ) at each assessed timepoint.
- SPIS through 24, 48, 72, and 96 hours.
- SPIS from 24-48, 48-72, and 72-96 hours.
- Total opioid consumption in IV morphine equivalents through 24, 48 and 96 hours.
- Total opioid consumption in IV morphine equivalents from 24-48, 48-72 and 72-96 hours.
- Percentage of subjects who are opioid-free through 24, 48 and 96 hours.
- Overall benefit of analgesia scale (OBAS) total score at 24 and 72 hours and Day 10.
- Subject satisfaction with overall analgesia at 24 and 72 hours and Day 10.
- Proportion of subjects ready for discharge at 12, 24, 36, 48, 60, 72, 84 and 96 hours
- Number of unscheduled phone calls or office visits related to pain after discharge through Day 29.
- Timed walk test at screening, postsurgically on day of surgery (Day 1) and q12h starting on Day 2 through hospital discharge.
- Timed up-and-go at screening, postsurgically on day of surgery (Day 1) and q12h starting on Day 2 through hospital discharge.
- Stair climb test at screening, postsurgically on day of surgery (Day 1) and q12h starting on Day 2 through hospital discharge.

#### 9.7.1.4. Area under the Curve

Area under the pain-time curve is derived using the trapezoidal rule (see formula below) on the pain scores adjusted for rescue medication use using the imputed values (see Section 9.1.1.1). AUC will start with the first pain assessment obtained after surgery and use all following pain assessments including those collected prior to rescue medication and unscheduled. Actual assessment times will be used in deriving AUC.

$$AUC = \left[\sum_{i=3}^{n} (p_i + p_{(i-1)})(t_i - t_{(i-1)})\right]/2$$

Where  $p_i$  is the VAS pain score at time i and  $t_i$  is the time, in hours, from end of surgery. Note that i starts at 3 since  $t_1$  is not used in AUC calculation (prior to surgery) and  $t_2$  is arrival at PACU.

# 9.7.1.5. Opioid Consumption

Opioids will be converted to IV morphine equivalent dose (MED mg) using the appropriate conversion factor from Table 3 for all summaries. Total opioid dose is the IV morphine equivalent sum of all opioids taken after surgery up to the timepoint of interest. Subjects with no opioid use during the period in question will be assigned a dose of 0 for summaries and changed


to the lesser of 0.1 or half of the smallest total amount observed in the study, whichever is smaller, prior to being transformed with the natural logarithm for analysis.

**Table 3: IV Morphine Equivalents** 

| Medication | Unit | Route | Conversion (Multiplication)<br>Factor |
|---|---|---|---|
| Oxycodone, Oxycocet, Percocet, acetaminophenoxycodone, Oxycontin | mg | PO,IV,IM,SC | 2 |
| Morphine | mg | IV,IM,SC | 1 |
| Morphine | mg | PO | 0.33 |
| Hydromorphone (Dilaudid), Hydromorphone hydrochloride | mg | IV,IM | 7.7 |
| Hydromorphone (Dilaudid), Hydromorphone hydrochloride | mg | РО | 1.3 |
| Hydromorphone (Dilaudid), Hydromorphone hydrochloride | mg | SC | 4 |
| Fentanyl | mg | IV,PO,IM | 100 |
| Vicodin, Norco, Lorcet, Lortab, hydrocodone-<br>acetaminophen | mg | РО | 2 |
| Codeine (Tylenol 3, acetaminophen-coedine,<br>Paracetamol Forte, Tylenol 4) | mg | РО | 0.05 |
| Ultram, Tramadol, Tramacol hydrochloride | mg | PO, IM | 0.08 |

PO = oral; IV = intravenous; VAS = visual analog scale.

**If other rescue medications are given then the conversion to IV Morphine Equivalent will be determined post-hoc.** If a combination opioid product is given then the IV Morphine Equivalent will be determined by the opioid part of the medication. Opioids given post surgically with an indication such as 'anesthesia maintenance' will not be included.

# 9.7.1.6. Time to First Opioid Rescue Medication Use

Time to first opioid rescue medication use will be calculated as the time from end of surgery to time of event in hours.

# 9.7.1.7. Pain-free

Pain-free is defined as an observed VAS score less than or equal to 1.5 with no prior rescue medication and all prior VAS scores less than or equal to 1.5.

# 9.7.1.8. Overall Benefit of Analgesia Score (OBAS)

The OBAS is derived as follows:

- 1. Add all of the scores of questions 1 to 6.
- 2. To this number, add four.
- 3. Subtract the score of question 7 from this number.

If a response is missing to any question in the OBAS, the total score will not be calculated.


# 9.7.2. Methods of Analysis

For Primary and Secondary Efficacy Analyses, descriptive statistics that are appropriate for the efficacy variable will also be shown by site but no statistical analyses will be performed within a site.

# 9.7.2.1. Primary Efficacy Analysis

The primary efficacy variable is the AUC of VAS scores through 72 hours [AUC(0-72)] using the multiple imputation method described in Section 9.1.1.1.

Tests for the treatment effect of EXPAREL versus placebo will be based on the following null hypothesis ( $H_0$ ) and two-sided alternative hypothesis ( $H_a$ ):

H<sub>o</sub>: 
$$\mu_s = \mu_p$$
 versus H<sub>a</sub>:  $\mu_s \neq \mu_p$ 

where  $\mu_{S}$  and  $\mu_{P}$  are the mean of AUC(0-72) for EXPAREL and the mean of AUC(0-72) for placebo, respectively. A two-sided test will be performed at 2.5% level of significance comparing each EXPAREL dose to placebo. The treatment effect of EXPAREL will be considered significantly better than that of placebo if the null hypothesis of no difference is rejected and a difference in mean of AUC(0-72) in favor of EXPAREL (mean for EXPAREL less than the mean for placebo) is observed.

For the primary efficacy variable of AUC(0-72), each EXPAREL dose will be compared to placebo using analysis of variance (ANOVA) with age, weight, and height as covariates. Based on the model, the LS mean, and the SE of the LS mean, will be reported for each treatment. The LS treatment difference for the active minus placebo, 95% CI for the active minus placebo treatment difference, and p-value will be reported as well as for each active treatment.

Descriptive statistics of the primary efficacy variable will also be shown by site but no statistical analyses will be performed within a site.

# 9.7.2.2. Secondary Efficacy Analyses

# 9.7.2.2.1. Postsurgical Opioid Consumption

Postsurgical narcotic consumption (MED mg) will be summarized (n, Geometric Mean, coefficient of variation, minimum, and maximum) by treatment group for the total dose consumed over the 72 hours after the end of surgery. The number and percentages of the types of opioids used will be presented by treatment group, subjects will be counted only once for each opioid used. This summary table will show summaries across all sites and for each site separately.

Prior to analysis, the natural logarithm transformation will be applied to the total opioid consumption amount. When total amount of opioids (IV Morphine Equivalent) used is 0, then the result will be changed to 0.1 or half of the smallest total amount observed in the study, whichever is smaller, prior to being transformed with the natural logarithm. To test for significant differences between EXPAREL and placebo, an ANOVA with age, weight, and height as covariates will be used. The LS means, LS mean difference between the two treatment groups, 95% CI for the LS mean difference between EXPAREL and placebo, and p-value will be reported. The LS means, LS mean differences and 95% CI will be back transformed for


presentation (note the LS mean difference becomes the ratio when back-transformed) along with the descriptive statistics (untransformed) by treatment.

### 9.7.2.2.2. Opioid-free

Percentage of opioid-free subjects through 72 hours will be analyzed using a Cochran-Mantel-Haenszel (CMH) test. The p-value from the CMH analysis and mean treatment difference and 95% CI about the mean difference derived using the Newcombe<sup>9</sup> method (SAS pseudo-code below) will be presented. The tabulation of opioid-free subjects will be presented across all sites and for each site separately. No inferential statistics will be calculated for individual sites.

The number and percentage of subjects opioid-free will also be tabulated by timepoint.

# Pseudo-code for Newcombe method:

PROC FREQ;

TABLE SITE\*TREATMENT\*RESPONSE / RISKDIFF(CL=NEWCOMBE COMMON);

RUN:

# 9.7.2.2.3. Time to First Opioid Rescue Medication

Time to first opioid rescue medication will be computed in hours as the date and time of the first opioid rescue medication minus the date and time of the end of surgery. If a subject is not administered an opioid rescue medication, the time to first administration will be censored at 72 hours after surgery or at the time of last follow-up, whichever is earliest. Time of last follow-up will be defined as the latter of (1) the last pain assessment, (2) the start time of the last concomitant medication, or (3) the start time of the last AE.

Time to first opioid rescue will be analyzed by the Kaplan-Meier method. The n (%) of subjects administered an opioid as well as the n (%) of censored observations will be presented for each treatment group. In addition, Kaplan-Meier estimates in terms of the median and its 95% CI, and the 25th and 75th percentiles will be presented for each treatment. Log-rank tests will be used to compare each EXPAREL dose to placebo.

#### 9.7.2.3. Tertiary Efficacy Analyses

P-values computed for the tertiary endpoints are for descriptive purposes only and are not adjusted for multiple comparisons.

# 9.7.2.3.1. Visual analog scale (VAS) AUC

Summary statistics will be presented by treatment for VAS AUC(0-12), VAS AUC(0-24), VAS AUC(0-48), VAS AUC(0-96), VAS AUC(24-48), VAS AUC(48-72) and VAS AUC(72-96). For each of these variables, each EXPAREL dose will be compared to placebo using analysis of variance (ANOVA) with age, weight, and height as covariates. Based on the model, the LS mean and SE of the LS mean will be reported for each treatment. The LS treatment difference for the active minus placebo, 95% CI for the active minus placebo treatment difference, and p-value will be reported as well as for each active treatment.

#### 9.7.2.3.2. Visual analog scale (VAS)

Summary statistics will be presented by treatment for VAS at each assessment timepoint. This summary will be based on the observed VAS values.


# 9.7.2.3.3. Proportion of Pain-Free Subjects

The proportion of pain-free subjects will be tabulated by treatment. The number and proportion of subjects who are pain-free and not pain-free (or VAS score is missing) will be presented at assessment timepoint. For the proportion of pain-free subjects, each EXPAREL dose will be compared to placebo using a Cochran-Mantel-Haenszel (CMH) test. The p-value from the CMH analysis and mean treatment difference and 95% CI about the mean difference derived using the Newcombe<sup>10</sup> method.

# 9.7.2.3.4. Sum of Pain Intensity Scores (SPIS)

Summary statistics will be presented by treatment for SPIS(0-12), SPIS(0-24), SPIS(0-48), SPIS(0-72), SPIS(0-96), SPIS(24-48), SPIS(48-72) and SPIS(72-96). For each of these variables, each EXPAREL dose will be compared to placebo using analysis of variance (ANOVA) with age, weight, and height as covariates. Based on the model, the LS mean and SE of the LS mean will be reported for each treatment. The LS treatment difference for the active minus placebo, 95% CI for the active minus placebo treatment difference, and p-value will be reported as well as for each active treatment.

# 9.7.2.3.5. Total Opioid Consumption through 24, 48 and 96 hours

Total opioid consumption through 24, 48, and 96 hours will each be summarized by treatment group. The summaries and analyses will be calculated similar as the postsurgical opioid consumption through the 72 hour secondary endpoint (see Section 9.7.2.2.1).

# 9.7.2.3.6. Total Opioid Consumption During Specific Time Intervals

Total opioid consumption from 24-48, 48-72 and 72-96 hours will be summarized by treatment group. The summaries and analyses will be calculated similar as the postsurgical opioid consumption through the 72 hour secondary endpoint (see Section 9.7.2.2.1).

# 9.7.2.3.7. Percentage of Opioid-free Subjects through 24, 48 and 96 hours

The percentage of opioid-free subjects at 24, 48, and 96 hours will be tabulated by treatment. The summaries and analyses of the percentage of opioid-free subjects at 24, 48, and 96 hours will be calculated similar as the percentage of opioid-free subjects at 72 hours secondary endpoint (see Section 9.7.2.2.2).

#### 9.7.2.3.8. Overall Benefit of Analgesia (OBAS)

The OBAS total score will be summarized by treatment and individual question responses tabulated at each assessment timepoint. For the OBAS total score, each EXPAREL dose will be compared separately to placebo using a Kruskal-Wallis test.

#### 9.7.2.3.9. Subject Satisfaction with Overall Analgesia

Subject satisfaction with overall analgesia (obtained using a 5-point Likert scale) will be summarized and individual responses tabulated by treatment for each assessment timepoint. The numeric value of the response will be presented using descriptive statistics. For each value of the scale the number and percentage of subjects selecting that value will also be presented. For the subject satisfaction with overall analgesia, each EXPAREL dose will be compared to placebo using a Kruskal-Wallis test.

# 9.7.2.3.10. Discharge Readiness


Time to discharge ready will be computed in hours as the date and time of subjects first meeting the discharge readiness criterion and time of the end of surgery. Time to discharge ready will be when the MPADSS criteria is met (total score of 9 or more) for discharge readiness or the time of discharge, whichever occurs first. If a subject has not met the discharge ready criteria prior to or at a given timepoint (12, 24, 36, 48, 60, 72, 84, 96 and 120 hours), then the time to discharge ready will be censored at the time of their last MPADSS assessment in the study or the specific assessment timepoint (12, 24, 36, 48, 60, 72, 84, 96 and 120 hours), whichever occurs sooner.

Time to discharge ready will be analyzed by the Kaplan-Meier method for each of the following assessment timepoints: 12, 24, 36, 48, 60, 72, 84, 96 and 120 hours. The n (%) of subjects administered an opioid as well as the n (%) of censored observations will be presented for each treatment group. In addition, Kaplan-Meier estimates in terms of the median and its 95% CI, and the 25th and 75th percentiles will be presented for each treatment at 12, 24, 36, 48, 60, 72, 84, 96 and 120 hours. Log-rank tests will be used to compare each EXPAREL dose to placebo at 12, 24, 36, 48, 60, 72, 84, 96 and 120 hours.

The number and percent of subjects meeting the discharge readiness criteria at 12, 24, 36, 48, 60, 72, 84, 96 and 120 hours will be summarized.

If a subject is discharge ready at an early timepoint, the subject will be considered discharge ready at all subsequent (future) timepoints. If a subject has a discharge readiness total score of less than 9 or if the total score is missing, the subject will be considered not discharge ready, unless they were previously considered discharge ready.

#### 9.7.2.3.11. Number of Pain-Related Visits/Phone Calls after Discharge

The number of pain-related unscheduled phone calls or office visits will be summarized (n, mean, SD, median, minimum, and maximum) by treatment group. The number and percentage of subjects reporting for each number of pain-related unscheduled phone calls or visits (0, 1, 2, ... maximum number observed) will be presented by treatment group. For the number of pain-related unscheduled phone calls or office visits, each EXPAREL dose will be compared to placebo using a Kruskal-Wallis test.

#### 9.7.2.3.12. Timed Walk Test

Subjects who did not perform the timed walk test will have a zero (0) imputed for distance walked in the analysis. The distance, in meters, covered during the timed walk test will be analyzed using a mixed model repeated measures (MMRM) analysis with fixed effects for treatment, site and time and a treatment-by-time interaction with subject within treatment as the random effect. The LS mean and SE of the LS mean will be reported for each treatment. The LS treatment difference for the active minus placebo, 95% CI for the active minus placebo treatment difference, and p-value will be reported as well as for each active treatment. Analyses will be performed on the efficacy and per-protocol analysis sets.

The MMRM will be fit with covariance matrices of UN (unstructured), CS (compound symmetry) and AR(1) (auto-regressive 1). The analysis with the lowest AIC criteria will be reported on the table. Other covariance matrix structures may be used if none of these converge.

The timed walk test summary will include tabulations of whether the test was performed and if not performed, reasons why not and the use of a walking aid (yes/no), level of physical assistance required, and descriptive statistics for the distance covered. Statistics overall sites,


pooled site(s) and site within pooled site will be presented. This summary will be provided for both the efficacy and per-protocol analysis set.

# 9.7.2.3.13. Timed Up-and-go Test (TUG)

Subjects who did not perform the timed walk test will have a zero (0) imputed for time in the analysis. The time, in seconds, to complete the TUG test will be analyzed using a mixed model repeated measures analysis with fixed effects for treatment, site and time and a treatment-by-time interaction with subject within treatment as the random effect. The LS mean, SE of the LS mean, LS treatment difference, 95% CI for the active minus placebo treatment difference and p-value will be reported as well as the treatment. Analyses will be performed on the efficacy and per-protocol analysis sets.

The MMRM will be fit with covariance matrices of UN, CS, and AR(1). The analysis with the lowest Akaike's information criterion (AIC) criteria will be reported on the table. Other covariance matrix structures may be used if none of these converge.

The TUG test summary will include tabulations of whether the test was performed and if not performed, reasons why not and the use of a walking aid (yes/no), level of physical assistance required, and descriptive statistics for the time to complete. Statistics for overall sites, pooled site(s) and site within pooled site will be presented. This summary will be provided for both the efficacy and per-protocol analysis set.

#### 9.7.2.3.14. Stair Climb Test

The stair climb test will be analyzed using a general mixed effect model with the logit link function and fixed effects for treatment, site and time with treatment-by-time interaction and subject within treatment as the repeated effect (PROC GENMOD; class ...; model ... / d=bin link=logit; LSMEANS ... /DIFF=CONTROL(...) CL alpha=0.05 ILINK EXP; repeated .../ type=...; run;). The odds ratio (each EXPAREL dose / Placebo) and its 95% CI and p-value will be reported as well as the odds ratio and its 95% CI at each testing timepoint as derived from the model. Analyses will be performed on the efficacy and per-protocol analysis sets. The number of subjects not completing and completing the test will be reported at each testing timepoint. This analysis will be provided for both the efficacy and per-protocol analysis set.

# 9.7.2.3.15. Region Analysis

Summaries and tabulations looking at region will be performed for the following:

- Disposition
- Demographics
- Baseline Characteristics
- Intraoperative medicines
- VAS AUC(0-72)
- Total opioid consumption through 72 hours
- Percentage opioid-free through 72 hours
- Sensation Loss and Return
- Motor Function Loss and Return
- Overall summary of adverse events
- Incidence of TEAEs
- Incidence of Serious TEAEs


The populations for each the summary and tabulation as planned for the non-region tables will be repeated for the region tables.

For analyses considering region, the age, weight, and height covariates will be replaced with region, this will be performed for the following:

- VAS AUC(0-72)
- Total opioid consumption through 72 hours
- Percentage opioid-free through 72 hours
- Sensation Loss and Return
- Motor Function Loss and Return

Region summaries, tabulations, and analyses will be the final block within the 14.1, 14.2 and 14.3 series of tables.

# 9.8. Safety Analyses

Safety assessments in this study consist of vital signs, 12-lead ECGs, neurological assessments, sensory and motor nerve block assessments, motor function assessments, and AEs. Vital signs, ECGs, neurological, nerve block assessments (sensory and motor), and motor function assessments will be serially collected (see Time and Events Schedule of Study Procedures). Adverse events will be collected from the time of informed consent through Day 30.

P-values computed for the safety endpoints are for descriptive purposes only and are not adjusted for multiple comparisons.

# 9.8.1. Vital Signs

Vitals signs are resting heart rate (bpm), systolic blood pressure (mmHg), and diastolic blood pressure (mmHg). Vital signs will be summarized by treatment group and the All EXPAREL group at each assessment timepoint. Summaries will present both actual and change-from-baseline results. Baseline statistics will be presented at each assessment timepoint for those subjects reporting data at that timepoint.

Vital signs will also be assessed for potentially clinically significant abnormal values (see Table 4). The number and percentage of subjects satisfying the potentially clinically significant abnormal criteria (critical value, critical change separately and then value and change concurrently) at any time during the study and at each assessment timepoint will be tabulated by treatment and overall treatments.

Table 4: Criteria for Potentially Clinically Significant Abnormal Vital Signs

| | , | | 1 |
|---|---|---|---|
| Vital Sign | Unit | Critical Value | Critical Change <sup>1</sup> |
| Resting Heart Rate | beats/minute (bpm) | High: ≥ 120 | Increase of at least 15 |
| | | Low: ≤ 50 | Decrease of at least 15 |
| Systolic Blood Pressure | mmHg | High: ≥ 180 | Increase of at least 20 |
| | | Low: ≤ 90 | Decrease of at least 20 |
| Diastolic Blood Pressure | mmHg | High: ≥ 105 | Increase of at least 15 |
| | | Low: ≤ 50 | Decrease of at least 15 |

<sup>&</sup>lt;sup>1</sup>Change criteria not applicable at baseline or screening.

# 9.8.2. Electrocardiograms


Investigators will classify ECG tracings as 'normal, 'abnormal not clinically significant' or 'abnormal clinically significant'. The investigator classifications will be tabulated by treatment and overall treatments at any time during the study and each assessment timepoint.

A shift table comparing the investigator classification of the ECG results at baseline to each timepoint will also be provided.

#### 9.8.3. Neurological Assessments

Neurological assessments include orientation (orientated, disoriented, not assessable), numbness (of lips, tongue, or around mouth), metallic taste, hearing problems, vision problems, and muscle twitching. The number and percentage of subjects will be tabulated for each neurological assessment by treatment group at any time after baseline and at each assessment timepoint.

#### 9.8.4. Sensation Tests

Sensations tests are assessed on the thigh (anterior cutaneous nerve) and foot (saphenous nerve).

The number and percentage of subjects will be tabulated for each response (present/absent) within each nerve and sensory test (cold, pinprick and light touch) by treatment group at each assessment timepoint.

The number and percentage of subjects will be tabulated for loss and return of sensation (see Section 7) across all locations and within each location (thigh and foot) and each sensory test (cold, pinprick and light touch) and combinations of sensory tests (ANY, CPL, CP, CL, and PL) by treatment group at each assessment timepoint. Where the combinations of ANY, CPL, CP, CL and PL are defined as follows:

- ANY = at least one sensation
- CPL = all sensations (cold, pinprick and light touch)
- CP = cold and pinprick
- CL = cold and light touch
- PL = pinprick and light touch

A subject will be considered as having a loss of sensation if either of the locations has a loss of sensation; a return of sensation is when both locations have sensation for the subject.

The times to first loss of, last loss of, first return of sensation, and last return of sensation (see Section 7 subsection loss of sensation and return of sensation) will be summarized by the Kaplan-Meier method. The n (%) of subjects administered an opioid as well as the n (%) of censored observations will be presented for each treatment group. In addition, Kaplan-Meier estimates in terms of the median and its 95% CI (using log-log method), and the 25th and 75th percentiles will be presented for each treatment. Log-rank tests will be used to compare each EXPAREL dose to placebo. This analysis will be performed across locations and within each location.

Duration of sensation loss will be summarized across locations and within each location. Total duration is defined as the sum of durations of each lost-return cycle for a subject. If more than 10% of the subjects in at least one treatment group experience multiple lost-return cycles, then duration will be summarized for total duration and within each cycle.


An additional table summarizing the number of cycles and tabulating the distribution number of cycles by treatment group will be presented within each location by treatment group.

# 9.8.5. Degree of motor nerve block Assessments

Degree of motor nerve block assessments includes active and passive flexion and extension. The actual and change from baseline values for each of these parameters will be summarized by treatment at each assessment timepoint. At each assessment timepoint the baseline values will be summarized for those subjects who have data at that timepoint.

At each assessment timepoint, the number and percent of subjects with loss and return of motor function (see Section 7) will be summarized by treatment.

For each active assessment the time to return to motor function will be analyzed by treatment in the same manner as time to first rescue medication (see Section 9.7.1.6).

#### 9.8.6. Adverse Events

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

An AE will be considered TEAE if the onset date and time is between the start date and time of study treatment and Day 30.

If an AE has a partial onset date and time the imputed start and stop dates and times will be used to determine treatment-emergence (e.g., stop date and time is before start date and time of study treatment). All AE summaries will present TEAEs only; AEs that are not treatment-emergent will be included in listings but not summarized.

The incidence of subjects reporting TEAEs will be tabulated by the number and percentage of subjects reporting the TEAE. Incidence is defined as a subject reporting at least one TEAE within the summary level. Summary levels are 'at least one TEAE', system organ class and preferred term. Subjects will be counted only once within each reporting level on the table. For example if a subject reports a TEAE of headache on two separate occasions, the subject will be counted only once in the headache row of the table. Similarly if a subject reports two separate TEAEs within the same system organ class the subject will only be counted once in the summary row for that system organ class. A summary of subjects reporting at least one TEAE during the study will also be presented.

The first row on every TEAE table will be the number and percentage of subjects reporting at least one TEAE. Subsequent rows will be presented in descending order of subject counts for the overall treatment group with the most common system organ class first, followed within each system organ class by the preferred terms in descending subject count order. For tables presenting the severity or relation to study treatment of AE, the sort order will be determined by the number and percentage of subjects reporting the preferred term, thus the sort order of rows will remain the same for the relation or severity tables as the tables by preferred term.

The following summaries will be presented for the AEs reported by the subjects:

An overview of all TEAEs, serious TEAEs and TEAEs of Special Interest will present the number and percentage of subjects in the following categories:

• Any TEAE


- o Maximum severity: Mild
- o Maximum severity: Moderate
- o Maximum severity: Severe
- At least one related TEAE
- At least one serious TEAE
- Subjects discontinued due to a TEAE
- Died on study

Subjects will be counted once in each of the above categories except for maximum severity. Subjects will be counted only once at the highest severity reported. For example, if a subject has a mild and severe headache and a moderate rash, the subject will be counted under maximum severity of severe only.

Adverse event tables will present the data by treatment group and across all treatment groups. Incidence tables will be created for the following groups of TEAEs:

- All TEAEs
- Study treatment related TEAEs
- TEAEs leading to study withdrawal
- Study treatment related TEAEs leading to study withdrawal
- All TEAEs by severity
- All TEAEs by relationship to study treatment
- All serious TEAEs
- Study treatment related serious TEAEs
- Serious TEAEs leading to study withdrawal
- Study treatment related serious TEAEs leading to study withdrawal
- Serious TEAEs resulting in death
- Study treatment related serious TEAEs resulting in death
- All TEAEs of special interest
- Study treatment related TEAEs of special interest
- TEAEs of special interest leading to study withdrawal
- Study treatment related TEAEs of special interest leading to study withdrawal
- TEAEs of special interest resulting in death
- Study treatment related TEAEs of special interest resulting in death

If there are no AEs to report on any of the above tables, the table should be created with the line 'no adverse events were reported' in the body of the table.

Adverse events will be considered related if the investigator assessment of relationship to study treatment is either 'possible', 'probable' or 'definite'.

All AE summaries based on related AEs will be produced based on the investigator assessment of relatedness. Below are the MedDRA terms for the adverse events of special interest:

| | | MedDRA 18.1 Dictionary Terms | |
|---|---|---|---|
| Group | Protocol term | Term Level Term | |
| Cardiac | Angina | Preferred term | Angina Pectoris |
| Cardiac | Myocardial infarction | Preferred term | Myocardial Infarction |


| | Bradycardia | Preferred term | Bradycardia |
|---|---|---|---|
| | Tachycardia | Preferred term | Tachycardia |
| | Extrasystoles | Preferred term | Extrasystoles |
| | Shortness of breath requiring intervention | Preferred term | Dyspnoea |
| | Altered mental status | Preferred term | Mental Status Changes |
| | Altered sensorium | Preferred term | Depressed level of consciousness |
| | Rigidity | Preferred term | Muscle Rigidity |
| | Dysarthria | Preferred term | Dysarthria |
| | Seizure | Preferred term | Seizure |
| | Tremors | Preferred term | Tremor |
| | Metallic taste | Preferred term | Dysgeusia |
| Neurologic | Tinnitus | Preferred term | Tinnitus |
| | Perioral numbness | Preferred term | Hypoaesthesia Oral |
| | Visual disturbance | Preferred term | Visual Impairment |
| | Dizziness | Preferred term | Dizziness |
| | Hyperesthesia | Preferred term | Hyperaesthesia |
| | Muscular twitching* | Preferred term | Muscle Twitching |
| | Tingling* | Preferred term | Paraesthesia |
| | Paresthesia* | Preferred term | Paraesthesia |
| Other | Fall | Preferred term | Fall |
| * if event pe | * if event persists beyond or occurs after 72 hours after start of study treatment dose. | | |

A listing of the mapping of the system organ class and preferred terms to verbatim terms will be presented.

#### 9.8.7. Laboratory Parameters

Clinical laboratory assessments are collected at screening, baseline and Day 10. Laboratory results will be summarized by treatment group and the All EXPAREL group at each assessment timepoint. Summaries will present both actual and change-from-baseline results. Baseline statistics will be presented at each assessment timepoint for those subjects reporting data at that timepoint.

Tabulations of the number and percentage of subjects with value below normal, normal or above normal will be provided by treatment group, All EXPAREL group and across all treatment groups at each timepoint.

Shifts in laboratory results categorized as low (below the lower limit of the normal range), normal (within the normal range, limits inclusive) and above (above the upper limit of the normal range) will be presented in shift tables with baseline categories across the columns and Day 10 down the rows for EXPAREL 133 mg, EXPAREL 266 mg, All EXPAREL and placebo separately. Each cell will present the number and percentage of subjects in that cell. Due to the width of these tables, only 2 treatments can be presented on a page. For ease of comparing active treatments to placebo, placebo data will be presented on each page. Thus the shift table will present all laboratory data for EXPAREL 133 mg and placebo then for EXPAREL 266 mg and placebo and finally for All EXPAREL and placebo.

#### 9.9. Pharmacokinetic Analysis

The analysis of the PK endpoints will be described in a separate document.

#### 9.10. Interim Analysis

#### 9.10.1. Pharmacokinetic Review


An interim PK analysis was completed by QuantPharm LLC after 30 subjects completed the assessments through post-surgical Day 10. All of the plasma samples from the subjects who received EXPAREL were analyzed and the plasma samples from the subjects randomized to placebo were analyzed through the 24-hour timepoint. Enrollment continued while the interim PK data were analyzed. The goal of this blinded analysis was to determine the appropriateness of the PK timepoints selected and make recommendations to keep, remove, or revise them in order to fully characterize the PK profile.

QuantPharm LLC indicated that the results of this analysis showed a median  $T_{max}$  of 60 hours for the 133 mg EXPAREL group and a median  $T_{max}$  of 78 hours for the 266 mg EXPAREL group. This information informed the changes to the PK collection schedule contained protocol amendment 2.

In addition, the safety assessment timepoints, including the neurological exam, vital signs, and ECG were adjusted based on the initial interim PK data.

# 9.11. Significance Testing

Significance testing will be based on "Graphical approaches for multiple comparison procedures using weighted Bonferroni, Simes, or parametric tests" (Bretz 2011). The initial alpha will be set to a two-sided 0.025 for each of the primary efficacy analyses. Subsequent testing will be conducted following the ideas of the paper.

In addition to the primary endpoint (VAS AUC) there are three key secondary endpoints (total opioid consumption, percentage of opioid-free subjects, and time to first rescue medication), and for each of these four endpoints there are two primary pairwise comparisons. The procedure for multiplicity adjustment for these eight comparisons is described below, together with demonstration that it provides strong control of the type 1 error.

Let  $H_{PrimLD}$ ,  $H_{Sec1LD}$ ,  $H_{Sec2LD}$ , and  $H_{Sec3LD}$  represent the null hypotheses for the comparison of EXPAREL 133 mg versus Placebo. Likewise let  $H_{PrimHD}$ ,  $H_{Sec1HD}$ ,  $H_{Sec2HD}$ , and  $H_{Sec3HD}$  represent the null hypotheses for the comparison of EXPAREL 266 mg versus Placebo. Where  $H_{PrimLD}$ ,  $H_{Sec1LD}$ ,  $H_{Sec2LD}$ , and  $H_{Sec3LD}$  are respectively VAS AUC, total opioid consumption, percentage of opioid-free subjects, and time to first rescue medication and similarly for  $H_{PrimHD}$ ,  $H_{Sec1HD}$ ,  $H_{Sec2HD}$ , and  $H_{Sec3HD}$ .

The first stage of the multiplicity adjustment will be carried out using a graphical approach to sequentially rejective multiple test procedures (Bretz et al, 2009). This will be applied to the set of the four null hypotheses  $F = \{H_{PrimLD}, H_{PrimHD}, H_{Sec1LD}, H_{Sec1LD}\}$  corresponding to the primary endpoint and the first key secondary endpoint (total post-surgical opioid consumption through 48 hours). Let  $F_L = \{H_{PrimLD}, H_{Sec1LD}\}$  and  $F_H = \{H_{PrimHD}, H_{Sec1HD}\}$  denote the families of null hypotheses corresponding to comparisons of EXPAREL 133 mg versus Placebo, and EXPAREL 266 mg versus Placebo, respectively. The particular graphical procedure used here initially assigns  $\alpha = 0.0250$  two-sided for testing of the first member of each family (corresponding to the primary endpoint) and then within each family the two endpoints are tested in a fixed sequence. If for either family null hypotheses for both endpoints can be rejected, then the fixed sequence for the other dose level can be conducted using  $\alpha = 0.05$  two-sided. This procedure can be viewed as a Bonferroni-Holm-type approach applied to the families  $F_L$  and  $F_H$ . This procedure can be depicted graphically for  $F = \{H_{PrimLD}, H_{PrimHD}, H_{Sec1LD}, H_{Sec1LD}\}$  as follows:



With  $F = \{H_{PrimLD}, H_{PrimHD}, H_{Sec1LD}, H_{Sec1HD}\}$  as above, in the notation of Bretz et al (2009), we start with  $\alpha = (0.0250, 0.0250, 0, 0)$ . A **G** matrix with elements  $g_{ij}$  is defined in that paper to denote the fraction of the local level  $\alpha_i$  that is allocated to null hypothesis j from set F in the case that null hypothesis i is rejected. This 4x4 matrix **G** takes a simple form in the procedure considered here because  $g_{I3} = g_{24} = g_{32} = g_{4I} = 1$ , but all other elements are zero. Bretz et al (2009) provides an updating procedure for the matrix **G** as successive null hypotheses are rejected, and prove that such procedures provide strong control of the type 1 error. The particular procedure used in the current study implements the updating of  $\alpha$  and **G** in accordance with Bretz et al's (2009) "Algorithm 1." Further, the regularity conditions  $0 \le g_{ij} \le 1$ ,  $g_{ii} = 0$ , and

 $\sum_{k=1}^{4} g_{ik} \le 1$  for all i, j = 1,...4, specified in equation (1) of that paper, are satisfied, and so strong

control of type 1 error at  $\alpha = 0.05$  two-sided for testing of the four null hypotheses  $F = \{H_{PrimLD}, H_{PrimHD}, H_{Sec1LD}, H_{Sec1HD}\}$  follows from Bretz et al's proof.

The particular procedure used for the current trial is also given as an example to illustrate the graphical procedure within both Alosh et al (2014) and Bretz et al (2011).

The second stage of the multiplicity adjustment procedure relates to  $S = \{H_{Sec2HD}, H_{Sec2LD}, H_{Sec3HD}\}$ , ie, the four null hypotheses related to the second key efficacy parameter (percentage of opioid-free subjects through 48 hours) and the third key efficacy parameter (time to first opioid rescue through 48 hours). These are only tested if all 4 null hypotheses from set F have already been rejected, and in that case  $H_{Sec2HD}$ ,  $H_{Sec3HD}$ , and  $H_{Sec3LD}$  are then tested sequentially in turn at  $\alpha = 0.05$  two-sided, where statistical significance is required for all preceding tests within set S as well as statistical significance for all tests from set F. If the required preceding null hypotheses have not been rejected then p-values for later tests in this sequence will be viewed only as descriptive and not as hypothesis testing.

Given that: (i) strong control of type 1 error at  $\alpha = 0.05$  two-sided has been demonstrated for testing of the four null hypotheses F; (ii) testing only proceeds to set S if all null hypotheses in set F have been rejected; and (iii) the null hypotheses within set S are tested in a single step-down procedure, the above procedure has strong control of type 1 error at  $\alpha = 0.05$  two-sided for testing of all eight null hypotheses.


# 10. SAMPLE SIZE CALCULATIONS

Under Amendments 1 and 2 a study population of approximately 300 subjects was planned with approximately 100 subjects in each treatment group (EXPAREL 133 mg, EXPAREL 266 mg and placebo). The sample size was estimated based on the results of a Phase 3 TKA study of EXPAREL versus placebo where the mean (SD) AUC of the NRS-R pain intensity scores through 72 hours was 420 (169) and 514 (160) for the EXPAREL and placebo groups, respectively. Assuming a 2.5% two-sided alpha, common SD of 170 and a 5% drop-out rate, a sample size of 85 subjects per arm will have at least 90% power to detect a difference of 100 in at least one of the active treatment arms.

Under Amendment 3 the sample size was estimate was revised by changing the power from 90% to 80% and the drop-out rate was reduced from 5% to 3%; no other assumptions were changed in the derivation of the sample size. Thus the sample size, under Amendment 3, was estimated based on the results of a Phase-3 study of EXPAREL versus placebo in patients undergoing TKA where the means (standard deviation [SD]) AUC of the NRS-R pain intensity scores through 72 hours were 420 (169) and 514 (160) for the EXPAREL and placebo groups, respectively. Assuming a 2.5% two-sided alpha, common SD of 170 and a 3% drop-out rate, a sample size of 77 subjects per treatment group will have at least 80% power to detect a difference of 100 in at least one of the active treatment groups. Approximately 231 subjects (77 subjects per treatment group) are planned for enrollment in this study in order to have at least 225 evaluable subjects.

# 11. REFERENCES

<sup>1</sup> American Statistical Association. Ethical Guidelines for Statistical Practice. Prepared by the Committee on

7 Rubin DB, Schenker N. Multiple imputation for interval estimation from simple random samples with ignorable nonresponse. J Am Stat Assoc 1986;81:366-374.


American Statistical Association. Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, 07 August 1999. http://www.amstat.org/profession/ethicalstatistics.html

<sup>&</sup>lt;sup>2</sup> US Federal Register. International Conference on Harmonisation; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. 16 September 1998.

<sup>&</sup>lt;sup>3</sup> Royal Statistical Society. The Royal Statistical Society: Code of Conduct, August 1993. http://www.rss.org.uk/about/conduct.html.

<sup>&</sup>lt;sup>4</sup> Rubin, D. B. (1987). Multiple Imputation for Nonresponse in Surveys. New York: John Wiley & Sons.

<sup>&</sup>lt;sup>5</sup> The National Academies Press. The Prevention and Treatment of Missing Data in Clinical Trials, prepared by the Panel on Handling Missing Data in Clinical Trials and Committee on National Statistics, 2010.

<sup>&</sup>lt;sup>6</sup> Schafer, J. L. (1997). Analysis of Incomplete Multivariate Data. New York: Chapman & Hall.

<sup>&</sup>lt;sup>8</sup> Bretz F, Posch M, Glimm E, et al. Graphical approaches for multiple comparison procedures using weighted Bonferroni, Simes, or parametric tests. Biom J. 2011;53(6): 894–913.

<sup>&</sup>lt;sup>9</sup> Newcombe RG, Interval Estimation for the Difference between Independent Proportions: Comparison of Eleven Methods. Statist. Med. 17, 873-890 (1998).

<sup>&</sup>lt;sup>10</sup>Bretz, F., Maurer, W., Brannath, W. and Posch, M. (2009). A graphical approach to sequentially rejective multiple test procedures. Statistics in Medicine 28, 586–604.

<sup>&</sup>lt;sup>11</sup>Alosh, M., Bretz, F., and Huque, M. (2014) Advanced multiplicity adjustment methods in clinical trials. Statistics in Medicine 33(4), 693-713.

# 12. TIME AND EVENTS SCHEDULE OF STUDY PROCEDURES

Please see the Protocol for the full "Time and Events Schedule of Study Procedures". Note that the study days defined in the table and footnotes start with surgery as Day 0 for the Protocol "Time and Events Schedule of Study Procedures"; however, the SAP definitions start with surgery as Day 1. The SAP follows the CDISC convention to define study day. Thus in the SAP preop Day 0 is Day 1, Day 7 is Day 8, Day 10 is Day 11 and Day 29 is Day 30.

## 13. MULTIPLE IMPUTATION EXAMPLE PROGRAM CODE

```
** Note: INPUT DATA is the dataset that contains the VAS data with the wWOCF imputation performed
** Step 1 use Markov-Chain Monte-Carlo (MCMC) method **;
** Note the value for the random seed is fixed to be 123 so that the results are reproducible
proc mi data= INPUT DATA seed=123 nimpute=10 out= OUTPUT STEP1 minimum=0 maximum=10;
    by TRT01P;
    mcmc impute=monotone nbiter=2000 niter=1000;
    var aval atptn;
run; quit;
*** Step 2 derive endpoint using appropriate techniques from INPUT DATA to create INPUT DATA2**;
*** Step 3 analyze imputations
DATA &a;
       set INPUT DATA2;
       if param = &select and efffl = 'Y' and trt01pn ne 2;
run; quit;
proc sort data=&a; by IMPUTATION; run; quit;
PROC MIXED DATA= &a METHOD=TYPE3;
       by _IMPUTATION_;
       class TRT01P:
       model AVAL = TRT01P AGE WEIGHT HEIGHT;
       Ismeans TRT01P/ diff= CONTROL('Placebo') CL:
       ods output LSMeans = &b;
       ods output diffs = &c;
run; quit;
proc sort data= &b; by TRT01P; run;
PROC MIANALYZE DATA=&b ALPHA=0.05 THETA0=0;
       by TRT01P;
       modeleffects ESTIMATE;
       stderr STDERR;
       ods output PARAMETERESTIMATES=&d;
run; quit;
** Step 4 build report
```

# LAYOUT OF TABLES, LISTINGS AND FIGURES

The following are planned summary tables. Tables will be numbered according to the nomenclature used to support the CSR. The final table numbering may be different from the SAP. No amendment will be made for changes in table numbering. All headers, titles,

footnotes, and footers specified in the table mock-ups will be displayed in the produced output unless otherwise specified. Notes to programmers will not be included in the tables.

Tables and listings will have 10 point font size. Listings font size may be reduced to 9 point if needed. The TLFs will have either Times New Roman, Courier New or SAS Monospace type face. All final TLFs will be provided in both PDF and Word (or RTF) file formats.

Percentages should not appear if the count is zero.

Italicized text in the TLF mock-ups indicate notes to programmers and is not to appear on any TLF.

Note headers and footers on mock-ups are reflective of the SAP document and are not intended to appear on the TLFs.

Titles on the TLFs in the mock-ups are presented left-justified as a single line of text. However, the presentation for final TFLs should be center-justified with the TLF number on one line and the remaining titles on multiple lines of text where the line breaks are delimited by hyphens (-) in the TLF mock-ups titles. For example, for Table 14.2-1.1.1 the title in the mock-up appears as:

```
Table 14.2-1.1.1: Analysis of AUC of VAS Pain Intensity Scores through 72 hours - Efficacy Analysis Set - Multiple Imputation Results
```

but should appear as follows on the final TLF:

```
Table 14.2-1.1.1

Analysis of AUC of VAS Pain Intensity Scores through 72 hours

Efficacy Analysis Set

Multiple Imputation Results
```

The title format in the mock-ups is due to limitations of MSWord. The mock-up format enables MSWord to generate a table of contents for the mock-ups.

On all listings the treatments, in order of appearance, are: EXPAREL 133 mg, EXPAREL 266 mg, PLACEBO and, if applicable, NOT RANDOMIZED. Always insert a page break between treatments.

On all listings sort within treatment by site, subject, with further sorts dependent on listing.

Table and listing shells follow.

For categorical variables, if subjects are missing data for a certain category (example Race), a missing subcategory should be added under the respective category.

CONFIDENTIAL 42 of 173 20Jun 2017

| 14. | TABLE | OF | CONTENTS | FOR TABLE MOCK | <b>C-UPS</b> |
|-----|-------|-----------|----------|----------------|--------------|
| 17. | | <b>\/</b> | | | |

| TABLE 14.1-1: SUMMARY OF SUBJECT DISPOSITION – ALL SCREENED SUBJECTS | 49 |
|---|---|
| TABLE 14.1-2.1.1: SUMMARY OF SUBJECT DEMOGRAPHICS - SAFETY ANALYSIS SET | 51 |
| TABLE 14.1-2.1.2: SUBJECT DEMOGRAPHICS – EFFICACY ANALYSIS SET | 52 |
| TABLE 14.1-2.1.3: SUBJECT DEMOGRAPHICS – PER-PROTOCOL ANALYSIS SET | 52 |
| TABLE 14.1-2.2.1: SUMMARY OF SUBJECT BASELINE CHARACTERISTICS - SAFETY ANALYSIS SET | 53 |
| TABLE 14.1-2.2.2: SUBJECT BASELINE CHARACTERISTICS – EFFICACY ANALYSIS SET | 57 |
| TABLE 14.1-2.2.3: SUBJECT BASELINE CHARACTERISTICS – PER-PROTOCOL ANALYSIS SE | T57 |
| TABLE 14.1-3.1: SUMMARY OF SURGERY CHARACTERISTICS - SAFETY ANALYSIS SET | 58 |
| TABLE 14.1-3.2: SUMMARY OF SURGERY CHARACTERISTICS – EFFICACY ANALYSIS SET | 59 |
| TABLE 14.1-3.3: SUMMARY OF SURGERY CHARACTERISTICS – PER-PROTOCOL ANALYSIS SET | S<br>59 |
| TABLE 14.1-4.1: INCIDENCE OF INTRAOPERATIVE MEDICATIONS - SAFETY ANALYSIS SET | Γ60 |
| TABLE 14.1-4.2: INCIDENCE OF INTRAOPERATIVE MEDICATIONS - EFFICACY ANALYSIS SET | 60 |
| TABLE 14.1-4.3: INCIDENCE OF INTRAOPERATIVE MEDICATIONS – PER-PROTOCOL ANALYSIS SET | 60 |
| TABLE 14.1-5.1: SUMMARY OF SUBJECT DISPOSITION – BY REGION – ALL SCREENED SUBJECTS | 61 |
| TABLE 14.1-5.2.1.1: SUMMARY OF SUBJECT DEMOGRAPHICS – BY REGION - SAFETY ANALYSIS SET | 61 |
| TABLE 14.1-5.2.1.3: SUBJECT DEMOGRAPHICS – BY REGION – PER-PROTOCOL ANALYSIS SET | 61 |
| TABLE 14.1-5.2.2.1: SUMMARY OF SUBJECT BASELINE CHARACTERISTICS – BY REGION - SAFETY ANALYSIS SET | 61 |
| TABLE 14.1-5.2.2.2: SUBJECT BASELINE CHARACTERISTICS – BY REGION – EFFICACY ANALYSIS SET | 61 |
| TABLE 14.1-5.2.2.3: SUBJECT BASELINE CHARACTERISTICS – BY REGION – PER-PROTOCO ANALYSIS SET | L<br>61 |
| TABLE 14.1-5.3.1: SUMMARY OF SURGERY CHARACTERISTICS – BY REGION - SAFETY ANALYSIS SET | 61 |
| TABLE 14.1-5.3.2: SUMMARY OF SURGERY CHARACTERISTICS – BY REGION – EFFICACY ANALYSIS SET | 61 |
| TABLE 14.1-5.3.3: SUMMARY OF SURGERY CHARACTERISTICS – BY REGION – PER-PROTOCOL ANALYSIS SET | 61 |
| TABLE 14.2-1.1.1: ANALYSIS OF AUC OF VAS PAIN INTENSITY SCORES THROUGH 72 HOU – EFFICACY ANALYSIS SET - MULTIPLE IMPUTATION RESULTS | RS<br>62 |
| TABLE 14.2-1.1.2: SUMMARY OF AUC OF VAS PAIN INTENSITY SCORES THROUGH 72<br>HOURS BY SITE – EFFICACY ANALYSIS SET - MULTIPLE IMPUTATION<br>RESULTS | 63 |


| TABLE 14.2 | 2-1.2.1: ANALYSIS OF AUC OF VAS PAIN INTENSITY SCORES THROUGH 72 HOUR<br>– PER-PROTOCOL ANALYSIS SET - MULTIPLE IMPUTATION RESULTS | S<br>65 |
|---|---|---|
| TABLE 14.2 | 2-1.2.2: SUMMARY OF AUC OF VAS PAIN INTENSITY SCORES THROUGH 72<br>HOURS BY SITE – PER-PROTOCOL ANALYSIS SET - MULTIPLE IMPUTATION<br>RESULTS | 65 |
| TABLE 14.2 | 2-2.1.1: ANALYSIS OF POSTSURGICAL TOTAL OPIOID CONSUMPTION (MED MG)<br>THROUGH 72 HOURS – EFFICACY ANALYSIS SET | 66 |
| TABLE 14.2 | 2-2.1.2: SUMMARY OF TOTAL OPIOID CONSUMPTION (MED MG) THROUGH 72<br>HOURS BY SITE - EFFICACY ANALYSIS SET | 67 |
| TABLE 14.2 | 2-2.1.3: ANALYSIS OF TOTAL OPIOID CONSUMPTION (MED MG) BY TIME PERIOD - EFFICACY ANALYSIS SET | )<br>68 |
| TABLE 14.2 | 2-2.1.4: SUMMARY OF THE NUMBER OF TIMES OPIOID (RESCUE) MEDICATION WAS USED BY SUBJECT - EFFICACY ANALYSIS SET | <b>7</b> 0 |
| TABLE 14.2 | 2-2.2.1: ANALYSIS OF POSTSURGICAL TOTAL OPIOID CONSUMPTION (MED MG)<br>THROUGH 72 HOURS – PER-PROTOCOL ANALYSIS SET | 71 |
| TABLE 14.2 | 2-2.2.2: SUMMARY OF TOTAL OPIOID CONSUMPTION (MED MG) THROUGH 72 HOURS BY SITE - PER-PROTOCOL ANALYSIS SET | 71 |
| TABLE 14.2 | 2-2.2.3: ANALYSIS OF TOTAL OPIOID CONSUMPTION (MED MG) BY TIME PERIOD - PER-PROTOCOL ANALYSIS SET | )<br>71 |
| TABLE 14.2 | 2-2.2.4: SUMMARY OF THE NUMBER OF TIMES OPIOID (RESCUE) MEDICATION WAS USED BY SUBJECT - PER-PROTOCOL ANALYSIS SET | 71 |
| TABLE 14.2 | 2-3.1.1: ANALYSIS OF OPIOID-FREE SUBJECTS THROUGH 72 HOURS - EFFICACY ANALYSIS SET | 72 |
| TABLE 14.2 | 2-3.1.2: SUMMARY OF OPIOID-FREE SUBJECTS THROUGH 72 HOURS BY SITE - EFFICACY ANALYSIS SET | 73 |
| TABLE 14.2 | 2-3.2.1: ANALYSIS OF OPIOID-FREE SUBJECTS THROUGH 72 HOURS -<br>PER-PROTOCOL ANALYSIS SET | 74 |
| TABLE 14.2 | 2-3.2.2: SUMMARY OF OPIOID-FREE SUBJECTS THROUGH 72 HOURS BY SITE -<br>PER-PROTOCOL ANALYSIS SET | 74 |
| TABLE 14.2 | 2-4.1: ANALYSIS OF TIME TO FIRST RESCUE MEDICATION USE (HOURS) - EFFICACY ANALYSIS SET | 75 |
| TABLE 14.2 | 2-5.1: SUMMARY OF VAS AUC AT VARIOUS TIME INTERVALS - EFFICACY ANALYSIS SET | 76 |
| TABLE 14.2 | 2-5.2: SUMMARY OF VAS AT ASSESSMENT TIMEPOINTS - EFFICACY ANALYSIS SET | <b>7</b> 8 |
| TABLE 14.2 | 2-5.3: SUMMARY OF VAS SPIS AT VARIOUS TIME INTERVALS - EFFICACY ANALYSIS SET | <b>7</b> 9 |
| TABLE 14.2 | 2-6: ANALYSIS OF PAIN-FREE SUBJECTS AT ASSESSMENT TIMEPOINTS -<br>EFFICACY ANALYSIS SET | 80 |
| TABLE 14.2 | 2-7: ANALYSIS OF OPIOID-FREE SUBJECTS THROUGH 24, 48, AND 96 HOURS - EFFICACY ANALYSIS SET | 81 |
| TABLE 14.2 | 2-8: SUMMARY OF OVERALL BENEFIT OF ANALGESIA SCALE BY TIMEPOINT AND QUESTION - EFFICACY ANALYSIS SET | 82 |
| TABLE 14.2 | 2-9: SUMMARY OF SATISFACTION WITH POSTSURGICAL PAIN CONTROL<br>OUESTIONNAIRE SCORE BY TIMEPOINT - EFFICACY ANALYSIS SET | 84 |


| TABLE 14.2-10.1: SUMMARY OF TIME TO DISCHARGE READY - EFFICACY ANALYSIS SET | 85 |
|---|---|
| TABLE 14.2-10.2: SUMMARY OF DISCHARGE READY BY ASSESSMENT - EFFICACY ANALYSIS SET | 86 |
| TABLE 14.2-11: SUMMARY OF NUMBER OF UNSCHEDULED PHONE CALLS OR OFFICE VISITS RELATED TO PAIN - EFFICACY ANALYSIS SET | 87 |
| TABLE 14.2-12.1: ANALYSIS OF DISTANCE WALKED (METERS) DURING TIMED WALK TES – EFFICACY ANALYSIS SET | 88 |
| TABLE 14.2-12.2: SUMMARY OF TIMED WALK TEST BY TIMEPOINT – EFFICACY ANALYSIS SET | S<br>90 |
| TABLE 14.2-13: ANALYSIS OF TIMED UP-AND-GO TEST (SECONDS) – EFFICACY ANALYSIS SET | S<br>91 |
| TABLE 14.2-14: ANALYSIS OF STAIR CLIMB TEST – EFFICACY ANALYSIS SET | 92 |
| TABLE 14.2-15.1.1.1: REGION ANALYSIS OF AUC OF VAS PAIN INTENSITY SCORES THROUGH 72 HOURS – EFFICACY ANALYSIS SET - MULTIPLE IMPUTATION RESULTS | 93 |
| TABLE 14.2-15.1.2.1: REGION ANALYSIS OF AUC OF VAS PAIN INTENSITY SCORES THROUGH 72 HOURS – PER-PROTOCOL ANALYSIS SET - MULTIPLE IMPUTATION RESULTS | 93 |
| TABLE 14.2-15.2.1.1: REGION ANALYSIS OF POSTSURGICAL TOTAL OPIOID CONSUMPTION (MED MG) THROUGH 72 HOURS – EFFICACY ANALYSIS SET | N<br>93 |
| TABLE 14.2-15.2.1.2: REGION SUMMARY OF TOTAL OPIOID CONSUMPTION (MED MG) THROUGH 72 HOURS BY REGION - EFFICACY ANALYSIS SET | 93 |
| TABLE 14.2-15.2.1.3: REGION SUMMARY OF TOTAL OPIOID CONSUMPTION (MED MG) BY TIME PERIOD - EFFICACY ANALYSIS SET | 93 |
| TABLE 14.2-15.2.1.4: REGION SUMMARY OF THE NUMBER OF TIMES OPIOID (RESCUE) MEDICATION WAS USED BY SUBJECT - EFFICACY ANALYSIS SET | 93 |
| TABLE 14.2-15.2.2.1: REGION ANALYSIS OF POSTSURGICAL TOTAL OPIOID CONSUMPTION (MED MG) THROUGH 72 HOURS – PER-PROTOCOL ANALYSIS SET | N<br>93 |
| TABLE 14.2-15.2.2.2: REGION SUMMARY OF TOTAL OPIOID CONSUMPTION (MED MG) THROUGH 72 HOURS BY SITE - PER-PROTOCOL ANALYSIS SET | 94 |
| TABLE 14.2-15.2.2.3: REGION SUMMARY OF TOTAL OPIOID CONSUMPTION (MED MG) BY TIME PERIOD - PER-PROTOCOL ANALYSIS SET | 94 |
| TABLE 14.2-15.2.2.4: REGION SUMMARY OF THE NUMBER OF TIMES OPIOID (RESCUE) MEDICATION WAS USED BY SUBJECT - PER-PROTOCOL ANALYSIS SET | 94 |
| TABLE 14.2-15.3.1.1: REGION ANALYSIS OF OPIOID-FREE SUBJECTS THROUGH 72 HOURS - EFFICACY ANALYSIS SET | 94 |
| TABLE 14.2-15.3.1.2: REGION SUMMARY OF OPIOID-FREE SUBJECTS THROUGH 72 HOURS BY SITE - EFFICACY ANALYSIS SET | 94 |
| TABLE 14.2-15.3.2.1: REGION ANALYSIS OF OPIOID-FREE SUBJECTS THROUGH 72 HOURS - PER-PROTOCOL ANALYSIS SET | 94 |
| TABLE 14.2-15.3.2.2: REGION SUMMARY OF OPIOID-FREE SUBJECTS THROUGH 72 HOURS BY SITE - PER-PROTOCOL ANALYSIS SET | 94 |
| TABLE 14.3-1.1.1: SUMMARY OF CLINICAL LABORATORY DATA BY TIMEPOINT – HEMATOLOGY - SAFETY ANALYSIS SET | 95 |


| TABLE 14.3-1.1.2: SUMMARY OF CLINICAL LABORATORY DATA BY TIMEPOINT – CHEMISTRY - SAFETY ANALYSIS SET | 96 |
|---|---|
| TABLE 14.3-1.1.3.1: SUMMARY OF CLINICAL LABORATORY DATA BY TIMEPOINT – URINALYSIS - SAFETY ANALYSIS SET | 96 |
| TABLE 14.3-1.1.3.2: TABULATION OF CLINICAL LABORATORY DATA BY TIMEPOINT – URINALYSIS - SAFETY ANALYSIS SET | 97 |
| TABLE 14.3-1.2.1: TABULATION OF CLINICAL LABORATORY RANGE BY TIMEPOINT – HEMATOLOGY - SAFETY ANALYSIS SET | 98 |
| TABLE 14.3-1.2.2: TABULATION OF CLINICAL LABORATORY RANGE BY TIMEPOINT – CHEMISTRY - SAFETY ANALYSIS SET | 98 |
| TABLE 14.3-1.2.3: TABULATION OF CLINICAL LABORATORY RANGE BY TIMEPOINT – URINALYSIS - SAFETY ANALYSIS SET | 98 |
| TABLE 14.3-1.3.1: SHIFT TABLE FOR CLINICAL LABORATORY DATA BY TIMEPOINT – HEMATOLOGY - SAFETY ANALYSIS SET | 99 |
| TABLE 14.3-1.3.2: SHIFT TABLE FOR CLINICAL LABORATORY DATA BY TIMEPOINT – CHEMISTRY - SAFETY ANALYSIS SET | 99 |
| TABLE 14.3-1.3.3: SHIFT TABLE FOR CLINICAL LABORATORY DATA BY TIMEPOINT – URINALYSIS - SAFETY ANALYSIS SET | 99 |
| TABLE 14.3-2.1: SUMMARY OF VITAL SIGNS BY TIMEPOINT – SAFETY ANALYSIS SET | 100 |
| TABLE 14.3-2.2: SUMMARY OF POTENTIALLY CLINICALLY SIGNIFICANT ABNORMAL VITAL SIGNS – SAFETY ANALYSIS SET | 102 |
| TABLE 14.3-3.1: SUMMARY OF ELECTROCARDIOGRAM INTERPRETATION – INVESTIGATION – INVESTIGATION – SAFETY ANALYSIS SET | ΓOR<br>105 |
| TABLE 14.3-3.2: SHIFT TABLE FOR ELECTROCARDIOGRAM INTERPRETATION – INVESTIGATOR READ - SAFETY ANALYSIS SET | 106 |
| TABLE 14.3-4: SUMMARY OF NEUROLOGICAL ASSESSMENTS BY TIMEPOINT- SAFETY ANALYSIS SET | 107 |
| TABLE 14.3-5.1: TABULATION OF SENSATION TESTS – SAFETY ANALYSIS SET | 108 |
| TABLE 14.3-5.2: SUMMARY OF SENSATION LOSS AND RETURN BY TIMEPOINT – SAFETY ANALYSIS SET | 109 |
| TABLE 14.3-5.3.1: ANALYSIS OF TIME TO FIRST SENSATION LOSS – SAFETY ANALYSIS S | SET110 |
| TABLE 14.3-5.4.1: ANALYSIS OF TIME TO FIRST SENSATION RETURN – SAFETY ANALYS SET | IS<br>112 |
| TABLE 14.3-5.5: SUMMARY OF DURATION (HRS) OF SENSATION LOSS – SAFETY ANALY SET | SIS<br>114 |
| TABLE 14.3-5.6: SUMMARY OF THE NUMBER OF SENSATION LOSS-RETURN CYCLES - SAFETY ANALYSIS SET | 115 |
| TABLE 14.3-6.1: SUMMARY OF ACTIVE MOTOR FUNCTION LOSS AND RETURN BY TIMEPOINT – SAFETY ANALYSIS SET | 116 |
| TABLE 14.3-6.2: ANALYSIS OF TIME TO ONSET OF MOTOR FUNCTION LOSS - EFFICACY ANALYSIS SET | 117 |
| TABLE 14.3-6.3: ANALYSIS OF TIME TO RETURN OF MOTOR FUNCTION - EFFICACY ANALYSIS SET | 118 |


| | 6.4: SUMMARY OF MOTOR FUNCTION ASSESSMENTS BY TIMEPOINT – SAFET ANALYSIS SET | Y<br>119 |
|---|---|---|
| TABLE 14.3- | 7.1: OVERVIEW OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) - SAFETY ANALYSIS SET | 121 |
| | 7.1.2: SUMMARY OF INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) - SAFETY ANALYSIS SET | 122 |
| TABLE 14.3- | 7.1.3: SUMMARY OF INCIDENCE OF STUDY DRUG-RELATED TREATMENT-<br>EMERGENT ADVERSE EVENTS (TEAES) - SAFETY ANALYSIS SET | 122 |
| | 7.1.4: SUMMARY OF INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) LEADING TO STUDY WITHDRAWAL - SAFETY ANALYSIS SE | ET122 |
| TABLE 14.3- | 7.1.5: SUMMARY OF INCIDENCE OF STUDY DRUG-RELATED TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) LEADING TO STUDY WITHDRAWAL -SAFETY ANALYSIS SET | 122 |
| TABLE 14.3- | 7.1.6: SUMMARY OF INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) BY SEVERITY - SAFETY ANALYSIS SET | 123 |
| TABLE 14.3- | 7.1.7: SUMMARY OF INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) BY RELATIONSHIP TO STUDY DRUG - SAFETY ANALYSIS SI | ET124 |
| TABLE 14.3- | 7.2.1: OVERVIEW OF SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) - SAFETY ANALYSIS SET | 125 |
| TABLE 14.3- | 7.2.2: SUMMARY OF INCIDENCE OF SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) - SAFETY ANALYSIS SET | 125 |
| TABLE 14.3- | 7.2.3: SUMMARY OF INCIDENCE OF STUDY DRUG-RELATED SERIOUS<br>TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) - SAFETY ANALYSIS SE | T125 |
| | 7.2.4: SUMMARY OF INCIDENCE OF SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) LEADING TO STUDY WITHDRAWAL - SAFETY ANALYSIS SET | 125 |
| TABLE 14.3- | 7.2.5: SUMMARY OF INCIDENCE OF STUDY DRUG-RELATED SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) LEADING TO STUDY WITHDRAWAL - SAFETY ANALYSIS SET | 125 |
| | 7.2.6: SUMMARY OF INCIDENCE OF SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) RESULTING IN DEATH - SAFETY ANALYSIS SET | 125 |
| TABLE 14.3- | 7.2.7: SUMMARY OF INCIDENCE OF STUDY DRUG-RELATED SERIOUS<br>TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) RESULTING IN DEATH -<br>SAFETY ANALYSIS SET | 125 |
| TABLE 14.3- | 7.3.1: OVERVIEW OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) OF SPECIAL INTEREST - SAFETY ANALYSIS SET | 125 |
| | 7.3.2: SUMMARY OF INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) OF SPECIAL INTEREST - SAFETY ANALYSIS SET | 125 |
| | 7.3.3: SUMMARY OF INCIDENCE OF STUDY DRUG-RELATED TREATMENT-<br>EMERGENT ADVERSE EVENTS (TEAES) OF SPECIAL INTEREST - SAFETY<br>ANALYSIS SET | 125 |
| | 7.3.4: SUMMARY OF INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) OF SPECIAL INTEREST LEADING TO STUDY WITHDRAWAL SAFETY ANALYSIS SET | -<br>125 |


| TABLE 14.3- | -7.3.5: SUMMARY OF INCIDENCE OF STUDY DRUG-RELATED TREATMENT-<br>EMERGENT ADVERSE EVENTS (TEAES) OF SPECIAL INTEREST LEADING TO<br>STUDY WITHDRAWAL - SAFETY ANALYSIS SET | 126 |
|---|---|---|
| TABLE 14.3- | -7.3.6: SUMMARY OF INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) OF SPECIAL INTEREST RESULTING IN DEATH - SAFETY ANALYSIS SET | 126 |
| TABLE 14.3- | -7.3.7: SUMMARY OF INCIDENCE OF STUDY DRUG-RELATED TREATMENT-<br>EMERGENT ADVERSE EVENTS (TEAES) OF SPECIAL INTEREST RESULTING II<br>DEATH - SAFETY ANALYSIS SET | N<br>126 |
| TABLE 14.3- | -8.1: INCIDENCE OF PRIOR MEDICATIONS – SAFETY ANALYSIS SET | 127 |
| TABLE 14.3- | -8.2: INCIDENCE OF CONCOMITANT MEDICATIONS – SAFETY ANALYSIS SET | 127 |
| TABLE 14.3- | -9.1.1: REGION TABULATION OF SENSATION TESTS – SAFETY ANALYSIS SET | 128 |
| TABLE 14.3- | -9.1.2: REGION SUMMARY OF SENSATION LOSS AND RETURN BY TIMEPOINT SAFETY ANALYSIS SET | _<br>128 |
| TABLE 14.3- | -9.1.3: REGION ANALYSIS OF TIME TO SENSATION LOSS – SAFETY ANALYSIS SET | 128 |
| TABLE 14.3- | -9.1.4: REGION ANALYSIS OF TIME TO SENSATION RETURN – SAFETY<br>ANALYSIS SET | 128 |
| TABLE 14.3- | -9.1.5: REGION SUMMARY OF DURATION (HRS) OF SENSATION LOSS – SAFETY<br>ANALYSIS SET | 7<br>128 |
| TABLE 14.3- | -9.2.1: REGION SUMMARY OF ACTIVE MOTOR FUNCTION LOSS AND RETURN BY TIMEPOINT – SAFETY ANALYSIS SET | 128 |
| TABLE 14.3- | -9.2.2: REGION ANALYSIS OF TIME TO ONSET OF MOTOR FUNCTION LOSS - EFFICACY ANALYSIS SET | 128 |
| TABLE 14.3- | -9.2.3: REGION ANALYSIS OF TIME TO RETURN OF MOTOR FUNCTION -<br>EFFICACY ANALYSIS SET | 128 |
| TABLE 14.3- | -9.2.4: REGION SUMMARY OF MOTOR FUNCTION ASSESSMENTS BY TIMEPOIN<br>– SAFETY ANALYSIS SET | JT<br>128 |
| TABLE 14.3- | -9.3.1: REGION OVERVIEW OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) - SAFETY ANALYSIS SET | 129 |
| TABLE 14.3- | -9.3.2: REGION SUMMARY OF INCIDENCE OF TREATMENT-EMERGENT<br>ADVERSE EVENTS (TEAES) - SAFETY ANALYSIS SET | 130 |
| TABLE 14.3- | -9.3.3: REGION SUMMARY OF INCIDENCE OF SERIOUS TREATMENT-EMERGEN | NT<br>130 |


Protocol: 402-C-326

Pacira Pharmaceuticals (Page X of Y) Table 14.1-1: Summary of Subject Disposition - All Screened Subjects

| Site: Overall | | EXPARI | EL | | |
|---|---|---|---|---|---|
| | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| | n (%) | n (응) | n (%) | n (응) | n (%) |
| Screened [1] | | | | | XX |
| Screen Failure [1] | | | | | xx (xx.x) |
| Enrolled [1] | | | | | xx (xx.x) |
| Randomized | XX | XX | XX | XX | XX |
| Not Treated | XX | XX | XX | XX | XX |
| Treated | XX | XX | XX | XX | XX |
| Safety Analysis Set [2]# | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Efficacy Analysis Set [3]@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Per-Protocol Analysis Set [4]@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol | | | | | |
| Enrolled under Amendment 2 [2]# | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Enrolled under Amendment 1 [2]# | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Study@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued from Study@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reasons for Discontinuation@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse Event@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lack of Efficacy@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to Follow-up@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal by Subject@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup># =</sup> as treated;

Percentages for screen failure and enrolled based on number screened; others on number randomized.

Subjects randomized to EXPAREL but treated with placebo: list subjects;

Subjects randomized to placebo but treated with EXPAREL: list subjects; Source: list SAS datasets used to create table


DDMONYYYYTHH:MM

<sup>@ =</sup> as randomized;

<sup>[1]</sup> Signed the informed consent form; [2] Received study drug; [3] Received study drug and surgery;

<sup>[4]</sup> All subjects in the efficacy analysis set who do not have any important protocol deviations;

SAS X.Y program name

Note to programmer: First page will present overall sites; subsequent pages will present each site - one site per page. For reasons for discontinuation only those reasons that appear in the data will appear on the table. For individual sites the label should be the site number. For the footnotes "Subjects treated with..." if no subjects were mistreated, then omit footnote.

Protocol: 402-C-326

Pacira Pharmaceuticals (Page X of Y)
Table 14.1-2.1.1: Summary of Subject Demographics - Safety Analysis Set

| Site: Overall | | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | Statistic | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| | | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| Age (yrs) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |
| Sex | | | | | | |
| Female | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Male | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity | | | | | | |
| Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race | | | | | | |
| American Indian/Alaska Native | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black/African American | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| White | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Native Hawaiian/Pacific Islander | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Country | | | | | | |
| Belgium | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Denmark | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| USA | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: list SAS datasets used to create table
SAS X.Y

DDMONYYYYTHH:MM
program\_name


Note to programmer: First page will present overall sites; subsequent pages will present each site - one site per page. Only categories available in the data will appear on the table. For individual sites the label should be the site number. If subjects are missing data for a category (example Race), a missing subcategory should be added under the respective category. Use this mock-up also for table:

Table 14.1-2.1.2: Subject Demographics - Efficacy Analysis Set Table 14.1-2.1.3: Subject Demographics - Per-protocol Analysis Set

Pacira Pharmaceuticals  Protocol: 402-C-326

Table 14.1-2.2.1: Summary of Subject Baseline Characteristics - Safety Analysis Set

| Site: Overall | | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| | Statistic | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| Neurological Assessments | | | | | | |
| Subject oriented | | | | | | |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Numb lips, tongue, mouth | ( - / | ( | ( , | , | , , , | , |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Metallic taste | , , | , | , | , , | , | , |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Problems hearing | | | | | | |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Problems with vision | | | | | | |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Muscle twitch | | | | | | |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| ECG | | | | | | |
| Normal | n (응) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Abnormal, NCS | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Abnormal, CS | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Source: list SAS datasets used to create table

DDMONYYYYTHH:MM program\_name

SAS X.Y

Note to programmer: If subjects are missing data for a category (example Race), a missing subcategory should be added under the respective category.

Pacira Pharmaceuticals  Protocol: 402-C-326 Table 14.1-2.2.1: Summary of Subject Baseline Characteristics - Safety Analysis Set

| Site: Overall | | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| | Statistic | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| Motor Assessments | | | | | | |
| Active Flexion (degrees) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |
| Active Extension (degrees) | n | XX | XX | xx | xx | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |
| Passive Flexion (degrees) | n | xx | xx | xx | xx | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |

Source: list SAS datasets used to create table
SAS X.Y

DDMONYYYYTHH:MM
program\_name

Pacira Pharmaceuticals  Protocol: 402-C-326

Table 14.1-2.2.1: Summary of Subject Baseline Characteristics - Safety Analysis Set

| Site: Overall | | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| | Statistic | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| Motor Assessments | | | | | | |
| Passive Extension (degrees) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |
| VAS Score (cm) | n | xx | xx | xx | xx | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

Pacira Pharmaceuticals  Protocol: 402-C-326 Table 14.1-2.2.1: Summary of Subject Baseline Characteristics - Safety Analysis Set

| Site: Overall | | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | Statistic | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| | | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| ASA Classification | | | | | | |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ≥ 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Height (cm) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |
| Weight (kg) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |
| | Maximum | XX | XX | XX | XX | XX |
| Body Mass Index $(kg/m^2)$ | | | | | | |
| | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |
| | Maximum | XX | XX | XX | XX | XX |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

Pacira Pharmaceuticals  Protocol: 402-C-326 Table 14.1-2.2.1: Summary of Subject Baseline Characteristics - Safety Analysis Set

| Site: Overall | | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | Statistic | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| | | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| Heart Rate (bpm) | n | XX | XX | XX | XX | XX |
| (1) | Mean | XX.X | XX.X | XX.X | XX.X | xx.x |
| | SD | X.XX | X.XX | X.XX | X.XX | x.xx |
| | Minimum | XX | XX | XX | XX | xx |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |
| Systolic Blood Pressure (mmHg) | n | XX | XX | XX | XX | XX |
| | Mean | xx.x | XX.X | XX.X | XX.X | xx.x |
| | SD | X.XX | X.XX | X.XX | X.XX | x.xx |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |
| Diastolic Blood Pressure (mmHg) | n | XX | XX | XX | XX | XX |
| . 5. | Mean | xx.x | XX.X | XX.X | XX.X | xx.x |
| | SD | x.xx | x.xx | X.XX | x.xx | x.xx |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |
| | Maximum | XX | XX | XX | XX | XX |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

**Note to programmer:** First page will present overall sites; subsequent pages will present each site - one site per page. For individual sites the label should be the site number. Use this mock-up also for table:

Table 14.1-2.2.2: Subject Baseline Characteristics - Efficacy Analysis Set Table 14.1-2.2.3: Subject Baseline Characteristics - Per-protocol Analysis Set

Protocol: 402-C-326

Pacira Pharmaceuticals (Page X of Y)
Table 14.1-3.1: Summary of Surgery Characteristics - Safety Analysis Set

| Site: Overall | | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| Characteristic | Statistic | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| Duration of Surgery (hours) | n | xx | xx | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX | XX | XX | XX | XX |
| | Minimum | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |
| Tourniquet | | | | | | |
| Used | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not Used | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Duration (hours) | n | xx | xx | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX | XX | XX | XX | XX |
| | Minimum | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | xx | xx | XX | XX | XX |
| Drain | | | | | | |
| Used | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not Used | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Duration (hours) | n | XX | xx | xx | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX | XX | XX | XX | XX |
| | Minimum | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

**Note to programmer:** First page will present overall sites; subsequent pages will present each site - one site per page. For individual sites the label should be the site number.

Use this mock-up also for tables:

Table 14.1-3.2: Summary of Surgery Characteristics - Efficacy Analysis Set Table 14.1-3.3: Summary of Surgery Characteristics - Per-protocol Analysis Set

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326
Table 14.1-4.1: Incidence of Intraoperative Medications - Safety Analysis Set

| Table III III I III I I I I I I I I I I I I | ve mearcacrome | Darcey IIIIa | TYDID DCC | | |
|---|---|---|---|---|---|
| | | EXPAREL | | | |
| | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| Anatomical Therapeutic Class (ATC) | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| Preferred Name | n (응) | n (응) | n (응) | n (%) | n (응) |
| Subjects taking at least one medication | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PN1.1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PN1.2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PN2.1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PN2.2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ETC. | | | | | |

Medications are coded using World Health Organization Drug Dictionary (WHO-DD) March 2015.

Sorted by descending total incidence by ATC for Total column. Subjects using the same intraoperative medication (PT) more than once or multiple medications within an ATC class are counted only once at each ATC summary level.

Intraoperatives medications are those indicated as such by the investigator.

Subjects using the same prior medication more than once are counted only once at each summary level.

Source: list SAS datasets used to create table DDMONYYYYTHH:MM program name

**Note to programmer:** Use mock-up 14.1-4.1 for tables:

Table 14.1-4.2: Incidence of Intraoperative Medications - Efficacy Analysis Set
Table 14.1-4.3: Incidence of Intraoperative Medications - Per-protocol Analysis Set

Note to programmer: For the following region summaries, 'Site:' will be replaced with 'Region:'. Regions, in order of appearance, are US and ROW. There will be no overall region summary presented on these tables. Use mock-up 14.1-1 for table: Table 14.1-5.1: Summary of Subject Disposition - By Region - All Screened Subjects Use mock-up 14.1-2.1.1 for tables: Table 14.1-5.2.1.1: Summary of Subject Demographics - By Region - Safety Analysis Set Table 14.1-5.2.1.2: Subject Demographics - By Region - Efficacy Analysis Set Table 14.1-5.2.1.3: Subject Demographics - By Region - Per-protocol Analysis Set Use mock-up 14.1-2.2.1 for tables: Table 14.1-5.2.2.1: Summary of Subject Baseline Characteristics - By Region - Safety Analysis Set Table 14.1-5.2.2.2: Subject Baseline Characteristics - By Region - Efficacy Analysis Set Table 14.1-5.2.2.3: Subject Baseline Characteristics - By Region - Per-protocol Analysis Set Use mock-up 14.1-3.1 for tables: Table 14.1-5.3.1: Summary of Surgery Characteristics - By Region - Safety Analysis Set Table 14.1-5.3.2: Summary of Surgery Characteristics - By Region - Efficacy Analysis Set Table 14.1-5.3.3: Summary of Surgery Characteristics - By Region - Per-protocol Analysis Set


Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-1.1.1: Analysis of AUC of VAS Pain Intensity Scores through 72 hours - Efficacy Analysis Set - Multiple Imputation Results

| | EXP | AREL | |
|---|---|---|---|
| | 133 mg | 266 mg | Placebo |
| Statistic | [N=XX] | [N=XX] | [N=XX] |
| N | XX | XX | XX |
| Mean | XXX.X | XXX.X | XXX.X |
| SD | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.X | XXX.X | XXX.X |
| Minimum | XX | XX | XX |
| Maximum | XXX | XXX | xxx |
| LS Mean [1] | xxx.x | XXX.X | xxx.x |
| Standard Error of LS Mean [1] | xxx.xx | xxx.xx | XXX.XX |
| LS Treatment Difference [1][2] | XX.X | xx.x | |
| Treatment Difference 95% Confidence Interval [1][2] | (xx.x, xx.x) | (xx.x, xx.x) | |
| Treatment Difference p-value [1][2] | 0.xxx | 0.xxx | |

AUC = area under the curve calculated using the trapezoidal method;

LS = least squares;

VAS = 10 cm visual analog scale for pain, where 0 = no pain and 10 = worst possible pain;

- [1] From an ANOVA with age, weight, and height as covariates.
- [2] Treatment difference is EXPAREL placebo.

Source: list SAS datasets used to create table

DDMONYYYYTHH:MM program name

SAS X.Y

Note to programmer: The raw SAS outputs from the procedures used to produce ALL 14.2-1.1.\* & 14.2-1.2 series tables should be saved as a possible appendix to the clinical study report (CSR).

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-1.1.2: Summary of AUC of VAS Pain Intensity Scores through 72 hours by Site - Efficacy Analysis Set - Multiple Imputation Results

| | | EXPAREL | | |
|-------|-----------|---------|--------|---------|
| | | 133 mg | 266 mg | Placebo |
| Site | Statistic | [N=XX] | [N=XX] | [N=XX] |
| XXX | N | XX | XX | XX |
| 12121 | Mean | XXX.X | XXX.X | XXX.X |
| | SD | XXX.XX | XXX.XX | xxx.xx |
| | Median | XXX.X | XXX.X | XXX.X |
| | Minimum | XX | XX | XX |
| | Maximum | XXX | XXX | XXX |
| YYY | N | XX | XX | XX |
| | Mean | XXX.X | XXX.X | xxx.x |
| | SD | XXX.XX | xxx.xx | xxx.xx |
| | Median | XXX.X | XXX.X | XXX.X |
| | Minimum | XX | XX | XX |
| | Maximum | XXX | XXX | XXX |
| ZZZ | N | XX | XX | xx |
| | Mean | XXX.X | XXX.X | xxx.x |
| | SD | xxx.xx | xxx.xx | xxx.xx |
| | Median | xxx.x | xxx.x | xxx.x |
| | Minimum | xx | XX | XX |
| | Maximum | XXX | xxx | xxx |

AUC = area under the curve calculated using the trapezoidal method;

LS = least squares;

VAS = 10 cm visual analog scale for pain, where 0 = no pain and 10 = worst possible pain;

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

**Note to programmer:** The raw SAS outputs from the procedures used to produce ALL 14.2-1.1.\* series tables should be saved as a possible appendix to the clinical study report (CSR).


### Mock-up 14.2-1.1.1:

Table 14.2-1.2.1: Analysis of AUC of VAS Pain Intensity Scores through 72 hours - Per-protocol Analysis Set - Multiple Imputation Results

### Mock-up 14.2-1.1.2:

Table 14.2-1.2.2: Summary of AUC of VAS Pain Intensity Scores through 72 hours by Site - Per-protocol Analysis Set - Multiple Imputation Results


Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-2.1.1: Analysis of Postsurgical Total Opioid Consumption (MED mg) through 72 hours - Efficacy Analysis Set

| Statistic | EXPAREL 133 mg<br>[N=XX] | EXPAREL 266 mg [N=XX] | Placebo<br>[N=XX] |
|---|---|---|---|
| N | | | |
| N<br>Geometric Mean | XX<br>XXX.X | XX<br>XXX.X | XX<br>XXX.X |
| %CV | XXX.XX | XXX.XX | XXX.XX |
| Minimum | xx | XX | XX |
| Maximum | XXX | XXX | XXX |
| LS Mean [1] | XXX.X | xxx.x | XXX.X |
| Standard Error of LS Mean [1] | xxx.xx | xxx.xx | XXX.XX |
| LS Treatment Ratio [1][2] | XX.X | xx.x | |
| Treatment Ratio 95% Confidence Interval [1][2] | (xx.x, xx.x) | (xx.x, xx.x) | |
| Treatment Ratio p-value [1][2] | 0.xxx | 0.xxx | |

<sup>[1]</sup> From an ANOVA with age, weight, and height as covariates on log-transformed total opioid consumption. Subjects without any opioid use are set to 0.1 or half of the smallest total amount observed in the study, whichever is smaller, prior to being transformed with the natural logarithm. Results are backtransformed.

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

<sup>[2]</sup> Treatment ratio is EXPAREL / placebo.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-2.1.2: Summary of Total Opioid Consumption (MED mg) through 72 hours by Site - Efficacy Analysis Set

| | | EXPAREL 133 mg | EXPAREL 266 mg | Placebo |
|------|----------------|----------------|----------------|---------|
| Site | Statistic | [N=XX] | [N=XX] | [N=XX] |
| XXX | n | XX | XX | XX |
| | Geometric Mean | XX.X | XX.X | XX.X |
| | %CV | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX |
| | Maximum | XX | XX | XX |
| YYY | n | XX | XX | XX |
| | Geometric Mean | XX.X | XX.X | XX.X |
| | %CV | x.xx | X.XX | X.XX |
| | Minimum | XX | XX | XX |
| | Maximum | XX | XX | XX |
| 777 | _ | | | |
| ZZZ | n | XX | XX | XX |
| | Geometric Mean | xx.x | XX.X | XX.X |
| | %CV | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX |
| | Maximum | XX | XX | XX |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

**Note to programmer:** Present for each site. For pooled sites, present the pooled site first and then each site contributing to the pool immediately after. Do not split a site's statistics across pages.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-2.1.3: Analysis of Total Opioid Consumption (MED mg) by Time Period - Efficacy Analysis Set

| | | EXPAREL 133 mg | EXPAREL 266 mg | Placebo |
|---|---|---|---|---|
| | Statistic | [N=XX] | [N=XX] | [N=XX] |
| 0-24 hrs | N | | | |
| 0-24 HIS | | XX | XX | XX |
| | Geometric Mean | XXX.X | XXX.X | XXX.X |
| | %CV | XXX.XX | XXX.XX | XXX.XX |
| | Minimum | XX | XX | XX |
| | Maximum | XXX | XXX | XXX |
| | LS Mean [1] | XXX.X | XXX.X | xxx.x |
| | Standard Error of LS Mean [1] | xxx.xx | xxx.xx | XXX.XX |
| | LS Treatment Ratio [1][2] | xx.x | xx.x | |
| | Treatment Ratio 95% Confidence | | | |
| | Interval [1][2] | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Treatment Ratio p-value [1][2] | 0.xxx | 0.xxx | |
| 0-48 hrs | N | XX | XX | XX |
| | Geometric Mean | XXX.X | XXX.X | XXX.X |
| | %CV | XXX.XX | XXX.XX | XXX.XX |
| | Minimum | XX | XX | XX |
| | Maximum | XXX | XXX | XXX |
| | LS Mean [1] | XXX.X | xxx.x | xxx.x |
| | Standard Error of LS Mean [1] | xxx.xx | xxx.xx | XXX.XX |
| | LS Treatment Ratio [1][2] | xx.x | XX.X | |
| | Treatment Ratio 95% Confidence | | | |
| | Interval [1][2] | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Treatment Ratio p-value [1][2] | XXX.X | XXX.X | XXX.X |

<sup>[1]</sup> From an ANOVA with age, weight, and height as covariates on log-transformed total opioid consumption. Subjects without any opioid use are set to 0.1 or half of the smallest total amount observed in the study, whichever is smaller, prior to being transformed with the natural logarithm. Results are backtransformed.

Source: list SAS datasets used to create table SAS  $\rm X.Y$ 

DDMONYYYYTHH:MM program name

<sup>[2]</sup> Treatment ratio is EXPAREL / placebo.

**Note to programmer:** Time periods to appear on this table, in order, are 0-24, 0-48, 0-96, 24-48, 48-72 and 72-96. Do not split a time period statistics across pages.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-2.1.4: Summary of the Number of Times Opioid (Rescue) Medication was used by Subject - Efficacy Analysis Set

| | | EXPAREL 133 mg | EXPAREL 266 mg | Placebo |
|--------------------|-----------|----------------|----------------|-----------|
| | Statistic | [N=XX] | [N=XX] | [N=XX] |
| Count Summary | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Minimum | XX.X | XX.X | XX.X |
| | Median | XX | XX | XX |
| | Maximum | XX | XX | XX |
| Count Distribution | | | | |
| 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| U | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM

program name

**Note to programmer:** Present overall sites and for each site. Distribution should present all counts up to the highest number of visits in the data (U) on each page.

Note to programmer: Use the mock-ups indicated to for following tables:

#### Mock-up 14.2.1.1:

Table 14.2-2.2.1: Analysis of Postsurgical Total Opioid Consumption (MED mg) through 72 hours - Per-protocol Analysis Set

#### Mock-up 14.2.1.2:

Table 14.2-2.2.2: Summary of Total Opioid Consumption (MED mg) through 72 hours by Site - Per-protocol Analysis Set

#### Mock-up 14.2.1.3:

Table 14.2-2.2.3: Analysis of Total Opioid Consumption (MED mg) by Time Period - Per-protocol Analysis Set Set.

### Mock-up 14.2.1.4:

Table 14.2-2.2.4: Summary of the Number of Times Opioid (Rescue) Medication was used by Subject - Per-protocol Analysis Set


Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-3.1.1: Analysis of Opioid-Free Subjects through 72 hours - Efficacy Analysis Set

| | EXPAREL | | | |
|---|---|---|---|---|
| | Statistic | 133 mg<br>[N=XX] | 266 mg<br>[N=XX] | Placebo<br>[N=XX] |
| No Opioid Use | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Opioid Used | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Treatment Difference [1] | XX.X | XX.X | |
| | 95% CI for Difference [1] p-value [2] | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx | |

<sup>[1]</sup> Treatment difference (EXPAREL - placebo) and confidence intervals (CI) are based on the normal approximation to the binomial distribution using SAS PROC FREQ with RISKDIFFC option.

Source: list SAS datasets used to create table SAS  $\rm X.Y$ 

DDMONYYYYTHH:MM program name

<sup>[2]</sup> From Cochran-Mantel-Haenszel (CMH) test.
SAS X.Y

Source: list SAS datasets used to create table

DDMONYYYYTHH:MM

program name

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-3.1.2: Summary of Opioid-Free Subjects through 72 hours by Site - Efficacy Analysis Set

| | EXPAREL | | | |
|---------------|-----------|-----------|-----------|-----------|
| Site | | 133 mg | 266 mg | Placebo |
| Opioid Use | Statistic | [N=XX] | [N=XX] | [N=XX] |
| XXX | | | | |
| No Opioid Use | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Opioid Used | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| YYY | | | | |
| No Opioid Use | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Opioid Used | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Etc. | | | | |
| No Opioid Use | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Opioid Used | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

**Note to programmer:** Present for each site. For pooled sites, present the pooled site first and then each site contributing to the pool immediately after. Do not split a site's statistics across pages.

Note to programmer: Use the mock-ups indicated to for following tables:

Mock-up 14.2-3.1.1:

Table 14.2-3.2.1: Analysis of Opioid-Free Subjects through 72 hours - Per-protocol Analysis Set

Mock-up 14.2-3.1.2:

Table 14.2-3.2.2: Summary of Opioid-Free Subjects through 72 hours by Site - Per-protocol Analysis Set

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-4.1: Analysis of Time to First Rescue Medication Use (hours) - Efficacy Analysis Set

| | Statistic | EXPAREL 133 mg<br>[N=XX] | EXPAREL 266 mg<br>[N=XX] | Placebo<br>[N=XX] |
|---|---|---|---|---|
| Number of Orbitation | | | | |
| Number of Subjects on | (0) | , | , | , |
| Rescue Medication (Opioid) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No Rescue Medication (censored) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time to Rescue | | | | |
| Quartiles [1] | | | | |
| First (25% rescued) | Estimate | xx.xx | XX.XX | XX.XX |
| 11100 (200 1000000) | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| | (90% C1) | (ΔΔ.ΔΔ, ΔΔ.ΔΔ) | (\(\lambda\), \(\lambda\), \(\la | (\lambda \lambda \lambd |
| Median (50% rescued) | Estimate | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx, xx.xx) | (xx.xx,xx.xx) |
| Third (75% rescued) | Estimate | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Minimum | Observed | XX.XX | XX.XX | XX.XX |
| Maximum | Observed | XX.XX* | xx.xx* | XX.XX |
| p-value [2] | | 0.xxxx | 0.xxxx | |

<sup>\*</sup> indicates censored observation

Source: list SAS datasets used to create table

SAS X.Y

CI = confidence interval

DDMONYYYYTHH:MM program name

Note to programmer: Use this mock-ups indicated to for following table:

Table 14.2-4.2: Analysis of Time to First Rescue Medication Use (hours) - Per-protocol Analysis Set

<sup>[1]</sup> Estimates from Kaplan-Meier analysis.

<sup>[2]</sup> p-value from Log-rank test comparing EXPAREL to placebo.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326

Table 14.2-5.1: Summary of VAS AUC at Various Time Intervals - Efficacy Analysis Set

| E | EXPAREL 133 | EXPAREL 266 | |
|---|---|---|---|
| | mg | mg | Placebo |
| | [N=XX] | [N=XX] | [N=XX] |
| | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| | X.XX | X.XX | X.XX |
| | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| | XX | XX | XX |
| | xxx.x | XXX.X | xxx.x |
| | XXX.XX | XXX.XX | XXX.XX |
| | XX.X | XX.X | |
| rval [1][2] | (xx.x, xx.x) | (xx.x, xx.x) | |
| | 0.xxx | 0.xxx | |
| | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| | X.XX | X.XX | X.XX |
| | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| | XX | XX | XX |
| | xxx.x | XXX.X | xxx.x |
| | XXX.XX | XXX.XX | XXX.XX |
| | XX.X | XX.X | |
| rval [1][2] | | | |
| | 0.xxx | 0.xxx | |
| 9 | erval [1][2] | erval [1][2] (xx.x, xx.x) | erval [1][2] (xx.x, xx.x) (xx.x, xx.x) |

AUC = area under the curve calculated using the trapezoidal method;

VAS = 10 cm visual analog scale for pain, where 0 = no pain and 10 = worst possible pain;

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

LS = least squares;

<sup>[1]</sup> From an ANOVA with age, weight, and height as covariates.

<sup>[2]</sup> Treatment difference is EXPAREL - placebo.

Note to programmer: VAS AUCs to be presented on this table are, in order, AUC(0-12), AUC(0-24), AUC(0-48), AUC(0-96), AUC(24-48), AUC(48-72) and AUC(72-96). Do not break an AUC's statistics across pages.


Protocol: 402-C-326

Pacira Pharmaceuticals (Page X of Y)
Table 14.2-5.2: Summary of VAS at Assessment Timepoints - Efficacy Analysis Set

| | | EXPAREL 133 mg | EXPAREL 266 mg | Placebo |
|-----------|-----------|----------------|----------------|---------|
| Timepoint | Statistic | [N=XX] | [N=XX] | [N=XX] |
| Baseline | n | XX | xx | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Minimum | XX | xx | XX |
| | Median | XX.X | XX.X | XX.X |
| | Maximum | xx | XX | XX |
| PACU | n | XX | xx | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | x.xx | X.XX | X.XX |
| | Minimum | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX |
| Etc. | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX |

PACU is Post Anesthesia Care Unit

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program\_name

Note to programmer: Timepoints to appear on this table are, in order, Baseline, PACU and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120 hours.

Note to programmer: Use the indicated mock-up for the following tables:

Use mock-up 14.2-5.1:

Table 14.2-5.3: Summary of VAS SPIS at Various Time Intervals - Efficacy Analysis Set

Note to programmer: Remove "AUC = area under the curve calculated using the trapezoidal method;" footnote. VAS SPIS to be presented on Table 14.2-5.3 are, in order, SPIS(0-12), SPIS(0-24), SPIS(0-48), SPIS(0-96), SPIS(24-48), SPIS(48-72) and SPIS(72-96). Do not break an SPIS's statistics across pages.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-6: Analysis of Pain-Free Subjects at Assessment Timepoints - Efficacy Analysis Set

| | EXPAREL | | | |
|---|---|---|---|---|
| Timepoint | | 133 mg | 266 mg | Placebo |
| Opioid Use | Statistic | [N=XX] | [N=XX] | [N=XX] |
| Baseline | | | | |
| Pain-Free | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pained | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Treatment Difference [1] | XX.X | XX.X | |
| | 95% CI for Difference [1] | (xx.x, xx.x) | (xx.x, xx.x) | |
| | p-value [2] | 0.xxxx | 0.xxxx | |
| Etc. | | | | |
| Pain-Free | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pained | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Treatment Difference [1] | XX.X | xx.x | |
| | 95% CI for Difference [1] | (xx.x, xx.x) | (xx.x, xx.x) | |
| | p-value [2] | 0.xxxx | 0.xxxx | |

<sup>[1]</sup> Pain-Free Treatment difference (EXPAREL - placebo) and confidence intervals (CI) are based on the normal approximation to the binomial distribution using SAS PROC FREQ with RISKDIFFC option.

Pain-free = VAS score  $\leq$  1.5 and no prior rescue medication use and all prior VAS scores  $\leq$  1.5.

Source: list SAS datasets used to create table SAS  $\rm X.Y$ 

DDMONYYYYTHH:MM program\_name

Note to programmer: Timepoints to appear on this table are, in order, Baseline, PACU and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120 hours. Do not split a timepoint across pages.

<sup>[2]</sup> From Cochran-Mantel-Haenszel (CMH) test.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-7: Analysis of Opioid-Free Subjects through 24, 48, and 96 hours - Efficacy Analysis Set

| | | EXPA | AREL | |
|---|---|---|---|---|
| Timepoint | | 133 mg | 266 mg | Placebo |
| Opioid Use | Statistic | [N=XX] | [N=XX] | [N=XX] |
| 0-24 | | | | |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Treatment Difference [1] | XX.X | XX.X | |
| | 95% CI for Difference [1] | (xx.x, xx.x) | (xx.x, xx.x) | |
| | p-value [2] | 0.xxxx | 0.xxxx | |
| 0-48 | | | | |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Treatment Difference [1] | XX.X | XX.X | |
| | 95% CI for Difference [1] | (xx.x, xx.x) | (xx.x, xx.x) | |
| | p-value [2] | 0.xxxx | 0.xxxx | |

<sup>[1]</sup> Opioid-Free Treatment difference (EXPAREL - placebo) and confidence intervals (CI) are based on the normal approximation to the binomial distribution using SAS PROC FREQ with RISKDIFFC option.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Note to programmer: Timepoints to appear on this table are, in order, 0-24, 0-48, 0-96 hours. Do not split a timepoint across pages.

<sup>[2]</sup> From Cochran-Mantel-Haenszel (CMH) test.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-8: Summary of Overall Benefit of Analgesia Scale by Timepoint and Question - Efficacy Analysis Set

| Timepoint | | | EXPAREL 133 mg | EXPAREL 266 mg | Placebo |
|---|---|---|---|---|---|
| Question | | Statistic | [N=XX] | [N=XX] | [N=XX] |
| 24 hours | | | | | |
| Total Score | Summary | n | xx | xx | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | X.XX | x.xx | X.XX |
| | | Minimum | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X |
| | | Maximum | XX | xx | XX |
| | | p-value[1] | 0.xxx | 0.xxx | |
| | Score | | | | |
| | 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1. Current Pain | Summary | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | X.XX | x.xx | X.XX |
| | | Minimum | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX |
| | Score | | | | |
| | 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Total score = sum of scores from questions 1 to 6 plus 4 minus question 7 score.

Source: list SAS datasets used to create table

program\_name

DDMONYYYYTHH:MM

SAS X.Y

Note to programmer: Timepoints to appear on this table, in order, are 24 and 72 hours and Day 10.

Questions to appear on this table, in order, are 'Total Score', '1. Current Pain', '2. Vomiting', '3.

<sup>[1]</sup> p-value from Kruskal-Wallis test.

Itching', '4. Sweating', '5. Freezing', '6. Dizziness', and '7. Satisfaction'. Do not split a question's statistics across pages. P-Values should only be generated for 'Total score'.

Note to programmer: Use the indicated mock-up for the following tables:

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-9: Summary of Satisfaction with Postsurgical Pain Control Questionnaire Score by Timepoint - Efficacy Analysis Set

| | | | EXPAREL 133 | EXPAREL 266 | |
|---|---|---|---|---|---|
| | | | mg | mg | Placebo |
| Timepoint | Score | Statistic | [N=XX] | [N=XX] | [N=XX] |
| 0.4.1 | _ | | | | |
| 24 hours | Summary | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX |
| | | p-value[1] | 0.xxx | 0.xxx | |
| | Score | | | | |
| | 1: Extremely dissatisfied | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | 2: Dissatisfied | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | 3: Neither satisfied nor dissatisfied | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | 4: Satisfied | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | 5: Extremely Satisfied | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |

<sup>[1]</sup> p-value from Kruskal-Wallis test.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

**Note to programmer:** Timepoints to appear on this table are 24 and 72 hours and Day 10. Do not split timepoint across pages.

Protocol: 402-C-326

Pacira Pharmaceuticals (Page X of Y)
Table 14.2-10.1: Summary of Time to Discharge Ready - Efficacy Analysis Set

| Assessment Time | | EXPAREL 133 mg | EXPAREL 266 mg | Placebo |
|---|---|---|---|---|
| Discharge Ready | Statistic | [N=XX] | [N=XX] | [N=XX] |
| 12 hours | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Time to Discharge Ready | | | | |
| Quartiles [1] | | | | |
| First (25% Discharge Ready) | Estimate | XX.XX | XX.XX | XX.XX |
| , | (95% CI) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Median (50% Discharge Ready) | Estimate | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Third (75% Discharge Ready) | Estimate | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx, xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Minimum | Observed | XX.XX | XX.XX | XX.XX |
| Maximum | Observed | xx.xx* | xx.xx* | xx.xx |
| p-value [2] | | 0.xxxx | 0.xxxx | |

<sup>\*</sup> indicates censored observation

Source: list SAS datasets used to create table

SAS X.Y

CI = confidence interval

DDMONYYYYTHH:MM program name

Note to programmer: Assessments Time to be presented are 12, 24, 36, 48, 60, and 72 hours.

<sup>[1]</sup> Estimates from Kaplan-Meier analysis.

<sup>[2]</sup> p-value from Log-rank test comparing EXPAREL to placebo.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326

Table 14.2-10.2: Summary of Discharge Ready by Assessment - Efficacy Analysis Set

| | | EXPA | AREL | _ |
|-----------------|-----------|-----------|-----------|-----------|
| Assessment Time | | 133 mg | 266 mg | Placebo |
| Discharge Ready | Statistic | [N=XX] | [N=XX] | [N=XX] |
| 12 hours | | | | |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 24 hours | | | | |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 36 hours | | | | |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 165 | 11 (%) | AA (AA.A) | AA (AA.A) | AA (AA.A) |
| 48 hours | | | | |
| No | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 60 hours | | | | |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 72 hours | | | | |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 96 hours | | | | |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes | n (웅) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: list SAS datasets used to create table

DDMONYYYYTHH:MM program name

SAS X.Y

Note to programmer: Do not split timepoint across pages.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.2-11: Summary of Number of Unscheduled Phone Calls or Office Visits Related to Pain - Efficacy Analysis Set

| | · | EXPAREL 133 mg | EXPAREL 266 mg | Placebo |
|---|---|---|---|---|
| | Statistic | [N=XX] | [N=XX] | [N=XX] |
| Count Summary | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Minimum | XX.X | XX.X | XX.X |
| | Median | XX | XX | XX |
| | Maximum | XX | xx | XX |
| | p-value[1] | 0.xxx | 0.xxx | |
| Count Distribution | | | | |
| 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| U | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

[1] p-value from Kruskal-Wallis test.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Note to programmer: Distribution should present all counts up to the highest number of visits in the data (U).

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-331 Table 14.2-12.1: Analysis of Distance Walked (meters) During Timed Walk Test - Efficacy Analysis Set

| Timepoint | Statistic | EXPAREL 133 mg<br>[N=XX] | EXPAREL 266 mg<br>[N=XX] | Placebo<br>[N=XX] |
|---|---|---|---|---|
| Overall | LS Mean | xxx.x | xxx.x | XXX.X |
| Overall | Standard Error of LS Mean | XXX.XX | XXX.XX | XXX.XX |
| | LS Treatment Difference | XX.X | XX.X | 212121 • 2121 |
| | Treatment Difference 95% Confidence | 22.4 | 222. • 22 | |
| | Interval | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Treatment Difference p-value | 0.xxx | 0.xxx | |
| At Day 1-PM | LS Mean | xxx.x | XXX.X | XXX.X |
| | Standard Error of LS Mean | XXX.XX | XXX.XX | XXX.XX |
| | LS Treatment Difference | XX.X | XX.X | |
| | Treatment Difference 95% Confidence | | | |
| | Interval | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Treatment Difference p-value | 0.xxx | 0.xxx | |
| At Day 2-AM | LS Mean | XXX.X | XXX.X | xxx.x |
| | Standard Error of LS Mean | XXX.XX | XXX.XX | XXX.XX |
| | LS Treatment Difference | XX.X | XX.X | |
| | Treatment Difference 95% Confidence | | | |
| | Interval | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Treatment Difference p-value | 0.xxx | 0.xxx | |
| At Day 2-PM | LS Mean | XXX.X | XXX.X | xxx.x |
| | Standard Error of LS Mean | XXX.XX | XXX.XX | XXX.XX |
| | LS Treatment Difference | XX.X | XX.X | |
| | Treatment Difference 95% Confidence | | | |
| | Interval | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Treatment Difference p-value | 0.xxx | 0.xxx | |

<sup>[1]</sup> MMRM with fixed effect of treatment and a random effect of subject within treatment with XXXX covariance structure.

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name


Note to programmer: Timepoints for this table are Day 1-PM, Day 2-AM, Day 2-PM, Day 3-AM, Day 3-PM, Day 4-AM, Day 4-PM, and Day 10.

Protocol: 402-C-331

Pacira Pharmaceuticals (Page X of Y)
Table 14.2-12.2: Summary of Timed Walk Test by Timepoint - Efficacy Analysis Set

| | | | | EXPAREL 266 | |
|---|---|---|---|---|---|
| | | | EXPAREL 133 mg | mg | Placebo |
| Timepoint | Parameter | Statistic | [N=XX] | [N=XX] | [N=XX] |
| Day 1-PM | Not performed | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Reasons not performed | | | | |
| | Pain | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Weakness | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Nausea/Vomiting | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Other | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Walking Aid | | | | |
| | No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Physical Assistance | | | | |
| | Total Assistance | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Maximal Assistance | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Minimal Assistance | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Supervision | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Modified Independence | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Complete Independence | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Distance (meters) | N | XX | xx | xx |
| | | Mean | xxx.x | XXX.X | XXX.X |
| | | SD | xxx.xx | XXX.XX | XXX.XX |
| | | Median | xxx.x | XXX.X | XXX.X |
| | | Minimum | xx | XX | XX |
| | | Maximum | xxx | XXX | XXX |

Source: list SAS datasets used to create table DDMONYYYYTHH:MM

SAS X.Y program\_name

Note to programmer: Break out by site. Timepoints for this table are Day 1-PM, Day 2-AM, Day 2-PM, Day 3-AM, Day 3-PM, Day 4-AM, Day 4 - PM, and Day 10 with one timepoint per page. If a subject did not have an evaluation at a given timepoint then they should be counted under "Not performed".

Note to programmer: Timepoints for this table are Day 1-PM, Day 2-AM, Day 2-PM, Day 3-AM, Day 3-PM, Day 4-AM, and Day 14. If a subject did not have an evaluation at a given timepoint then they should be counted under "Not performed". Use mock-up 14.2-12.1 for the following tables:

Table 14.2-13: Analysis of Timed Up-and-Go Test (Seconds) - Efficacy Analysis Set

Protocol: 402-C-331

Pacira Pharmaceuticals (Page X of Y)
Table 14.2-14: Analysis of Stair Climb Test - Efficacy Analysis Set

| Timepoint | Completed Test? | Statistic | EXPAREL 266 mg [N=XX] | EXPAREL 266 mg [N=XX] | No EXPAREL [N=XX] |
|---|---|---|---|---|---|
| Day 1-PM | No | n (%) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| 1 | Yes | n (%) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| | | Odds Ratio EXAPAREL/Placebo | XXX.X | XXX.X | |
| | | Odds Ratio 95% Confidence Interval | (XX.X, XX.X) | (XX.X, XX.X) | |
| Day 2-AM | No | n (%) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| | Yes | n (%) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| | | Odds Ratio EXAPAREL/Placebo | XXX.X | XXX.X | |
| | | Odds Ratio 95% Confidence Interval | (XX.X, XX.X) | (XX.X, XX.X) | |
| Day 2-PM | No | n (%) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| | Yes | n (%) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| | | Odds Ratio EXAPAREL/Placebo | XXX.X | XXX.X | |
| | | Odds Ratio 95% Confidence Interval | (XX.X, XX.X) | (XX.X, XX.X) | |
| Day 3-AM | No | n (%) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| | Yes | n (%) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| | | Odds Ratio EXAPAREL/Placebo | XXX.X | XXX.X | |
| | | Odds Ratio 95% Confidence Interval | (XX.X, XX.X) | (XX.X, XX.X) | |
| Day 3-PM | No | n (%) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| _ | Yes | n (%) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| | | Odds Ratio EXAPAREL/Placebo | XXX.X | XXX.X | |
| | | Odds Ratio 95% Confidence Interval | (XX.X, XX.X) | (XX.X, XX.X) | |
| Etc. | | | | | |

Odds ratio from GEE with effect of treatment and subject within treatment as the repeated effect and logit linking function.

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

**Note to programmer:** Break out by site. Timepoints for this table are Day 1-PM, Day 2-AM, Day 2-PM, Day 3-AM, Day 3-PM, Day 4-AM, Day 4 - PM, and Day 10. If a subject did not have an evaluation at a given timepoint then they should be counted under "No".

**Note to programmer:** For the following region summaries, 'Site:' will be replaced with 'Region:' in the statistical models, row labels, footnotes and by lines of summaries as appropriate. When summarizing by region, the regions are, in order of appearance, US and ROW. There will be no overall region summary presented on these tables.

Use mock-up 14.2-1.1.1 for tables:

Table 14.2-15.1.1.1: Region Analysis of AUC of VAS Pain Intensity Scores through 72 hours - Efficacy Analysis Set - Multiple Imputation Results

Table 14.2-15.1.2.1: Region Analysis of AUC of VAS Pain Intensity Scores through 72 hours - Per-protocol Analysis Set - Multiple Imputation Results

Use mock-up 14.2-2.1.1 for table:

Table 14.2-15.2.1.1: Region Analysis of Postsurgical Total Opioid Consumption (MED mg) through 72 hours - Efficacy Analysis Set

Use mock-up 14.2-2.1.2 for table:

Table 14.2-15.2.1.2: Region Summary of Total Opioid Consumption (MED mg) through 72 hours by Region - Efficacy Analysis Set

Use mock-up 14.2-2.1.3 for table:

Table 14.2-15.2.1.3: Region Summary of Total Opioid Consumption (MED mg) by Time Period - Efficacy Analysis Set

*Use mock-up 14.2-2.1.4 for table:* 

Table 14.2-15.2.1.4: Region Summary of the Number of Times Opioid (Rescue) Medication was used by Subject - Efficacy Analysis Set

*Use mock-up 14.2-2.1.1 for table:* 

Table 14.2-15.2.2.1: Region Analysis of Postsurgical Total Opioid Consumption (MED mg) through 72 hours - Per-protocol Analysis Set

Use mock-up 14.2-2.1.2 for table:


Table 14.2-15.2.2.2: Region Summary of Total Opioid Consumption (MED mg) through 72 hours by Site - Perprotocol Analysis Set

Use mock-up 14.2-2.1.3 for table:

Table 14.2-15.2.2.3: Region Summary of Total Opioid Consumption (MED mg) by Time Period - Per-protocol Analysis Set

Use mock-up 14.2-2.1.4 for table:

Table 14.2-15.2.2.4: Region Summary of the Number of Times Opioid (Rescue) Medication was used by Subject - Per-protocol Analysis Set

Use mock-up 14.2-3.1.1 for table:

Table 14.2-15.3.1.1: Region Analysis of Opioid-Free Subjects through 72 hours - Efficacy Analysis Set

Use mock-up 14.2-3.1.2 for table:

Table 14.2-15.3.1.2: Region Summary of Opioid-Free Subjects through 72 hours by Site - Efficacy Analysis Set

Use mock-up 14.2-3.1.1 for table:

Table 14.2-15.3.2.1: Region Analysis of Opioid-Free Subjects through 72 hours - Per-protocol Analysis Set

Use mock-up 14.2-3.1.2 for table:

Table 14.2-15.3.2.2: Region Summary of Opioid-Free Subjects through 72 hours by Site - Per-protocol Analysis Set


Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-1.1.1: Summary of Clinical Laboratory Data by Timepoint - Hematology - Safety Analysis Set

| Laboratory p | parameter (units) | | | EXPAREL | - <del></del> | | |
|---|---|---|---|---|---|---|---|
| Timepoint | Value | Statistic | 133 mg<br>[N=XXX] | 266 mg<br>[N=XXX] | All<br>EXPAREL<br>[N=XXX] | Placebo<br>[N=XXX] | Total<br>[N=XXX] |
| - | | | | | | | |
| Baseline | Actual | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX | XX | XX |
| Day 10 | Baseline [1] | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX | XX | XX |
| | Actual | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX | XX | XX |
| | Change | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | x.xx |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX | XX | xx |

<sup>[1]</sup> Baseline (prior to surgery) for subjects with data at the timepoint.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

**Note to programmer:** Only present overall sites. Timepoints to appear on this table are, in order of appearance, Baseline (prior to surgery) and Day 10. Do not split timepoint statistics across pages. See

protocol for list of lab analytes. Analytes should be sorted in alphabetical order. Use this mock-up for the following tables:

Table 14.3-1.1.2: Summary of Clinical Laboratory Data by Timepoint - Chemistry - Safety Analysis Set Table 14.3-1.1.3.1: Summary of Clinical Laboratory Data by Timepoint - Urinalysis - Safety Analysis Set

For urinalysis results only numeric results will appear on this table.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-1.1.3.2: Tabulation of Clinical Laboratory Data by Timepoint - Urinalysis - Safety Analysis Set

| | | | | | EXPAREL | | _ | |
|---|---|---|---|---|---|---|---|---|
| | | | | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| Analyte | Timepoint | Category | Statistic | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] |
| Analyte 1 | Baseline | Cat 1 | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Cat 2 | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Etc. | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Day 10 | Cat 1 | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Cat 2 | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Etc. | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Analyte 2 | Baseline | Cat 1 | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Cat 2 | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Etc. | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Day 10 | Cat 1 | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Cat 2 | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Etc. | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Etc. | | | | | | | | |

[1] Baseline (prior to surgery) for subjects with data at the timepoint.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Note to programmer: Only present overall sites. Timepoints to appear on this table are, in order of appearance, Baseline (prior to surgery) and Day 10. Do not split timepoint statistics across pages, if possible. Present all avaliable lab analytes. Categories are the superset of those reported in the data for both timepoints combined. All categories should appear for both timepoints with zeros (0) as counts where needed.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326
Table 14.3-1.2.1: Tabulation of Clinical Laboratory Range by Timepoint - Hematology - Safety Analysis Set

| Laboratory | parameter (ı | ınits) | | EXPAREL | | | |
|---|---|---|---|---|---|---|---|
| | Normal | | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| Timepoint | Range | Statistic | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] |
| Baseline | Below | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Normal | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Above | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Day 10 | Below | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Normal | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Above | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

Note to programmer: Only present overall sites. Timepoints to appear on this table are, in order of appearance, Baseline (prior to surgery) and Day 10. Do not split timepoint statistics across pages. Present all avaliable analytes. Analytes should be sorted in alphabetical order. Use this mock-up for the following tables:

Table 14.3-1.2.2: Tabulation of Clinical Laboratory Range by Timepoint - Chemistry - Safety Analysis Set Table 14.3-1.2.3: Tabulation of Clinical Laboratory Range by Timepoint - Urinalysis - Safety Analysis Set

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-1.3.1: Shift Table for Clinical Laboratory Data by Timepoint - Hematology - Safety Analysis Set

| | | | | Base | line | | |
|---|---|---|---|---|---|---|---|
| | Normal Range | EXPA | REL XXXXXXX [N= | XXX] | I | Placebo [N=XXX | [] |
| Analyte | Day 10 | Below | Normal | Above | Below | Normal | Above |
| Analyte 1 | Below | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Above | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Analyte 2 | Below | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Above | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Analyte 3 | Below | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Above | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ETC . | Below | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Above | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

**Note to programmer:** Only present overall sites. Do not split an analyte across pages. EXPAREL 133 mg and EXPAREL 266 mg will appear on separate pages. All analytes for an EXPAREL group (combined, 133 mg, 266 mg) should appear on consecutive pages before starting the next EXPAREL group. Analytes should be sorted in alphabetical order. Use this mock-up for the following tables:

Table 14.3-1.3.2: Shift Table for Clinical Laboratory Data by Timepoint - Chemistry - Safety Analysis Set Table 14.3-1.3.3: Shift Table for Clinical Laboratory Data by Timepoint - Urinalysis - Safety Analysis Set

Protocol: 402-C-326

Pacira Pharmaceuticals (Page X of Y)
Table 14.3-2.1: Summary of Vital Signs by Timepoint - Safety Analysis Set

| Heart Rate ( | bpm) | | | EXPAREL | | | |
|---|---|---|---|---|---|---|---|
| Timepoint | Value | Statistic | 133 mg<br>[N=XXX] | 266 mg<br>[N=XXX] | All<br>EXPAREL<br>[N=XXX] | Placebo<br>[N=XXX] | Total<br>[N=XXX] |
| Baseline | Actual | n | XX | XX | XX | XX | XX |
| Daseille | ACCUAI | Mean | | | | | |
| | | SD | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | x.xx | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX | XX | XX |
| PACU | Baseline [1] | n | xx | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | X.XX | x.xx | x.xx | X.XX | x.xx |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | XX.X | xx.x | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX | XX | XX |
| | Actual | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | xx.x | xx.x |
| | | SD | X.XX | x.xx | x.xx | x.xx | x.xx |
| | | Minimum | XX | XX | XX | XX | xx |
| | | Median | XX.X | XX.X | XX.X | xx.x | xx.x |
| | | Maximum | XX | XX | XX | XX | XX |
| | Change | n | XX | XX | XX | XX | XX |
| | 5 - | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | X.XX | x.xx | x.xx | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX | XX | XX |

<sup>[1]</sup> Baseline (prior to surgery) for subjects with data at the timepoint.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Note to programmer: Only present overall sites. Vital signs are 'Resting Heart Rate (bpm)', 'Systolic Blood Pressure (mmHg)' and 'Diastolic Blood Pressure (mmHg)'. Timepoints to appear on this table are, in order of

appearance, Baseline (prior to surgery), PACU and, 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120 hours and Days 7 and 10. Do not split timepoint statistics across pages.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-2.2: Summary of Potentially Clinically Significant Abnormal Vital Signs - Safety Analysis Set

| Heart Rate | (bpm) | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | | 133 mg<br>[N=XX] | 266 mg<br>[N=XX] | All EXPAREL [N=XX] | Placebo<br>[N=XX] | Total<br>[N=XXX] |
| Timepoint | Criteria | n (응) | n (%) | n (응) | n (%) | n (응) |
| Baseline | <= 50 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Decrease >= 15 | NA | NA | NA | NA | NA |
| | <= 50 & Decrease >= 15 | NA | NA | NA | NA | NA |
| | >= 120 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <pre>Increase &gt;= 15</pre> | NA | NA | NA | NA | NA |
| | >= 120 & Increase >= 15 | NA | NA | NA | NA | NA |
| Any Time | <= 50 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| After | Decrease >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Baseline | <= 50 & Decrease >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 120 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <pre>Increase &gt;= 15</pre> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 120 & Increase >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc. | <= 50 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Decrease >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <= 50 & Decrease >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 120 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <pre>Increase &gt;= 15</pre> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 120 & Increase >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-2.2: Summary of Potentially Clinically Significant Abnormal Vital Signs - Safety Analysis Set

| Systolic Bl | lood Pressure (mmHg) | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| | | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XXX] |
| Timepoint | Criteria | n (응) | n (응) | n (응) | n (응) | n (응) |
| Baseline | <= 90 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Decrease >= 20 | NA | NA | NA | NA | NA |
| | <= 90 & Decrease >= 20 | NA | NA | NA | NA | NA |
| | >= 180 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <pre>Increase &gt;= 20</pre> | NA | NA | NA | NA | NA |
| | >= 180 & Increase >= 20 | NA | NA | NA | NA | NA |
| Any Time | <= 90 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| After | Decrease >= 20 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Baseline | <= 90 & Decrease >= 20 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 180 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <pre>Increase &gt;= 20</pre> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 180 & Increase >= 20 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc. | <= 90 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Decrease >= 20 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <= 90 & Decrease >= 20 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 180 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <pre>Increase &gt;= 20</pre> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 180 & Increase >= 20 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Source: list SAS datasets used to create table SAS  $\rm X.Y$ 

DDMONYYYYTHH:MM program\_name

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-2.2: Summary of Potentially Clinically Significant Abnormal Vital Signs - Safety Analysis Set

| Diastolic E | Blood Pressure (mmHg) | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | | 133 mg<br>[N=XX] | 266 mg<br>[N=XX] | All EXPAREL [N=XX] | Placebo<br>[N=XX] | Total<br>[N=XXX] |
| Timepoint | Criteria | n (%) | n (%) | n (%) | n (%) | n (%) |
| Baseline | <= 50 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Decrease >= 15 | NA | NA | NA | NA | NA |
| | <= 50 & Decrease >= 15 | NA | NA | NA | NA | NA |
| | >= 105 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <pre>Increase &gt;= 15</pre> | NA | NA | NA | NA | NA |
| | >= 105 & Increase >= 15 | NA | NA | NA | NA | NA |
| Any Time | <= 50 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| After | Decrease >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Baseline | <= 50 & Decrease >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 105 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <pre>Increase &gt;= 15</pre> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 105 & Increase >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc. | <= 50 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Decrease >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <= 50 & Decrease >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 105 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <pre>Increase &gt;= 15</pre> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | >= 105 & Increase >= 15 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Source: list SAS datasets used to create table SAS  $\rm X.Y$ 

DDMONYYYYTHH:MM program\_name

**Note to programmer:** Only present overall sites. Timepoints to appear on this table are, in order of appearance, Baseline (prior to surgery), Any Time After Baseline, PACU and, 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120 hours and Days 7 and 10. Do not split timepoint statistics across pages.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326
Table 14.3-3.1: Summary of Electrocardiogram Interpretation - Investigator Read - Safety Analysis Set

| | | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| Time Point | Interpretation | 133 mg<br>[N=XX]<br>n (%) | 266 mg<br>[N=XX]<br>n (%) | All<br>EXPAREL<br>[N=XX]<br>n (%) | Placebo<br>[N=XX]<br>n (%) | Total<br>[N=XXX]<br>n (%) |
| Baseline (Prior to Surgery) | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, NCS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, CS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Any Time After Baseline | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, NCS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, CS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| At Tmax* | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | N/A | N/A |
| | Abnormal, NCS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | N/A | N/A |
| | Abnormal, CS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | N/A | N/A |
| Etc. | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, NCS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, CS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

\*QuantPharm LLC indicated that the results of the interim PK analysis showed a median Tmax of 60 hours for the 133 mg EXPAREL group and a median Tmax of 78 hours for the 266 mg EXPAREL group. The 'at Tmax' timepoint is the time nearest in absolute value to the population PK estimated median Tmax.

NCS = not clinically significant

CS = clinically significant

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM

program name

Note to programmer: Only present overall sites. Timepoints to appear on this table are, in order of appearance, Baseline (prior to surgery), At any time after baseline, At Tmax, PACU and, 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120 hours and Days 7 and 10. Do not split a timepoint across pages. For the timepoint 'any time after baseline' report the worst interpretation reported at any timepoint but baseline. The 'at Tmax' timepoint is the time nearest in absolute value to the population PK estimated median Tmax.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-3.2: Shift Table for Electrocardiogram Interpretation - Investigator Read - Safety Analysis Set

| | | Baseline | | | |
|---|---|---|---|---|---|
| | | All | L EXPAREL [N=XXX] | Plac | ebo [N=XXX] |
| | | | Abnormal | | Abnormal |
| Time Point | Interpretation | Normal | NCS CS | Normal | NCS CS |
| Any Time | Normal | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) xx (xx.x%) x | x (xx.x%) xx (xx.x%) |
| After | NCS | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) xx (xx.x%) x | x (xx.x%) xx (xx.x%) |
| Baseline | CS | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) xx (xx.x%) x | x (xx.x%) xx (xx.x%) |
| | Normal | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) xx (xx.x%) x | x (xx.x%) xx (xx.x%) |
| | NCS | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) xx (xx.x%) x | x (xx.x%) xx (xx.x%) |
| | CS | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) xx (xx.x%) x | x (xx.x%) xx (xx.x%) |
| At Tmax* | Normal | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) N/A | N/A N/A |
| | NCS | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) N/A | N/A N/A |
| | CS | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) N/A | N/A N/A |
| Etc. | Normal | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) xx (xx.x%) x | x (xx.x%) xx (xx.x%) |
| | NCS | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) xx (xx.x%) x | x (xx.x%) xx (xx.x%) |
| | CS | xx (xx.x%) | xx (xx.x%) xx (xx. | x%) xx (xx.x%) x | x (xx.x%) xx (xx.x%) |

\*QuantPharm LLC indicated that the results of the interim PK analysis showed a median Tmax of 60 hours for the 133 mg EXPAREL group and a median Tmax of 78 hours for the 266 mg EXPAREL group. The 'at Tmax' timepoint is the time nearest in absolute value to the population PK estimated median Tmax.

NCS = not clinically significant

Source: list SAS datasets used to create table

DDMONYYYYTHH:MM program name

Note to programmer: Only present overall sites. Timepoints to appear on this table are, in order of appearance, Baseline (prior to surgery), At any time after baseline, At Tmax, PACU and, 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120 hours and Days 7 and 10. Do not split a timepoint across pages. For the timepoint 'any time after baseline' report the worst interpretation reported at any timepoint but baseline. The 'at Tmax' timepoint is the time nearest in absolute value to the population PK estimated median Tmax. EXPAREL 133 mg and EXPAREL 266 mg will appear on separate pages. All timepoints for an EXPAREL group (All EXPAREL, 133 mg, 266 mg) should appear on consecutive pages before starting the next EXPAREL group.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326

| Table 14.3-4: Summary of Neurological Assessments by Timepoint- Safety Analysis Set | | | | | | |
|---|---|---|---|---|---|---|
| | | | EXPAREL | | | |
| | | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| | | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XXX] |
| Timepoint Assessment | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Baseline (Prior to Surgery) | | | | | | |
| Subject Oriented | No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Numb lips, tongue or mouth | No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Metallic taste | No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Hearing problems | No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Vision problems | No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| - | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Muscle twitching | No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Source: list SAS datasets used to create table
SAS X.Y

DDMONYYYYTHH:MM
program\_name

Note to programmer: Only present overall sites. Timepoints to appear on this table are, in order of appearance, Baseline (prior to surgery), At any time after baseline, PACU and, 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120 hours and Days 7 and 10. Put one timepoint per page. For the timepoint 'any time after baseline' if there is at least one 'yes' at any timepoint other than baseline, the subject will be a 'yes'.

Protocol: 402-C-326

Pacira Pharmaceuticals (Page X of Y)
Table 14.3-5.1: Tabulation of Sensation Tests - Safety Analysis Set

| Location: | location-name (nerv | e name) | | EXPAREL | | | |
|---|---|---|---|---|---|---|---|
| | | | 133 mg<br>[N=XXX] | 266 mg<br>[N=XXX] | All EXPAREL [N=XXX] | Placebo<br>[N=XXX] | Total<br>[N=XXX] |
| Timepoint | Sensation | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Baseline | Cold | Absent<br>Present | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |
| | Pinprick | Absent<br>Present | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |
| | Light Touch | Absent<br>Present | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |
| Pinp | Cold | Absent<br>Present | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |
| | Pinprick | Absent<br>Present | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |
| | Light Touch | Absent<br>Present | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM

program\_name

Note to programmer: Locations to appear on this table, in order, are 'Thigh (Anterior Cutaneous)' and 'Foot (Saphenous)'. Timepoints to appear on this table are, in order, are: Baseline, 15, 30 and 45 minutes and 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108 and 120 hours. Do not split a timepoint across pages.
Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-5.2: Summary of Sensation Loss and Return by Timepoint - Safety Analysis Set

| Location: 10 | cation-name (nerve | name) | | EXPAREL | | | |
|---|---|---|---|---|---|---|---|
| | | 133 mg | | lg 266 mg A | All EXPAREL | Placebo | Total |
| | | | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] |
| Timepoint | Sensation | | n (%) | n (%) | n (%) | n (%) | n (%) |
| At Any Time | Any | Loss | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| _ | _ | Return | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | CPL | Loss | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Return | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | CP | Loss | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Return | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | CL | Loss | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Return | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | PL | Loss | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Return | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Cold (C) | Loss | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Return | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Pinprick (P) | Loss | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Return | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Light Touch (L) | Loss | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Return | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Loss is the absence of sensation

Return is the presence of sensation after a loss of sensation

Sensation: CPL = All; CP = cold & pinprick; CL = cold & light touch; PL = pinprick & light touch

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM

program\_name

Note to programmer: Nerves to appear on this table, in order, are 'All' 'Thigh (Anterior Cutaneous)' and 'Foot (Saphenous)'. Timepoints to appear on this table are, in order, are: At Any Time, 15, 30 and 45 minutes and 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108 and 120 hours. For 'at any time' timepoint subjects' experiencing a loss/return at any time during the study will be counted only once. For 'any' sensation, subjects' experiencing a loss/return for at least one of the sensation at that timepoint will be counted only once. Do not split a timepoint across pages.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-5.3.1: Analysis of Time to First Sensation Loss - Safety Analysis Set

| Location: location-name | e (nerve name) | | | | |
|---|---|---|---|---|---|
| | | 133 mg | 266 mg | All EXPAREL | Placebo |
| | | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] |
| Sensation | Statistic | n (%) | n (%) | n (%) | n (%) |
| Loss | | | | | |
| Ever | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Never* | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Time to First Loss (hrs | 5) | | | | |
| Quartiles [1] | | | | | |
| First (25%) | Estimate | XX.XX | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx, xx.xx) |
| Median (50%) | Estimate | XX.XX | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx, xx.xx) |
| Third (75%) | Estimate | XX.XX | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx, xx.xx) |
| Minimum | Observed | XX.XX | XX.XX | XX.XX | XX.XX |
| Maximum | Observed | xx.xx* | xx.xx* | XX.XX | XX.XX |
| p-value [2] | | 0.xxxx | 0.xxxx | 0.xxxx | |

Loss: absence of at least one of cold, pinprick or light touch sensation.

Time to sensation loss is the time from end of surgery to first loss of sensation.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

\* = censored

Note to programmer: Nerves to appear on this table, in order, are 'All' 'Thigh (Anterior Cutaneous)' and 'Foot (Saphenous)'.

<sup>[1]</sup> Estimates from Kaplan-Meier analysis.

<sup>[2]</sup> p-value from log-rank test with a term for treatment comparing EXPAREL to placebo.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-5.3.2: Analysis of Time to Last Sensation Loss - Safety Analysis Set

| Location: location-name ( | nerve name) | e) EXPAREL | | | |
|---|---|---|---|---|---|
| | | 133 mg | 266 mg | All EXPAREL | Placebo |
| | | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] |
| Sensation | Statistic | n (%) | n (%) | n (%) | n (%) |
| Time to Last Loss (hrs) | | | | | |
| Quartiles [1] | | | | | |
| First (25%) | Estimate | XX.XX | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Median (50%) | Estimate | XX.XX | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Third (75%) | Estimate | XX.XX | xx.xx | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Minimum | Observed | XX.XX | xx.xx | XX.XX | XX.XX |
| Maximum | Observed | XX.XX* | XX.XX* | XX.XX | XX.XX |
| p-value [2] | | 0.xxxx | 0.xxxx | 0.xxxx | |

Loss: absence of at least one of cold, pinprick or light touch sensation.

\* = censored

Return: all 3 (cold, pinprick and light touch) sensations are present after loss of sensation Time to sensation return is the time from first sensation loss to first sensation return.

[1] Estimates from Kaplan-Meier analysis.

[2] p-value from log-rank test with a term for treatment comparing EXPAREL to placebo.

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

Note to programmer: Nerves to appear on this table, in order, are 'All' 'Thigh (Anterior Cutaneous)' and 'Foot (Saphenous)'. If a subject meets the loss criteria at any timepoint, the subject will be counted in 'loss ever' category; otherwise the subject will be counted in 'loss never' category. Note time to last loss will only be provided if more than 10% of the subjects in a treatment arm have more than 1 sensation loss-return cycle.

Protocol: 402-C-326

Pacira Pharmaceuticals (Page X of Y)
Table 14.3-5.4.1: Analysis of Time to First Sensation Return - Safety Analysis Set

| Location: location-name | ne (nerve name) | | EXPAREL | | |
|---|---|---|---|---|---|
| | | 133 mg | 266 mg | All EXPAREL | Placebo |
| | | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] |
| Sensation | Statistic | n (%) | n (%) | n (%) | n (%) |
| Loss Ever | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Return | | | | | |
| Ever | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Never* | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Time to First Return | (hrs) | | | | |
| Quartiles [1] | ( | | | | |
| First (25%) | Estimate | XX.XX | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx, xx.xx) |
| Median (50%) | Estimate | XX.XX | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Third (75%) | Estimate | XX.XX | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx,xx.xx) |
| Minimum | Observed | XX.XX | XX.XX | XX.XX | XX.XX |
| Maximum | Observed | xx.xx* | xx.xx* | XX.XX | XX.XX |
| p-value [2] | | 0.xxxx | 0.xxxx | 0.xxxx | |

Loss: absence of at least one of cold, pinprick or light touch sensation.

Return: all 3 (cold, pinprick and light touch) sensations are present after loss of sensation

Time to sensation return is the time from first sensation loss to first sensation return.

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

\* = censored

Note to programmer: Nerves to appear on this table, in order, are 'All' 'Thigh (Anterior Cutaneous)' and 'Foot (Saphenous)'. This table based on only those subjects who lost sensation (ie, the loss ever row is the population appearing in analyses).

<sup>[1]</sup> Estimates from Kaplan-Meier analysis.

<sup>[2]</sup> p-value from log-rank test with a term for treatment comparing EXPAREL to placebo.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326

Table 14.3-5.4.2: Analysis of Time to Last Sensation Return - Safety Analysis Set

| Location: location-name | | | | | |
|---|---|---|---|---|---|
| (nerve name) | | _ | | | |
| | | 133 mg 266 mg | | All EXPAREL | Placebo |
| | | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] |
| Sensation | Statistic | n (%) | n (%) | n (%) | n (%) |
| Time to Last Return (hrs) | | | | | |
| Quartiles [1] | | | | | |
| First (25%) | Estimate | XX.XX | xx.xx | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx, xx.xx) | (xx.xx,xx.xx) |
| Median (50%) | Estimate | XX.XX | xx.xx | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Third (75%) | Estimate | XX.XX | xx.xx | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Minimum | Observed | XX.XX | XX.XX | XX.XX | XX.XX |
| Maximum | Observed | XX.XX* | XX.XX* | XX.XX | XX.XX |
| p-value [2] | | 0.xxxx | 0.xxxx | 0.xxxx | |

Loss: absence of at least one of cold, pinprick or light touch sensation.

\* = censored

Return: all 3 (cold, pinprick and light touch) sensations are present after loss of sensation Time to sensation return is the time from first sensation loss to first sensation return.

[1] Estimates from Kaplan-Meier analysis.

[2] p-value from log-rank test with a term for treatment comparing EXPAREL to placebo.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Note to programmer: Nerves to appear on this table, in order, are 'All' 'Thigh (Anterior Cutaneous)' and 'Foot (Saphenous)'. 'Loss Ever' counts on this table should agree with 'loss ever' counts on Table 14.3-5.1.1. If a subject meets the return criteria at any time, the subject will be counted in 'return ever' category; otherwise the subject will be counted in the 'return never' category. The sum of 'return ever' and 'return never' should add up to 'loss ever'; subjects who did not experience a loss of sensation cannot have a return of sensation. Only subjects experiencing a 'loss ever' will contribute to the body of this table. Note time to last return will only be provided if more than 10% of the subjects in a treatment arm have more than 1 sensation loss-return cycle.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326

Table 14.3-5.5: Summary of Duration (hrs) of Sensation Loss - Safety Analysis Set

| Location: location-name (nerve name) | | | EXPAREL | | |
|---|---|---|---|---|---|
| (Herve Hame) | | 133 mg | 266 mg | All EXPAREL | Placebo |
| | | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] |
| | Statistic | n (%) | n (%) | n (%) | n (%) |
| otal Duration | n | XX | XX | XX | XX |
| Juliusian | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X . XX | X • XX | x . xx | X.XX |
| | Minimum | XX | XX | XX | XX |
| | Median | XX.X | XX.X | xx.x | XX.X |
| | Maximum | XX | XX | XX | XX |
| Cycle 1 | n | XX | XX | XX | XX |
| - | Mean | XX.X | XX.X | XX.X | xx.x |
| | SD | X.XX | X.XX | x.xx | X.XX |
| | Minimum | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX |
| Etc. | n | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | x.xx | X.XX |
| | Minimum | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX |

Duration is the time between loss and return of sensation.

Total duration is the sum, within a subject, of all sensation loss-return cycles.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Note to programmer: Nerves to appear on this table, in order, are 'All' 'Thigh (Anterior Cutaneous)' and 'Foot (Saphenous)'. Only subjects experiencing a sensation loss will contribute to the body of this table. Note summaries of cycles will only be provided if more than 10% of the subjects in a treatment arm have more than 1 sensation loss-return cycle.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-5.6: Summary of the Number of Sensation Loss-Return Cycles - Safety Analysis Set

| Location: locati | on-name (nerve name) | | EXPAREL | | |
|---|---|---|---|---|---|
| | | 133 mg | 266 mg | All EXPAREL | Placebo |
| | Statistic | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| Count Summary | n | XX | XX | XX | XX |
| - | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | x.xx | X.XX |
| | Minimum | XX.X | XX.X | xx.x | XX.X |
| | Median | XX | XX | xx | XX |
| | Maximum | XX | XX | XX | XX |
| Count Distributi | on | | | | |
| 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| U | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

Note to programmer: Locations to appear on this table, in order, are 'Thigh (Anterior Cutaneous)' and 'Foot (Saphenous)'. Distribution should present all counts up to the highest number of loss-return cycles in the data (U). Only subjects experiencing a sensation loss will contribute to the body of this table. This table will only be provided if at least 1 subject has more than 1 sensation loss-return cycle.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-6.1: Summary of Active Motor Function Loss and Return by Timepoint - Safety Analysis Set

| | | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| | | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] |
| Timepoint | | n (%) | n (%) | n (%) | n (%) | n (응) |
| At Any Time | Loss | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Flexion | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Extension | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | FE | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Return | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| 15 min | Loss | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Flexion | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Extension | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | FE | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Return | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x% |

FE = flexion and extension loss;

Loss (at least one of active flexion or active extension motor functions is lost):

Flexion = angle <  $80^{\circ}$  if baseline  $\geq$   $80^{\circ}$ , otherwise post-baseline change >  $-10^{\circ}$ 

Extension = angle > 10° if baseline  $\leq$  10°, otherwise post-baseline change  $\geq$  10°

Return (Flexion and Extension must return):

Flexion = angle  $\geq$  80° if baseline  $\geq$  80°, otherwise post-baseline change  $\leq$  -10° Extension = angle  $\leq$  10° if baseline  $\leq$  10°, otherwise post-baseline change  $\leq$  10°

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

Note to programmer: Timepoints to appear on this table are, in order, are: At Any Time, 15, 30 and 45 minutes and 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108 and 120 hours. For at any time, the criteria must be met at the same time point to be counted. For example loss in extension need only be met any timepoint during the study, but flexion and extension loss (FE) must be met at the same timepoint to be counted under at any time.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-6.2: Analysis of Time to Onset of Motor Function Loss - Efficacy Analysis Set

| | Statistic | EXPAREL 133 mg<br>[N=XX] | EXPAREL 266 mg<br>[N=XX] | Placebo<br>[N=XX] |
|---|---|---|---|---|
| Number of Subjects with | | | | |
| Motor Function Loss | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No Motor Function Loss | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time to Loss | | | | |
| Quartiles [1] | | | | |
| First (25%) | Estimate | xx.xx | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx, xx.xx) |
| Median (50%) | Estimate | xx.xx | xx.xx | xx.xx |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx, xx.xx) |
| Third (75%) | Estimate | XX.XX | XX.XX | xx.xx |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx, xx.xx) |
| Minimum | Observed | XX.XX | xx.xx | xx.xx |
| Maximum | Observed | xx.xx* | xx.xx* | xx.xx |
| p-value [2] | | 0.xxxx | 0.xxxx | |

Loss (at least one of active flexion or active extension motor functions is lost):

Flexion = angle  $< 80^{\circ}$  if baseline  $\geq 80^{\circ}$ , otherwise post-baseline change  $> -10^{\circ}$ 

Extension = angle >  $10^{\circ}$  if baseline  $\leq 10^{\circ}$ , otherwise post-baseline change  $\geq 10^{\circ}$ 

CI = confidence interval

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM

program\_name

<sup>\*</sup> indicates censored observation

<sup>[1]</sup> Estimates from Kaplan-Meier analysis.

<sup>[2]</sup> p-value from log-rank test with a term for treatment comparing EXPAREL to placebo.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326

Table 14.3-6.3: Analysis of Time to Return of Motor Function - Efficacy Analysis Set

| | Statistic | EXPAREL 133 mg<br>[N=XX] | EXPAREL 266 mg<br>[N=XX] | Placebo<br>[N=XX] |
|---|---|---|---|---|
| Number of Subjects with | | | | |
| Motor Function Return | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No Motor Function Return | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time to Return | | | | |
| Quartiles [1] | | | | |
| First (25%) | Estimate | xx.xx | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Median (50%) | Estimate | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Third (75%) | Estimate | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Minimum | Observed | XX.XX | xx.xx | XX.XX |
| Maximum | Observed | xx.xx* | xx.xx* | XX.XX |
| p-value [2] | | 0.xxxx | 0.xxxx | |

Return (Flexion and Extension must return):

Flexion = angle  $\geq$  80° if baseline  $\geq$  80°, otherwise post-baseline change  $\leq$  -10°

Extension = angle  $\leq$  10° if baseline  $\leq$  10°, otherwise post-baseline change  $\leq$  10°

CI = confidence interval

Source: list SAS datasets used to create table

DDMONYYYYTHH:MM program name

SAS X.Y

<sup>\*</sup> indicates censored observation

<sup>[1]</sup> Estimates from Kaplan-Meier analysis.

<sup>[2]</sup> p-value from log-rank test with a term for treatment comparing EXPAREL to placebo.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-6.4: Summary of Motor Function Assessments by Timepoint - Safety Analysis Set

| Active Fle | xion (degrees) | | | EXPAREL | | | |
|---|---|---|---|---|---|---|---|
| | | | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| Timepoint | Value | Statistic | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] | [N=XXX] |
| Baseline | Actual | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX | XX | XX |
| 15 | Danalina [1] | | | | | | |
| 15 min | Baseline [1] | n<br>Marana | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX | XX | XX |
| | Actual | n | XX | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX | xx | XX |
| | Change | n | XX | XX | XX | XX | XX |
| | Change | Mean | XX.X | | XX.X | XX.X | |
| | | SD | | XX.X | | | XX.X |
| | | Minimum | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | XX | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Maximum | XX | XX | XX | XX | XX |

<sup>[1]</sup> Baseline (prior to surgery) for subjects with data at the timepoint.

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

Note to programmer: Motor assessments to appear on this table, in order, are: 'Active Flexion (degrees)', 'Active Extension (degrees)', 'Passive Flexion (degrees)' and 'Passive Extension (degrees)'. Timepoints to appear on this table are, in order, are: Baseline, 15, 30 and 45 minutes and 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108 and 120 hours.


Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-7.1: Overview of Treatment-Emergent Adverse Events (TEAEs) - Safety Analysis Set

| | | EXPAREL | | | |
|---|---|---|---|---|---|
| | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| Number of | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Maximum Severity of Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Maximum Severity of Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Maximum Severity of Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| At least one Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| At least one Serious | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects Discontinued due to TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Died on Study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Related TEAEs are those AEs indicated as 'possible', 'probable' or 'definite' related by the investigator on the AE CRF.

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

Note to programmer: Only present overall sites. All categories on this table should appear, even if not present in the data.

SAS X.Y

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-7.1.2: Summary of Incidence of Treatment-Emergent Adverse Events (TEAEs) - Safety Analysis Set

| | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
|---|---|---|---|---|---|
| System Organ Class | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| Preferred Term | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with at least one TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1.1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1.2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2.1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2.2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ETC. | | | | | |

Adverse events coded using the Medical Dictionary for Regulatory Activities (MedDRA TBD).

Sorted by descending total incidence by system organ class and preferred term within system organ class.

Subjects experiencing the same TEAE more than once are counted only once at each summary level.

Source: list SAS datasets used to create table

DDMONYYYYTHH:MM program name

Note to programmer: Only present overall sites. Use mock-up Table 14.3-2.1.2 for the following tables:

Table 14.3-7.1.3: Summary of Incidence of Study Drug-Related Treatment-Emergent Adverse Events (TEAEs) -Safety Analysis Set

Table 14.3-7.1.4: Summary of Incidence of Treatment-Emergent Adverse Events (TEAEs) Leading to Study Withdrawal - Safety Analysis Set

Table 14.3-7.1.5: Summary of Incidence of Study Drug-Related Treatment-Emergent Adverse Events (TEAEs) Leading to Study Withdrawal - Safety Analysis Set

For related tables add the following footnote to the table:

Related TEAEs are those AEs indicated as 'possible', 'probable' or 'definite' related by the investigator on the AE CRF.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-7.1.6: Summary of Incidence of Treatment-Emergent Adverse Events (TEAEs) by Severity - Safety Analysis Set

| | | | EXPAREL | | | |
|---|---|---|---|---|---|---|
| | | | 266 mg | All | _ | Total |
| | | 133 mg | [N=XX] | EXPAREL | Placebo | [N=XX] |
| System Organ Class | | [N=XX] | n (%) | [N=XX] | [N=XX] | n (%) |
| Preferred Term | Severity | n (%) | | n (%) | n (%) | |
| Subjects with at least one TEAE | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| - | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1.1 | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Adverse events coded using the Medical Dictionary for Regulatory Activities (MedDRA TBD).

Sorted by descending total incidence by system organ class and preferred term within system organ class.

Subjects experiencing the same TEAE more than once are counted only once at each summary level.

Source: list SAS datasets used to create table
SAS X.Y

DDMONYYYYTHH:MM program name

Pacira Pharmaceuticals Protocol: 402-C-326 (Page X of Y) Table 14.3-7.1.7: Summary of Incidence of Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug - Safety Analysis Set

EXPAREL 266 mg All Total

| System Organ Class<br>Preferred Term | Relation | 133 mg<br>[N=XX]<br>n (%) | [N=XX]<br>n (%) | EXPAREL [N=XX] n (%) | Placebo<br>[N=XX]<br>n (%) | [N=XX]<br>n (%) |
|---|---|---|---|---|---|---|
| Subjects with at least one TEAE | Unrelated Unlikely Possible Probable Definite | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| SOC1 | Unrelated Unlikely Possible Probable Definite | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| PT1.1 | Unrelated<br>Unlikely<br>Possible<br>Probable<br>Definite | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

Adverse events coded using the Medical Dictionary for Regulatory Activities (MedDRA TBD). Sorted by descending total incidence by system organ class and preferred term within system organ class.

Subjects experiencing the same TEAE more than once are counted only once at each summary level.

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name Note to programmer: Only present overall sites. For related tables add the following footnote to the table, "Related TEAEs are those AEs indicated as 'possible', 'probable' or 'definite' related by the investigator on the AE CRF." Use indicated mock-up for the following tables:

Use mock-up 14.7-1.1

Table 14.3-7.2.1: Overview of Serious Treatment-Emergent Adverse Events (TEAEs) - Safety Analysis Set  $Use\ mock-up\ 14.7-1.2$ 

Table 14.3-7.2.2: Summary of Incidence of Serious Treatment-Emergent Adverse Events (TEAEs) - Safety Analysis Set

Use mock-up 14.7-1.3

Table 14.3-7.2.3: Summary of Incidence of Study Drug-Related Serious Treatment-Emergent Adverse Events (TEAEs) - Safety Analysis Set

Use mock-up 14.7-1.4

Table 14.3-7.2.4: Summary of Incidence of Serious Treatment-Emergent Adverse Events (TEAEs) Leading to Study Withdrawal - Safety Analysis Set

Use mock-up 14.7-1.5

Table 14.3-7.2.5: Summary of Incidence of Study Drug-Related Serious Treatment-Emergent Adverse Events (TEAEs) Leading to Study Withdrawal - Safety Analysis Set

Use mock-up 14.7-1.6

Table 14.3-7.2.6: Summary of Incidence of Serious Treatment-Emergent Adverse Events (TEAEs) Resulting in Death - Safety Analysis Set

Use mock-up 14.7-1.7

Table 14.3-7.2.7: Summary of Incidence of Study Drug-Related Serious Treatment-Emergent Adverse Events (TEAEs) Resulting in Death - Safety Analysis Set

Use mock-up 14.7-1.1

Table 14.3-7.3.1: Overview of Treatment-Emergent Adverse Events (TEAEs) of Special Interest - Safety Analysis Set

Use mock-up 14.7-1.2

Table 14.3-7.3.2: Summary of Incidence of Treatment-Emergent Adverse Events (TEAEs) of Special Interest - Safety Analysis Set

Use mock-up 14.7-1.3

Table 14.3-7.3.3: Summary of Incidence of Study Drug-Related Treatment-Emergent Adverse Events (TEAEs) of Special Interest - Safety Analysis Set

Use mock-up 14.7-1.4

Table 14.3-7.3.4: Summary of Incidence of Treatment-Emergent Adverse Events (TEAEs) of Special Interest Leading to Study Withdrawal - Safety Analysis Set

Use mock-up 14.7-1.5


Table 14.3-7.3.5: Summary of Incidence of Study Drug-Related Treatment-Emergent Adverse Events (TEAEs) of Special Interest Leading to Study Withdrawal - Safety Analysis Set

Use mock-up 14.7-1.6

Table 14.3-7.3.6: Summary of Incidence of Treatment-Emergent Adverse Events (TEAEs) of Special Interest Resulting in Death - Safety Analysis Set

Use mock-up 14.7-1.7

Table 14.3-7.3.7: Summary of Incidence of Study Drug-Related Treatment-Emergent Adverse Events (TEAEs) of Special Interest Resulting in Death - Safety Analysis Set

**Note to programmer:** Use mock-up 14.1-4.1 for tables:

Table 14.3-8.1: Incidence of Prior Medications - Safety Analysis Set.

On this table change the footnote 'Intraoperatives medications are those indicated as such by the investigator' to read 'Prior medications are those stopped before start of study drug administration.'

Table 14.3-8.2: Incidence of Concomitant Medications - Safety Analysis Set.

On this table change the footnote 'Intraoperatives medications are those indicated as such by the investigator' to read 'Concomitant medications are those taken between the start of study drug administration and discharge from study and are not designated intraoperative medications.'

**Note to programmer:** For the following tables, only present US and ROW regions; there is no overall regions group. All of the following mock-ups will put the region as a by-line title in the table.

Use mock-up 14.3-5.1 for table:

Table 14.3-9.1.1: Region Tabulation of Sensation Tests - Safety Analysis Set

Use mock-up 14.3-5.2 for table:

Table 14.3-9.1.2: Region Summary of Sensation Loss and Return by Timepoint - Safety Analysis Set

Use mock-up 14.3-5.3 for table:

Table 14.3-9.1.3: Region Analysis of Time to Sensation Loss - Safety Analysis Set

Use mock-up 14.3-5.4 for table:

Table 14.3-9.1.4: Region Analysis of Time to Sensation Return - Safety Analysis Set

Use mock-up 14.3-5.5 for table:

Table 14.3-9.1.5: Region Summary of Duration (hrs) of Sensation Loss - Safety Analysis Set

Use mock-up 14.3-6.1 for table:

Table 14.3-9.2.1: Region Summary of Active Motor Function Loss and Return by Timepoint - Safety Analysis Set

Use mock-up 14.3-6.2 for table:

Table 14.3-9.2.2: Region Analysis of Time to Onset of Motor Function Loss - Efficacy Analysis Set

Use mock-up 14.3-6.3 for table:

Table 14.3-9.2.3: Region Analysis of Time to Return of Motor Function - Efficacy Analysis Set

Use mock-up 14.3-6.4 for table:

Table 14.3-9.2.4: Region Summary of Motor Function Assessments by Timepoint - Safety Analysis Set


Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-9.3.1: Region Overview of Treatment-Emergent Adverse Events (TEAEs) - Safety Analysis Set

| Region: US | | EXPAREL | | | |
|---|---|---|---|---|---|
| | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| Number of | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Maximum Severity of Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Maximum Severity of Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Maximum Severity of Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| At least one Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| At least one Serious | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects Discontinued due to TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Died on Study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

**Note to programmer:** Only present US and ROW regions; there is no overall regions group. All categories on this table should appear, even if not present in the data.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Table 14.3-9.3.2: Region Summary of Incidence of Treatment-Emergent Adverse Events (TEAEs) - Safety

| 70 | 1 | | O - L |
|-----|--------|-------|-------|
| Ana | 1 77.5 | 3 I S | Set |

| Region: | | EXPAREL | | _ | • |
|---|---|---|---|---|---|
| | 133 mg | 266 mg | All EXPAREL | Placebo | Total |
| System Organ Class | [N=XX] | [N=XX] | [N=XX] | [N=XX] | [N=XX] |
| Preferred Term | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with at least one TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1.1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1.2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2.1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2.2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ETC. | | | | | |

Adverse events coded using the Medical Dictionary for Regulatory Activities (MedDRA TBD).

Sorted by descending total incidence by system organ class and preferred term within system organ class.

Sorted by descending total incidence by system organ class and preferred term within system organ class. Subjects experiencing the same TEAE more than once are counted only once at each summary level.

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

**Note to programmer:** Only present US and ROW regions; there is no overall regions group. Use this mock-up for table:

Table 14.3-9.3.3: Region Summary of Incidence of Serious Treatment-Emergent Adverse Events (TEAEs) - Safety Analysis Set

# 15. TABLE OF CONTENTS FOR LISTING MOCK-UPS

| LISTING 16.2-1: SUBJECT DISPOSITION – ALL SUBJECTS | 133 |
|---|---|
| LISTING 16.2-2: RANDOMIZATION AND ANALYSIS SETS – RANDOMIZED SUBJECTS | 134 |
| LISTING 16.2-3: DEMOGRAPHICS – ALL SUBJECTS | 135 |
| LISTING 16.2-4: HEIGHT AND WEIGHT – ALL SUBJECTS | 136 |
| LISTING 16.2-5: SURGERY – RANDOMIZED SUBJECTS | 137 |
| LISTING 16.2-6: VISUAL ANALOG SCALE (VAS) – RANDOMIZED SUBJECTS | 138 |
| LISTING 16.2-7.1: RESCUE MEDICATION TOTAL DOSE (MED MG) AND OPIOID-FREE STAR - RANDOMIZED SUBJECTS | ATUS<br>139 |
| LISTING 16.2-7.2: RESCUE MEDICATION – RANDOMIZED SUBJECTS | 140 |
| LISTING 16.2-8: OVERALL BENEFIT OF ANALGESIA – RANDOMIZED SUBJECTS | 141 |
| LISTING 16.2-9: SUBJECT SATISFACTION WITH POST-SURGICAL PAIN CONTROL – RANDOMIZED SUBJECTS | 142 |
| LISTING 16.2-10: MODIFIED POST-ANESTHESIA DISCHARGE SCORING SYSTEM (MPADS RANDOMIZED SUBJECTS | SS)–<br>143 |
| LISTING 16.2-11: DAY 29 PHONE CALL – RANDOMIZED SUBJECTS | 144 |
| LISTING 16.2-12: HEMATOLOGY – RANDOMIZED SUBJECTS | 145 |
| LISTING 16.2-13: CHEMISTRY – RANDOMIZED SUBJECTS | 145 |
| LISTING 16.2-14.1: URINALYSIS – NUMERIC RESULTS – RANDOMIZED SUBJECTS | 145 |
| LISTING 16.2-14.2: URINALYSIS – CHARACTER RESULTS – RANDOMIZED SUBJECTS | 146 |
| LISTING 16.2-15: VITAL SIGNS ASSESSMENT – ALL SUBJECTS | 147 |
| LISTING 16.2-16: ELECTROCARDIOGRAM FINDINGS – INVESTIGATOR ASSESSMENT – A SUBJECTS | ALL<br>148 |
| LISTING 16.2-17: NEUROLOGICAL ASSESSMENT – ALL SUBJECTS | 149 |
| LISTING 16.2-18.1: SENSORY FUNCTION ASSESSMENT – ALL SUBJECTS | 150 |
| LISTING 16.2-18.2: TIME TO LOSS AND RETURN OF SENSORY FUNCTION – RANDOMIZE SUBJECTS | D<br>151 |
| LISTING 16.2-19.1.1: ACTIVE MOTOR FUNCTION ASSESSMENT – ALL SUBJECTS | 152 |
| LISTING 16.2-19.1.2: PASSIVE MOTOR FUNCTION ASSESSMENT – ALL SUBJECTS | 153 |
| LISTING 16.2-19.2: TIME TO LOSS AND RETURN OF MOTOR FUNCTION – RANDOMIZED SUBJECTS | 154 |
| LISTING 16.2-20: TIMED WALK TEST – RANDOMIZED SUBJECTS | 155 |
| LISTING 16.2-21: TIMED UP-AND-GO TEST – RANDOMIZED SUBJECTS | 156 |
| LISTING 16.2-22: STAIR CLIMBING TEST – RANDOMIZED SUBJECTS | 157 |
| LISTING 16.2-23.1: ALL ADVERSE EVENTS – ALL SUBJECTS | 158 |
| LISTING 16.2-23.2.1: TREATMENT-EMERGENT ADVERSE EVENTS – RANDOMIZED SUBJ | ECTS158 |
| LISTING 16.2-23.2.2: TREATMENT-EMERGENT STUDY DRUG RELATED ADVERSE EVEN RANDOMIZED SUBJECTS | TS –<br>158 |
| LISTING 16.2-23.3; ALL SERIOUS ADVERSE EVENTS – ALL SUBJECTS | 158 |

| SUBJECTS 15 | _ |
|---|---|
| LISTING 16.2-23.4.2: TREATMENT-EMERGENT STUDY DRUG RELATED SERIOUS ADVERSE EVENTS – RANDOMIZED SUBJECTS 15 | 58 |
| LISTING 16.2-23.5.1: TREATMENT-EMERGENT ADVERSE EVENTS OF SPECIAL INTEREST – RANDOMIZED SUBJECTS 15 | 58 |
| LISTING 16.2-23.5.2: TREATMENT-EMERGENT STUDY DRUG RELATED ADVERSE EVENTS OF SPECIAL INTEREST – RANDOMIZED SUBJECTS 15 | 58 |
| LISTING 16.2-24.1: ALL PRIOR AND CONCOMITANT MEDICATIONS – ALL SUBJECTS 15 | 59 |
| LISTING 16.2-24.2: PRIOR MEDICATIONS – RANDOMIZED SUBJECTS 15 | 59 |
| LISTING 16.2-24.3: CONCOMITANT MEDICATIONS – RANDOMIZED SUBJECTS 15 | 59 |
| LISTING 16.2-25: MEDICAL HISTORY – ALL SUBJECTS 16 | 50 |
| LISTING 16.2-26: INTRAOPERATIVE OPIOIDS – RANDOMIZED SUBJECTS 16 | 51 |
| LISTING 16.2-27: STUDY DRUG ADMINISTRATION – RANDOMIZED SUBJECTS 16 | 52 |
| LISTING 16.2-28: URINE DRUG SCREEN, ALCOHOL BLOOD TEST AND PREGNANCY TEST – ALL SUBJECTS 16 | 53 |
| LISTING 16.2-29: ADMISSION AND DISCHARGE – RANDOMIZED SUBJECTS 16 | 54 |
| LISTING 16.2-30: UNIQUE ADVERSE EVENTS TERMS AND ASSOCIATED CODED TERMS 16 | 55 |
| LISTING 16.2-31: UNIQUE MEDICATION TERMS AND ASSOCIATED CODED TERMS 16 | 56 |
| LISTING 16.2-32: PROTOCOL DEVIATIONS 16 | 57 |

| Pacira Pharmaceuticals, | Inc. |
|-------------------------|------|
| EXPAREL | |

### 402-C-326 (TKA FNB) Statistical Analysis Plan

| Pacira Pharmac | ra Pharmaceuticals (Page X | | (of Y) | Protocol: 402-C-326 |
|---|---|---|---|---|
| Listing 16.2-1 | : Subject Dispos | | | |
| TREATMENT: tre | eatment-name | | | _ |
| | Date of | | | _ |
| Site Subject | Last Visit | End of Study Status | Specify | |
| XXX XXX-YYYY | DDMONYYYY | | | |

Source: list SAS datasets used to create table SAS  $\rm X.Y$ 

DDMONYYYYTHH:MM program\_name

Note to programmer: End of study status for subject who early terminated from the study is the primary reason for termination. If subject discontinued due to an AE then the reason should read 'ADVERSE EVENT, AE # X'. If subject discontinued due to death the reason should read 'DEATH ON DDMONYYYY'. For those reasons that also collected a specify text, that text belongs in the specify column.

Pacira Pharmaceuticals, Inc. EXPAREL

402-C-326 (TKA FNB) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-2: Randomization and Analysis Sets - Randomized Subjects

TREATMENT: treatment-name

| Randomization | | | n | | Analys | is Set | |
|---|---|---|---|---|---|---|---|
| Site | Subject | Date and Time | Number | Safety | Efficacy | Per-protocol | PK |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | XXXXX | X | X | X | Х |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

Protocol: 402-C-326

Note to programmer: Analysis set will by 'Y' if subject in set, blank otherwise.

| Pacira Pharmaceuticals, Inc |
|-----------------------------|
| EXPAREL |

## 402-C-326 (TKA FNB) Statistical Analysis Plan

| Pacir | a Pharmace | uticals | | | (Page | X of Y) | Protocol: 402-C-32 | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Listi | ng 16.2-3: | Demograph | ics - All Sub | jects | | | | | | |
| TREAT | MENT: trea | tment-name | | | | | | | | |
| | Subject | Subject | | Age | | | | ASA | | |
| Site | ID | Initials | Birth Date | (yrs) | Sex | Race | Ethnicity | Class | Region | Country |
| XXX | XXX-YYYY | AMZ | DDMONYYYY | ΥΥ | XXXXXX | XXXXXXXXXXXXXXXXXXX | xxxxxxxx | V | XXX | XXXXXXX |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

Note to programmer: If race is 'other' then race should be 'Other: other-specify-text'.

Pacira Pharmaceuticals, Inc. EXPAREL

402-C-326 (TKA FNB) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-4: Height and Weight - All Subjects

TREATMENT: treatment-name

| Site | Subject | Height and Weight<br>Collection Date | Height (cm) | Weight (kg) | Body Mass<br>Index<br>(kg/m²) |
|---|---|---|---|---|---|
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | XXX.X | XXX.X | XX.X |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

Pacira Pharmaceuticals, Inc. EXPAREL

402-C-326 (TKA FNB) Statistical Analysis Plan

Pacira Pharmaceuticals
Listing 16.2-5: Surgery - Randomized Subjects

(Page X of Y)

| TREAT | TMENT: trea | atment-name | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| , | | | | | | | Incision | Bupivacaine HCl | |
| | | | Start | Stop | Duration | | Length | Administration | |
| Site | Subject | Date | Time | Time | (hrs) | Location | (cm) | Time | Anesthesia Type |
| XXX | XXX-YYYY | DDMONYYYY | HH:MM | HH:MM | X.X | XXXXX | XX.X | HH:MM | XXXXXXXXXXXXXXXXXXXX |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program\_name

Protocol: 402-C-326

Note to programmer: If anesthesia type is 'other' then text should read 'other: specify-text'.

(Page X of Y)

Listing 16.2-6: Visual Analog Scale (VAS) - Randomized Subjects

TREATMENT: treatment-name

| | | | Ti | me From Do | se | | |
|---|---|---|---|---|---|---|---|
| | | | Scheduled | Actual | Deviation | VAS | Pain-Free |
| Site | Subject | Date Time | (hr) | (hr) | (hrs) | (cm) | $(VAS \leq 1.5cm)$ |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | XX.XX | XX.XX | XXXX | XX.X | V |

VAS: 0=No pain to 10=Worst Pain Imaginable

ND=Not Done NA=Not Applicable

\* = out of window

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

Note to programmer: Sort by VAS collection date and time. If VAS was taken due to rescue medication dosing, put RESCUE in scheduled column and hours from dose in actual column - leave deviation column blank. Do not split a subject's data across pages if it can be avoided. Pain-free will have Y if VAS  $\leq$  1.5 otherwise blank. An asterisk (\*) will be placed next to the deviation if an assessment is out of window. See Table of Time and Events for windows.

### 402-C-326 (TKA FNB) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Listing 16.2-7.1: Rescue Medication Total Dose (MED mg) and Opioid-free Status - Randomized Subjects TREATMENT: treatment-name 96 hrs 24-48hrs 48-72hrs 72-96 hrs Site Subject 72 hrs 24 hrs 48 hrs Opioid-Free XXX XXX-YYYY XXXX.X XXXX.X XXXX.X XXXX.X XXXX.X XXXX.X XXXX.X NO XXX XXX-YYYY YES

Total dose is dose from end of surgery through timepoint.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

**Note to programmer:** If medication is 'Other', text should read 'Other: specify-text'. Sort by date and time within subject.

## 402-C-326 (TKA FNB) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-7.2: Rescue Medication - Randomized Subjects

| | | | Time to | | Dose | Conversion | Dose<br>(MED | |
|---|---|---|---|---|---|---|---|---|
| Site | Subject | Date and Time | Rescue (hr) | Medication | (units) | Factor | mg) | Route |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | XXX.X | XXXXXXXXXXX | XX (XXXX) | X.XX | XXX.X | XXXXXXX |
| | | DDMONYYYYTHH:MM | XXX.X | XXXXXXXXXXX | XX(XXXX) | X.XX | XXX.X | XXXXXXX |
| | | DDMONYYYYTHH:MM | XXX.X | XXXXXXXXXXX | XX (XXXX) | X.XX | XXX.X | XXXXXXX |
| | | DDMONYYYYTHH:MM | XXX.X | XXXXXXXXXXX | XX (XXXX) | X.XX | XXX.X | XXXXXXX |

Time to rescue is time from end of surgery to rescue medication dose.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program\_name

Protocol: 402-C-326

**Note to programmer:** If medication is 'Other', text should read 'Other: specify-text'. Sort by date and time within subject.

Protocol: 402-C-326

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-8: Overall Benefit of Analgesia - Randomized Subjects

| | | Assessment | | | | Question | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Schedule | Actual | Deviation | | | | | | | | Total |
| Site | Subject | Date and Time | (hrs) | (hrs) | (hrs) | 1 | 2 | 3 | 4 | 5 | 6 | 7 | Score |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | 24 | XX.X | XX.X | Х | Х | Х | Х | Х | Х | Х | XX |
| | | DDMONYYYYTHH:MM | 72 | XX.X | XX.X | X | Χ | Χ | X | X | Χ | Χ | XX |
| | | DDMONYYYYTHH:MM | 240 (D10) | XXX.X | XX.X | X | X | X | X | X | X | X | XX |

Total score = sum of questions 1 to 6 scores minus question 7 score plus 4.

- 1) Please rate your current pain at rest on a scale between 0=minimal pain and 4=maximum imaginable pain
- 2) Please grade any distress and bother from vomiting in the past 24 h (0=not at all to 4=very much)
- 3) Please grade any distress and bother from itching in the past 24 h (0=not at all to 4=very much)
- 4) Please grade any distress and bother from sweating in the past 24 h (0=not at all to 4=very much)
- 5) Please grade any distress and bother from freezing in the past 24 h (0=not at all to 4=very much)
- 6) Please grade any distress and bother from dizziness in the past 24 h (0=not at all to 4=very much)
- 7) How satisfied are you with your pain treatment during in the past 24 h (0=not at all to 4=very much)

Source: list SAS datasets used to create table

DDMONYYYYTHH:MM

program name

(Page X of Y)

Listing 16.2-9: Subject Satisfaction with Post-Surgical Pain Control - Randomized Subjects

| Site | Subject | Assessment | Date and Time | Rating | Score |
|---|---|---|---|---|---|
| XXX | XXX-YYYY | 24 hr | DDMONYYYYTHH:MM | EXTREMELY DISSATISFIED | 1 |
| ΛΛΛ | XXX-1111 | 72 hr | DDMON11111HH:MM | DISSATISFIED | 2 |
| | | Day 10 | DDMONYYYYTHH:MM | NEITHER SATISFIED NOR DISSATISFIED | 3 |
| XXX | XXX-YYYY | 24 hr | DDMONYYYYTHH:MM | SATISFIED | 4 |
| | | 72 hr | DDMONYYYYTHH:MM | EXTREMELY SATISIFIED | 5 |
| | | Day 10 | DDMONYYYYTHH:MM | EXTREMELY SATISIFIED | 5 |

Time to rescue is time from end of surgery to rescue medication dose.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

(Page X of Y)

Listing 16.2-10: Modified Post-Anesthesia Discharge Scoring System (MPADSS) - Randomized Subjects

| TREATMENT: treati | ment-name |
|-------------------|-----------|
|-------------------|-----------|

| | | Assessment | | | | | Question | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Schedule | Actual | Deviation | | | | | | Total |
| Site | Subject | Date and Time | (hrs) | (hrs) | (hrs) | 1 | 2 | 3 | 4 | 5 | Score |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | 24 | XX.X | XX.X | X | X | X | Χ | X | XX |
| | | DDMONYYYYTHH:MM | 72 | XX.X | XX.X | Χ | Χ | Χ | Χ | Χ | XX |
| | | DDMONYYYYTHH:MM | 240 (D10) | XXX.X | XX.X | X | Χ | Χ | Χ | Χ | XX |

\*=out of window

Total score = sum of scores.

- 1) Vital signs:  $2 = \le 20\%$ ; 1 = 20-40%; 0 = >40% of preoperative value.
- 2) Ambulation: 2 = steady gait/no dizziness; 1 = with assistance; 0 = none/dizziness
- 3) Nausea and Vomiting: 2 = minimal; 1 = moderate; 0 = severe
- 4) Pain: 2 = minimal; 1 = moderate; 0 = severe
- 5) Surgical bleeding: 2 = minimal; 1 = moderate; 0 = severe

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

(Page X of Y)

Listing 16.2-11: Day 29 Phone Call - Randomized Subjects

| TREATMENT: | treatment-name |
|------------|----------------|

| | | | | | | Number of | pain-related | |
|---|---|---|---|---|---|---|---|---|
| Site | Subject | Date | Schedule<br>(days) | Actual<br>(days) | Deviation<br>(days) | Phone<br>Calls | Visits | Total |
| XXX | XXX-YYYY | DDMONYYYY | 29 | XX.X | XX.X | XX | XX | XXXX |
| XXX | XXX-YYYY | DDMONYYYY | 29 | XX.X | XX.X | XX | XX | XXXX |
| XXX | XXX-YYYY | DDMONYYYY | 29 | XX.X | XX.X | XX | XX | XXXX |

Total = sum of calls and visits.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326
## 402-C-326 (TKA FNB) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-12: Hematology - Randomized Subjects

| TREAT | MENT: trea | tment-name | · | | • | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Normal | Range | | | |
| Site | Subject | Visit | Date and Time | Analyte (units) | | Low | High | Result | Change | Flag |
| XXX | XXX-YYYY | Screening | DDMONYYYYTHH:MM | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | _ | Н |
| | | | | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | _ | |
| | | | | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | _ | L |
| | | | | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | _ | |
| | | Baseline | DDMONYYYYTHH:MM | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | _ | |
| | | | | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | _ | |
| | | | | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | _ | L |
| | | | | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | _ | |
| | | Day 10 | DDMONYYYYTHH:MM | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | XX.X | |
| | | | | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | XX.X | |
| | | | | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | XX.X | L |
| | | | | XXXXXXXXXXXXXXX | (units) | XXX.XX | XXX.XX | XXX.XX | XX.X | |

Flag: L=below normal range; H=above normal range.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

**Note to programmer:** Sort by date and time within subject and analyte alphabetically within date. Change is only calculated for Day 10 visit. Use this mock-up for the following listings:

Listing 16.2-13: Chemistry - Randomized Subjects

Listing 16.2-14.1: Urinalysis - Numeric Results - Randomized Subjects

(Page X of Y)

Listing 16.2-14.2: Urinalysis - Character Results - Randomized Subjects

| TREAT | MENT: treatm | ent-name | | | | | |
|---|---|---|---|---|---|---|---|
| Site | Subject | Visit | Date and Time | Analyte | Normal Criteria | Result | Flag |
| XXX | XXX-YYYY | Screening | DDMONYYYYTHH:MM | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXXX | A |
| | | | | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXX | |
| | | | | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXX | |
| | | | | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXXX | |
| | | Baseline | DDMONYYYYTHH:MM | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXX | А |
| | | | | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXX | |
| | | | | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXXX | |
| | | | | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXXX | |
| | | Day 10 | DDMONYYYYTHH:MM | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXX | |
| | | | | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXXX | |
| | | | | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXX | |
| | | | | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXXX | |

Flag: A = abnormal.

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program\_name

Protocol: 402-C-326

Note to programmer: Sort by date and time within subject and analyte alphabetically within date.

(Page X of Y)

Listing 16.2-15: Vital Signs Assessment - All Subjects

| TREATMENT: | treatment-name |
|------------|----------------|

| | | | | | | Heart | Rate | Bl | ood Press | sure (mml | Hg) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Assessment | | | (b | pm) | Syst | olic | Dias | tolic |
| | | | Schedule | Actual | Dev. | | | | | | |
| Site | Subject | Date and Time | (hrs) | (hrs) | (hrs) | Actual | Change | Actual | Change | Actual | Chang |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | Screening | _ | _ | XX | _ | XXX | _ | XX | _ |
| | | DDMONYYYYTHH:MM | Baseline | - | - | XX | _ | XXX | _ | XX | _ |
| | | DDMONYYYYTHH:MM | PACU | - | - | XX | XX | XXX | -X | XX | X |
| | | DDMONYYYYTHH:MM | 6 | XXX.XX | XXX | XX | -XX | XXX | X | XX | -X |
| | | DDMONYYYYTHH:MM | 12 | XXX.XX | XXX | XX | XX | XXX | X | XX | X |
| | | DDMONYYYYTHH:MM | 24 | XXX.XX | XXX | XX | XX | XXX | -X | XX | X |
| | | DDMONYYYYTHH:MM | 36 | XXX.XX | XXX | XX | XX | XXX | X | XX | X |
| | | DDMONYYYYTHH:MM | 48 | XXX.XX | XXX | 0XX | -XX | XXX | X | XX | -X |
| | | DDMONYYYYTHH:MM | 60 | XXX.XX | XXX | XX | XX | XXX | -X | XX | X |
| | | DDMONYYYYTHH:MM | 66 | XXX.XX | XXX | XX | XX | XXX | -X | XX | -X |
| | | DDMONYYYYTHH:MM | 72 | XXX.XX | XXX | XX | -XX | XXX | X | XX | X |
| | | DDMONYYYYTHH:MM | 78 | XXX.XX | XXX* | XX | XX | XXX | -X | XX | -X |
| | | DDMONYYYYTHH:MM | 84 | XXX.XX | XXX | XX | -XX | XXX | X | XX | X |
| | | DDMONYYYYTHH:MM | 96 | XXX.XX | XXX | XX | XX | XXX | X | XX | X |
| | | DDMONYYYYTHH:MM | 108 | XXX.XX | XXX | XX | -XX | XXX | -X | XX | X |
| | | DDMONYYYYTHH:MM | 120 | XXX.XX | XXX | XX | XX | XXX | X | XX | -X |
| | | DDMONYYYYTHH:MM | 168 (D7) | XXX.XX | XXX | XX | XX | XXX | X | XX | X |
| | | DDMONYYYYTHH:MM | 240 (D10 | XXX.XX | XXX | XX | -XX | XXX | -X | XX | X |

\*=out of window

Change is change from baseline (Preop).

Source: list SAS datasets used to create table

SAS X.Y

@=potentially clinically significant value

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

**Note to programmer:** Sort by date and time within subject. An asterisk (\*) will be placed next to the deviation if an assessment is out of window. See Table of Time and Events for windows.

(Page X of Y)

Listing 16.2-16: Electrocardiogram Findings - Investigator Assessment - All Subjects

| | | | Assessment | | | | |
|---|---|---|---|---|---|---|---|
| | | | Schedule | Actual | Deviation | _ | |
| Site | Subject | Date and Time | (hrs) | (hrs) | (hrs) | Finding | |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | Screening | _ | _ | Normal | |
| | | DDMONYYYYTHH:MM | Preop | _ | _ | Abnormal, | clinically significant |
| | | DDMONYYYYTHH:MM | PACU | _ | _ | Abnormal, | not clinically significant |
| | | DDMONYYYYTHH:MM | 6 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 12 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 24 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 36 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 48 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 60 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 66 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 72 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 78 | XXX.XX | XXX* | Normal | |
| | | DDMONYYYYTHH:MM | 84 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 96 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 108 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 120 | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 168 (D7) | XXX.XX | XXX | Normal | |
| | | DDMONYYYYTHH:MM | 240 (D10 | XXX.XX | XXX | Normal | |

<sup>\*=</sup>out of window

Source: list SAS datasets used to create table SAS  ${\tt X.Y}$ 

DDMONYYYYTHH:MM program\_name

Protocol: 402-C-326

**Note to programmer:** Sort by date and time within subject. An asterisk (\*) will be placed next to the deviation if an assessment is out of window. See Table of Time and Events for windows.


(Page X of Y)

Listing 16.2-17: Neurological Assessment - All Subjects

| | | | Assessment | | | | | Ques | tion | L | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Schedule | Actual | Deviation | | | | | | |
| ite | Subject | Date and Time | (hrs) | (hrs) | (hrs) | 1 | 2 | 3 | 4 | 5 | ( |
| XX | XXX-YYYY | DDMONYYYYTHH:MM | Screening | _ | _ | Х | Х | Х | Χ | Х | 2 |
| | | DDMONYYYYTHH:MM | Preop | _ | _ | X | Χ | Χ | Χ | Χ | |
| | | DDMONYYYYTHH:MM | PACU | _ | _ | X | Χ | Χ | Χ | Χ | |
| | | DDMONYYYYTHH:MM | 6 | XXX.XX | XXX | X | X | Χ | X | Χ | |
| | | DDMONYYYYTHH:MM | 12 | XXX.XX | XXX | X | X | Χ | X | Χ | |
| | | DDMONYYYYTHH:MM | 24 | XXX.XX | XXX | X | Χ | Χ | Χ | Χ | |
| | | DDMONYYYYTHH:MM | 36 | XXX.XX | XXX | X | Χ | X | X | X | |
| | | DDMONYYYYTHH:MM | 48 | XXX.XX | XXX | X | X | Χ | X | Χ | |
| | | DDMONYYYYTHH:MM | 60 | XXX.XX | XXX | X | Χ | Χ | X | Χ | |
| | | DDMONYYYYTHH:MM | 66 | XXX.XX | XXX | X | Χ | Χ | X | Χ | |
| | | DDMONYYYYTHH:MM | 72 | XXX.XX | XXX | X | X | Χ | X | Χ | |
| | | DDMONYYYYTHH:MM | 78 | XXX.XX | XXX* | X | Χ | Χ | X | Χ | |
| | | DDMONYYYYTHH:MM | 84 | XXX.XX | XXX | X | Χ | Χ | X | Χ | |
| | | DDMONYYYYTHH:MM | 96 | XXX.XX | XXX | X | Χ | Χ | X | Χ | |
| | | DDMONYYYYTHH:MM | 108 | XXX.XX | XXX | X | Χ | Χ | Χ | Χ | |
| | | DDMONYYYYTHH:MM | 120 | XXX.XX | XXX | X | Χ | Χ | X | X | |
| | | DDMONYYYYTHH:MM | 168 (D7) | XXX.XX | XXX | X | Χ | Χ | X | X | |
| | | DDMONYYYYTHH:MM | 240 (D10 | XXX.XX | XXX | Х | Χ | X | Χ | Χ | |

<sup>\*=</sup>out of window

- 1) Is subject oriented?
- 2) Do you have numbness of the lips, the tongue or around the mouth?
- 3) Do you have a metallic taste in your mouth?
- 4) Are you having problems with your hearing not related to the use of a hearing aid?
- 5) Are you having problems with your vision not related to the use of eye glasses?
- 6) Are your muscles twitching?

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

**Note to programmer:** Sort by date and time within subject. An asterisk (\*) will be placed next to the deviation if an assessment is out of window. See Table of Time and Events for windows.

(Page X of Y)

Listing 16.2-18.1: Sensory Function Assessment - All Subjects
TREATMENT: treatment-name

| | | | Assessment | | | Anterio | or Cutaneo | us Nerve | Sapl | henous N | erve |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Schedule | Actual | Dev. | | Pin- | Light | | Pin- | Light |
| Site | Subject | Date and Time | (hrs) | (hrs) | (hrs) | Cold | prick | Touch | Cold | prick | Touch |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | Screening | _ | _ | + | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | Baseline | _ | _ | + | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | PACU | - | - | + | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | 6 | XXX.XX | XXX | + | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | 9 | XXX.XX | XXX | -L | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | 12 | XXX.XX | XXX | _ | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | 18 | XXX.XX | XXX | _ | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | 24 | XXX.XX | XXX | _ | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | 36 | XXX.XX | XXX | _ | -L | + | + | + | + |
| | | DDMONYYYYTHH:MM | 48 | XXX.XX | XXX | +R | +R | + | + | + | + |
| | | DDMONYYYYTHH:MM | 60 | XXX.XX | XXX | + | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | 72 | XXX.XX | XXX | + | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | 84 | XXX.XX | XXX | + | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | 96 | XXX.XX | XXX | + | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | 108 | XXX.XX | XXX | + | + | + | + | + | + |
| | | DDMONYYYYTHH:MM | 120 | XXX.XX | XXX | + | + | + | -L | + | + |
| | | DDMONYYYYTHH:MM | Unsched. | _ | _ | + | + | + | _ | + | + |

\*=out of window

'-/+'=Absent/Present; L/R=Loss/Return of sensation Source: list SAS datasets used to create table

Unsched=Unscheduled DDMONYYYYTHH:MM program name

SAS X.Y

Protocol: 402-C-326

Note to programmer: Sort by date and time within subject. An asterisk (\*) will be placed next to the deviation if an assessment is out of window. See Table of Time and Events for windows.

## 402-C-326 (TKA FNB) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-18.2: Time to Loss and Return of Sensory Function - Randomized Subjects

| TREATI | MENT: trea | tment-nan | пе | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Loss | s-Return | | Date and Time of | | Time t | o (hrs) |
| | | Cycle | | | | | Loss | Return |
| Site | Subject | Number | Location | Dose | Loss | Return | [1] | [2] |
| | XXX- | | | | | | | |
| XXX | YYYY | 1 | Anterior | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM | XXX.X | XXX.X |
| | | 2 | Saphenous | _ | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM | XXX.X | XXX.X |
| | | ••• | Saphenous | _ | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM | XXX.X | XXX.X |
| | | n | Anterior | _ | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM* | XXX.X | XXX.X* |
| | | Total | | _ | _ | _ | _ | D.D |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

**Note to programmer:** Sort by date and time within subject. In total row, D.D is sum of durations from all cycles. Some subjects may have more losses of sensation than returns.


<sup>[1]</sup> Time to loss is the time from start of study drug administration to loss of sensation

<sup>[2]</sup> Time to return is time the time from most recent loss of sensation to return of sensation

<sup>\*=</sup>Censored return (time of last sensory assessment)

(Page X of Y)

Listing 16.2-19.1.1: Active Motor Function Assessment - All Subjects

TREATMENT: treatment-name

| | | | Assessment | | | Flexion<br>(degrees) | | Extension (degrees) | |
|---|---|---|---|---|---|---|---|---|---|
| Site | Subject | Date and Time | Schedule<br>(hrs) | Actual<br>(hrs) | Dev.<br>(hrs) | Act | Chg | Act | Chọ |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | Screening | _ | _ | XXX | _ | XXX | _ |
| | | DDMONYYYYTHH:MM | Baseline | _ | _ | XXX | _ | XXX | _ |
| | | DDMONYYYYTHH:MM | PACU | _ | _ | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 6 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 9 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 12 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 18 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 24 | XXX.XX | XXX | XXX | XXX | XXX | XX |
| | | DDMONYYYYTHH:MM | 36 | XXX.XX | XXX | XXX | XXX | XXX | XX |
| | | DDMONYYYYTHH:MM | 48 | XXX.XX | XXX | XXXL | XXX | XXX | XX |
| | | DDMONYYYYTHH:MM | 60 | XXX.XX | XXX | XXX | XXX | XXX | XX |
| | | DDMONYYYYTHH:MM | 72 | XXX.XX | XXX | XXX | XXX | XXX | XX |
| | | DDMONYYYYTHH:MM | 84 | XXX.XX | XXX | XXXR | XXX | XXX | XX |
| | | DDMONYYYYTHH:MM | 96 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 108 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 120 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | Unsched. | _ | - | XXX | XXX | XXX | XX |

\*=out of window

L=Loss of function/R=Return of function

Unsched=Unscheduled

Protocol: 402-C-326

Act = Actual; Chg = Change from Baseline (Preop) Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program\_name

**Note to programmer:** Sort by date and time within subject. An asterisk (\*) will be placed next to the deviation if an assessment is out of window. See Table of Time and Events for windows.

(Page X of Y)

Listing 16.2-19.1.2: Passive Motor Function Assessment - All Subjects

TREATMENT: treatment-name

| | | | Assessment | | | Flexion<br>(degrees) | | Extension (degrees) | |
|---|---|---|---|---|---|---|---|---|---|
| Site | Subject | Date and Time | Schedule<br>(hrs) | Actual<br>(hrs) | Dev.<br>(hrs) | Act | Chg | Act | Chọ |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | Screening | _ | _ | XXX | _ | XXX | _ |
| | | DDMONYYYYTHH:MM | Baseline | _ | _ | XXX | _ | XXX | _ |
| | | DDMONYYYYTHH:MM | PACU | _ | _ | XXX | XXX | XXX | XXΣ |
| | | DDMONYYYYTHH:MM | 6 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 9 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 12 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 18 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 24 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 36 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 48 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 60 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 72 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 84 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 96 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 108 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | 120 | XXX.XX | XXX | XXX | XXX | XXX | XXX |
| | | DDMONYYYYTHH:MM | Unsched. | _ | _ | XXX | XXX | XXX | XX |

\*=out of window

SAS X.Y

L=Loss of function/R=Return of function

Unsched=Unscheduled

Protocol: 402-C-326

Act = Actual; Chg = Change from Baseline (Preop) Source: list SAS datasets used to create table

DDMONYYYYTHH:MM program\_name

**Note to programmer:** Sort by date and time within subject. An asterisk (\*) will be placed next to the deviation if an assessment is out of window. See Table of Time and Events for windows.

(Page X of Y)

Listing 16.2-19.2: Time to Loss and Return of Motor Function - Randomized Subjects

| TREAT | MENT: trea | tment-name | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Loss-Re | eturn | | Date and Time of | | Time to (hrs) | |
| | | | Active | | | | Loss | Return |
| Site | Subject | Cycle Number | Assessment | Dose | Loss | Return | [1] | [2] |
| XXX | XXX-YYYY | 1 | Flexion | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM | XXX.X | XXX.X |
| | | 2 | Extension | - | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM | XXX.X | XXX.X |
| | | | Flexion | _ | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM | XXX.X | XXX.X |
| | | n | Flexion | _ | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM* | XXX.X | XXX.X* |
| | | Total | | _ | _ | _ | _ | D.D |

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

**Note to programmer:** Sort by date and time within subject. In total row, D.D is the time from first loss of motor function to last return of motor function. Some subjects may have more losses of motor function than returns.


<sup>[1]</sup> Time to loss is the time from start of study drug administration to loss of motor function

<sup>[2]</sup> Time to return is time the time from most recent loss of to return of motor function Total Return is the time from first loss to last return of motor function.

<sup>\*=</sup>Censored return (time of last sensory assessment)

## 402-C-326 (TKA FNB) Statistical Analysis Plan

Protocol: 402-C-326

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-20: Timed Walk Test - Randomized Subjects

| Site | Subject | Timepoint | Date and Time | Done? | Reason not done | Distance<br>(m) | Walking<br>Aid? | Physical<br>Assistance |
|---|---|---|---|---|---|---|---|---|
| XXX | XXX-YYYY | Day 1-PM | DDMONYYYYTHH:MM | Y | | XX | XXX | X |
| | | Day 2-AM | DDMONYYYYTHH:MM | N | XXXXXXXXXXXXXXX | | | |
| | | Day 2-PM | DDMONYYYYTHH:MM | Y | | XX | XX | X |
| | | Day 3-AM | DDMONYYYYTHH:MM | Y | | XX | XX | X |
| | | Day 3-PM | DDMONYYYYTHH:MM | Y | | XX | XX | X |
| | | Day 4-AM | DDMONYYYYTHH:MM | Y | | XX | XX | X |
| | | Day 4-PM | DDMONYYYYTHH:MM | Y | | XX | XX | X |
| | | Day 15 | DDMONYYYYTHH:MM | Y | | XX | XX | X |

Physical Assistance: 1=Total Assistance 2=Maximal Assistance 3=Moderate Assistance 4=Minimal Assistance 5=Supervision 6=Modified Independence 7=Complete Independence DDMONYYYYTHH:MM

SAS X.Y program\_name

Protocol: 402-C-331

Pacira Pharmaceuticals (Page X of Y) Listing 16.2-21: Timed Up-and-go Test - Randomized Subjects

DDMONYYYYTHH:MM

DDMONYYYYTHH:MM

Day 4-PM

Day 15

TREATMENT: treatment-name Change Duration from of Test Aid Physical Reason not Subject Timepoint Baseline (seconds) Assistance Site Date and Time Done? done Used? XXX XXX-YYYY Baseline N/A Υ DDMONYYYYTHH:MM Day 1-PM DDMONYYYYTHH:MM XX.X Υ Day 2-AM XX.X Ν XXX DDMONYYYYTHH:MM XXXXXXXXX XXX Day 2-PM XX.X Υ DDMONYYYYTHH:MM Υ Day 3-AM XX.X DDMONYYYYTHH:MM Day 3-PM XX.X Υ DDMONYYYYTHH:MM Day 4-AM Υ DDMONYYYYTHH:MM XX.X

> XX.X XX.X

| Physical Assistance: | 1=Total Assistance | 2=Maximal Assistance | 3=Moderate Assistance |
|---|---|---|---|
| 4=Minimal Assistance | 5=Supervision | 6=Modified Independence | 7=Complete Independence |
| Source: list SAS datase | ts used to create table | | DDMONYYYYTHH:MM |
| SAS X.Y | | | program name |

Υ

Υ

Note to Programmer: All of the Not Done visits should be included in this listing. In addition, in ADQS, variable CHG, (Change from Baseline), is present, include this in the listing.

Pacira Pharmaceuticals
Listing 16 2-22: Stair Climbing Tost - P

(Page X of Y)

Listing 16.2-22: Stair Climbing Test - Randomized Subjects

| | | | | | | Successfully |
|---|---|---|---|---|---|---|
| Site | Subject | Timepoint | Date and Time | Done? | Reason not done | Completed |
| | XXX- | | | | | |
| XXX | YYYY | Day 1-PM | DDMONYYYYTHH:MM | Y | | |
| | | Day 2-AM | DDMONYYYYTHH:MM | N | XXXXXXXXXXXXXX | XXX |
| | | Day 2-PM | DDMONYYYYTHH:MM | Y | | |
| | | Day 3-AM | DDMONYYYYTHH:MM | Y | | |
| | | Day 3-PM | DDMONYYYYTHH:MM | Y | | |
| | | Day 4-AM | DDMONYYYYTHH:MM | Y | | |
| | | Day 4-PM | DDMONYYYYTHH:MM | Y | | |
| | | Day 15 | DDMONYYYYTHH:MM | Y | | |
| | | Day 15 | DDMON11111IIII.MM | 1 | | |

Physical Assistance: 1=Total Assistance 4=Minimal Assistance 5=Supervision Source: list SAS datasets used to create table SAS X.Y 2=Maximal Assistance 6=Modified Independence 3=Moderate Assistance 7=Complete Independence DDMONYYYYTHH:MM program\_name

Protocol: 402-C-331

Pacira Pharmaceuticals (Page X of Y)

Listing 16.2-23.1: All Adverse Events - All Subjects

Treatment: treatment-name

| Site | Subject | TEAE | Data Type | Data | | |
|---|---|---|---|---|---|---|
| XXX | XXX-YYYY | N | Start | DDMONYYYYTHH:MM | | |
| | | | Stop | DDMONYYYYTHH:MM | | |
| | | | AE Number | X | | |
| | | | System Organ Class | XXXXXXXXXXXXXXX | | |
| | | | Preferred | XXXXXXXXXXXXXXXXX | | |
| | | | Verbatim | XXXXXXXXXXXXXXXXXXX | | |
| | | | Severity | XXXXXXX | | |
| | | | Relationship to Study Drug | XXXXXXX | | |
| | | | Action Taken | XXXXXXXXXXXXXXXXXX | | |
| | | | | | Outcome | XXXXXXXXXXXX |
| | | | Serious | XXX | | |
| | | | Serious Cause(s) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | |

TEAE: Treatment-emergent AE (Y=TEAE/N=Not TEAE) Source: list SAS datasets used to create listing

SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

Note to programmer: If AE is ongoing, put ONGOING in stop row. Do not split an AE across pages. Insert a page break between subjects. Use this mock-up for the following listings:

Listing 16.2-23.2.1: Treatment-emergent Adverse Events - Randomized Subjects

Listing 16.2-23.2.2: Treatment-emergent Study Drug Related Adverse Events - Randomized Subjects

Listing 16.2-23.3: All Serious Adverse Events - All Subjects

Listing 16.2-23.4.1: Treatment-emergent Serious Adverse Events - Randomized Subjects

Listing 16.2-23.4.2: Treatment-emergent Study Drug Related Serious Adverse Events - Randomized Subjects

Listing 16.2-23.5.1: Treatment-emergent Adverse Events of Special Interest - Randomized Subjects

Listing 16.2-23.5.2: Treatment-emergent Study Drug Related Adverse Events of Special Interest - Randomized Subjects

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326

Listing 16.2-24.1: All Prior and Concomitant Medications - All Subjects

Treatment: treatment-name

| Site | Subject | Category | Data Type | Data |
|---|---|---|---|---|
| XXX | XXX-YYYY | | Start | DDMONYYYYTHH:MM |
| | | | Stop | DDMONYYYYTHH:MM |
| | | | Medication Number | X |
| | | | ATC Level 1 | XXXXXXXXXXXXXXX |
| | | | ATC Level 2 | XXXXXXXXXXXXXXXXX |
| | | | ATC Level 3 | XXXXXXXXXXXXXXXXXXX |
| | | | ATC Level 4 | XXXXXXXXXXXXXXXXX |
| | | | Preferred Name | XXXXXXXXXXXXXXXXXX |
| | | | Verbatim | XXXXXXXXXXXXXXXXX |
| | | | Route | XXXXXXX |
| | | | Frequency | XXXXXXX |
| | | | Given for AE or MH? | XXXXXXXXXXXXXXXXXX AE # XX (or MH # XX) |

ATC=Anatomical therapeutic class

Source: list SAS datasets used to create listing

SAS X.Y

DDMONYYYYTHH:MM program name

Note to programmer: If medication is ongoing, put ONGOING in stop row. Do not split a medication across pages. Insert a page break between subjects. Values for category column are: CONCOMITANT; SURGICAL/ANESTHESIA; NON-MEDICATION; PRIOR. Use this mock-up for the following listings:

Listing 16.2-24.2: Prior Medications - Randomized Subjects

Listing 16.2-24.3: Concomitant Medications - Randomized Subjects

Pacira Pharmaceuticals (Page X of Y)

Listing 16.2-25: Medical History - All Subjects

Treatment: treatment-name

| Site | Subject | Data Type | Data |
|------|----------|--------------------|---------------------|
| XXX | XXX-YYYY | Start | DDMONYYYY |
| | | Stop | DDMONYYYY |
| | | System Organ Class | XXXXXXXXXXXXXXX |
| | | Preferred | XXXXXXXXXXXXXXXXX |
| | | History Verbatim | XXXXXXXXXXXXXXXXXX |
| | | Start | DDMONYYYY |
| | | Stop | DDMONYYYY |
| | | System Organ Class | XXXXXXXXXXXXXXX |
| | | Preferred | XXXXXXXXXXXXXXXXX |
| | | History Verbatim | XXXXXXXXXXXXXXXXXXX |

Source: list SAS datasets used to create listing SAS X.Y

DDMONYYYYTHH:MM program\_name

Protocol: 402-C-326

Pacira Pharmaceuticals, Inc. EXPAREL

402-C-326 (TKA FNB) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-26: Intraoperative Opioids - Randomized Subjects

| | | <u> </u> | - | | | |
|---|---|---|---|---|---|---|
| TREAT | MENT: treat | ment-name | | | | |
| Site | Subject | Administered | Name | Dose | Unit | Route |
| XXX | XXX-YYYY | YES | <i>OPIOID-NAME</i> | XXX.XX | (UNITS) | XXXX |
| XXX | XXX-YYYY | NO | | | | |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

XXX-YYYY

DDMONYYYY

HH:MM

HH:MM

XXX

| Pacira | . Pharmaceuti | cals | | | (Page X of Y) | Protocol: | 402-C-326 |
|---|---|---|---|---|---|---|---|
| Listing 16.2-27: Study Drug Administration - Randomized Subjects | | | | | | | |
| TREATM | MENT: treatme | nt-name | | | | | |
| | | | Start | Stop | Total Volume | | |
| Site | Subject | Date | Time | Time | (mL) | | |

XXX

Source: list SAS datasets used to create table
SAS X.Y

DDMONYYYYTHH:MM
program\_name

XXXXXXXX

XXXXXXXX

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-326 Listing 16.2-28: Urine Drug Screen, Alcohol Blood Test and Pregnancy Test - All Subjects

TREATMENT: treatment-name Blood Site Subject Visit Urine Drug Alcohol Pregnancy XXX Screening XXXXXXXX XXX-YYYY XXXXXXXX XXXXXXXX Day 0 (Preop) XXXXXXXX XXXXXXXX XXXXXXXX Screening XXX XXX-YYYY XXXXXXXX XXXXXXXX XXXXXXXX Day 0 (Preop) XXXXXXXX XXXXXXXX XXXXXXXX Screening XXX XXX-YYYY XXXXXXXX XXXXXXXX XXXXXXXX Day 0 (Preop) XXXXXXXX XXXXXXXX XXXXXXXX XXX Screening XXX-YYYY XXXXXXXX XXXXXXXX XXXXXXXX

Source: list SAS datasets used to create table DDMONYYYYTHH:MM program name

XXXXXXXX

Day 0 (Preop)

Pacira Pharmaceuticals (Page X of Y)
Listing 16.2-29: Admission and Discharge - Randomized Subjects

| TREATMENT: treat | ment-name |
|------------------|-----------|
|------------------|-----------|

| | Date and Time | | |
|------|---------------|-----------------|------------------|
| Site | Subject | Admission | Discharge |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | DDMONYYYYTHH: MM |
| XXX | XXX-YYYY | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM |

\*=out of window

Total score = sum of scores.

- 1) Vital signs:  $2 = \le 20\%$ ; 1 = 20-40%; 0 = >40% of preoperative value.
- 2) Ambulation: 2 = steady gait/no dizziness; 1 = with assistance; 0 = none/dizziness
- 3) Nausea and Vomiting: 2 = minimal; 1 = moderate; 0 = severe
- 4) Pain: 2 = minimal; 1 = moderate; 0 = severe
- 5) Surgical bleeding: 2 = minimal; 1 = moderate; 0 = severe

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-326

| Pacira Pharmaceuticals, Inc. |
|------------------------------|
| EXPAREL |

| Listing 16.2-30: Unique Adverse | E Events Terms and Associated Coded Terms |
|---|---|
| MedDRA Terms | |
| SOC | |
| Preferred Term | Verbatim(s) |
| SOC1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| PT1.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| PT1.2 | xxxxxxxxxxxxxxxxxxxxxxx |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| SOC2 | |
| PT2.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | xxxxxxxxxxxxxxxxxxxxxxx |

402-C-326 (TKA FNB) Statistical Analysis Plan

program\_name

Note to programmer: Sort by SOC and preferred term in alphabetical order

SAS X.Y

SAS X.Y

program\_name

| Pacira Pharmaceuticals | (Page X of Y) | Protocol: 402-C-327 |
|---|---|---|
| Listing 16.2-31: Unique Medication | Terms and Associated Coded Terms | |
| Who Drug Dictionary Terms | | |
| ACT1 | | |
| ACT2 | | |
| ACT3 | | |
| ACT4 | | |
| Preferred name | Verbatim(s) | |
| ATC1 | | |
| ATC1.2 | | |
| PN1.2.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXX | |
| PN1.2.2 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| ATC2 | | |
| ATC2.2 | | |
| ATC2.3 | | |
| ATC2.4 | | |
| PN2.2.3.4.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXX | |
| Coded using Who Drug Dictionary Source: list SAS datasets used to | create listing | DDMONYYYYTHH:MM |
| bource. Itse bab databets used to | oreace insting | |

Note to programmer: Sort by ATC1, ATC2, ATC3, ATC4 and preferred name in alphabetical order

Pacira Pharmaceuticals, Inc. EXPAREL

402-C-326 (TKA FNB) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

TREATMENT: treatment-name

Surgery: surgery-type

Nerve Block: nerve-block type

Listing 16.2-32: Protocol Deviations

| | ier ve proci | | | | |
|------|--------------|----------|-----------|------|--------------------|
| Site | Subject | Category | Important | Date | Description |
| XXX | XXX-YYYY | XXXXXX | XXX | | XXXXXXXXXXXXXXXXX |
| ΛΛΛ | XXX-1111 | ^^^^ | AAA | | XXXXXXXXXXXXXXXXXX |

Categories: Important, might significantly impact; not-important, none to minimal impact on study outcomes. Important:

Source: list SAS datasets used to create listing SAS X.Y

DDMONYYYYTHH:MM program name

Protocol: 402-C-327

Note to programmer: Subjects may have multiple deviations. Sort deviations by treatment, surgery type, nerve block type, site, subject, then category 'Important' followed by 'Not-Important' and finally important ('YES' then 'NO'). Date may or may not include time.

# 16. TABLE OF CONTENTS FOR FIGURE MOCK-UPS

| PLOT OF MEAN PAIN INTENSITY SCORE (VAS) VS TIME THROUGH 72 HOURS – EFFICACY ANALYSIS SET | 73 |
|---|---|
| PLOT OF MEAN PAIN INTENSITY SCORE (VAS) VS TIME THROUGH 72 HOURS – PER-PROTOCOL ANALYSIS SET | 73 |
| PLOT OF MEAN PAIN INTENSITY SCORE (VAS) VS TIME THROUGH 96 HOURS – EFFICACY ANALYSIS SET | 73 |
| PLOT OF MEAN PAIN INTENSITY SCORE (VAS) VS TIME THROUGH 96 HOURS – PER-PROTOCOL ANALYSIS SET | 73 |
| LOT OF INDIVIDUAL SUBJECT PAIN INTENSITY SCORE (VAS) VS TIME<br>THROUGH 72 HOURS – EFFICACY ANALYSIS SET | 73 |
| LOT OF INDIVIDUAL SUBJECT PAIN INTENSITY SCORE (VAS) VS TIME THROUGH 96 HOURS – EFFICACY ANALYSIS SET | 73 |

Figure Mock-up 1



Figure Mock-up 2



Figure Mock-up 3

Subject=XXX-XXX-XXXX Treatment=EXPAREL XXX mg



Gray bars indicate rescue medication windows

Figure Mock-up 4





Gray bars indicate rescue medication windows

Note to programmers: The colors and symbols used in the figure mock-ups are not correct per the SAP description; all figures created should use the SAP defined colors and symbols. In figure mock-ups 3 and 4: the gray bars highlight the rescue medication windows for that subject; the time axes are set to ensure the entire period is captured and doesn't end at the limits of the figure. Use the indicated figure mock-up for the following figures.

### Use Figure mock-up 1 for the following the x-axis should track through 76 hours:

Figure 1.1: Plot of Mean Pain Intensity Score (VAS) vs Time through 72 hours - Efficacy Analysis Set Figure 1.2: Plot of Mean Pain Intensity Score (VAS) vs Time through 72 hours - Per-protocol Analysis Set

### Use Figure mock-up 2 for the following (the x-axis should track through 100 hours):

Figure 2.1: Plot of Mean Pain Intensity Score (VAS) vs Time through 96 hours - Efficacy Analysis Set Figure 2.2: Plot of Mean Pain Intensity Score (VAS) vs Time through 96 hours - Per-protocol Analysis Set

Use Figure mock-up 3 for the following (use actual hours since the end of surgery and not scheduled hours, include all VAS scores collected, the x-axis should track through 76 hours):

Figure 3: Plot of Individual Subject Pain Intensity Score (VAS) vs Time through 72 hours - Efficacy Analysis Set

Use Figure mock-up 4 for the following (use actual hours since the end of surgery and not scheduled hours, include all VAS scores collected, the x-axis should track through 100 hours):

Figure 4: Plot of Individual Subject Pain Intensity Score (VAS) vs Time through 96 hours - Efficacy Analysis Set